## **CLINICAL STUDY PROTOCOL**

CiloMecT: Effect of Cilostazol as an add-on treatment to a single antiplatelet agent (Acetylsalicylic acid or Clopidogrel) on platelet function testing and bleeding time in healthy volunteers

NCT Number: NCT02554721

PRT NO.: 21-13-102

Version Date: 07 March 2018 (Version 11.0)

# Protocol and/or Protocol Amendments Table of Contents

| Table of Contents | 1 |
|---------------------------------------------------------|----|
| Study 21-13-102 Protocol Amendment 10; 07 March 2018 | 2 |
| Protocol_21-13-102_SmPC Pletal Tabletten Ger_Jan2017 | 81 |
| Protocol_21-13-102_SmPC Aspirin protect 100 Ger_Mar2017 | 86 |
| Protocol 21-13-102 SmPC Plavix Ger Jan2018 | 90 |

## Investigational Medicinal Product OPC-13013

## CLINICAL TRIAL PROTOCOL

Protocol Title: CiloMecT: Effect of Cilostazol as an add-on treatment to a single antiplatelet agent (Acetylsalicylic acid or Clopidogrel) on platelet function testing and bleeding time in healthy volunteers

Protocol No. 21-13-102 EudraCT No. 2013-002633-38

| Drug Development Phase: | 1 |
|---|---|
| Sponsor: | Otsuka Pharmaceutical Co., Ltd.<br>2-9 Kanda-Tsukasamachi, Chiyoda-ku<br>Tokyo<br>Japan |
| Sponsor Representatives: | |
| Clinical Director: | PPD |
| Immediately Reportable Events: | Pharmacovigilance Region Europe<br>Phone: +49 69 955 044 0<br>Fax: +49 69 955 044 63<br>Email: Global_Intake@otsuka-us.com<br>SAE phone: +49 172 61 44 932 |
| EU-QPPV: | D |
| Version: | Version 11.0 |
| Issue Date: | 7 March 2018 |

## CONFIDENTIAL – PROPRIETARY INFORMATION

This document is a confidential communication of Otsuka. Acceptance of this document constitutes agreement by the recipient that no unpublished information contained herein shall be published or disclosed without prior written approval, except that this document may be disclosed to the appropriate Institutional Review Board(s)/Independent Ethics Committee(s) under the condition that they keep it confidential.

## Signatures of Sponsor Representatives

I have read and agree to the protocol 21-13-102 version 11.0, entitled 'CiloMecT: Effect of Cilostazol as an add-on treatment to a single antiplatelet agent (Acetylsalicylic acid or Clopidogrel) on platelet function testing and bleeding time in healthy volunteers'. I am aware of my responsibilities under the guidelines of Good Clinical Practice, local regulations (as applicable) and the study protocol. I agree to conduct the study according to these guidances.




## **Protocol Synopsis**

| Name of Company:<br>Otsuka Pharmaceuti<br>Name of Investigati<br>Pletal <sup>®</sup> , Cilostazol, | onal Medicinal Product: | Protocol # 21-13-102 |
|---|---|---|
| Protocol Title: CiloMecT: Effect of Cilostazol as an add-on treatment to a single antiplatelet agent (Acetylsalicylic acid or Clopidogrel) or platelet function testing and bleeding time in healthy volunteers | | |
| Clinical Phase: | 1 | |
| Treatment | Healthy subjects | |
| Indication(s): | Cilostazol Mechanistic Trial | |
| Objective(s): | Primary: Trial to investigate | |
| <ul> <li>effects of Cilostazol, Acetylsalycylic acid and<br/>Clopidogrel alone as well as combinations of Cilostazol<br/>Acetylsalicylic acid and Cilostazol/ Clopidogrel on ex-<br/>vivo Platelet Function (PF) testing.</li> </ul> | | |
| • effects on PF in <i>CYP2C19</i> wild-type subjects when compared to subjects identified as carriers of heterozygous or homozygous <i>CYP2C19*2</i> loss-of-function allele(s). | | |
| | [Time Frame: Prior to first dose and after each trial period] | |
| | Secondary: | |
| effects of Cilostazol, Acetylsalycylic acid and<br>Clopidogrel alone as well as combinations of Cilostaz<br>Acetylsalicylic acid and Cilostazol/ Clopidogrel on<br>Bleeding Time (BT). | | |
| | <ul> <li>effects on BT in CYP2C19 wild<br/>compared to subjects identified a<br/>heterozygous or homozygous CY<br/>function allele(s).</li> </ul> | as carriers of |


## • association between PF and BT

Safety variables (vital signs, physical examination, ECG, safety lab, adverse events):

[Time Frame: After first dose and during each trial period]

## Trial Design:

Open-label, single centre, parallel group trial in healthy volunteers. The trial will be conducted at one (1) investigational site in Germany.

After signing screening informed consent approximately 2000 subjects will be screened to evaluate inclusion/ exclusion criteria and to determine subjects *CYP2C19* genotype.

Screening will be performed until:

at least 38 (34 + 4 replacements) subjects with *CYP2C19* wildtype genotype(\*1/\*1) (normal *CYP2C19* activity)

and

at least 19 (17 + 2 replacements) subjects identified as CYP2C19 heterozygous (\*1/\*2) alleles have been screened (intermediate CYP2C19 activity)

and

at least 19 (17 + 2 replacements) subjects identified as CYP2C19 homozygous (\*2/\*2) alleles have been screened (poor CYP2C19 activity).

All determined subjects are required to meet all inclusion and no exclusion criterion.

The *CYP2C19* genotype will be determined by commercially-available technology. The Spartan RX<sup>®</sup> System will be used, allowing determination of the *CYP2C19\*2* phenotype within 60 minutes in the patient's saliva. The assay discriminates between the *CYP2C19* wildtype allele (\*1/\*1, normal *CYP2C19* activity), heterozygous (\*1/\*2, intermediate *CYP2C19* activity) and homozygous (\*2/\*2, poor *CYP2C19* activity) isoforms. The

Spartan RX® *CYP2C19* system is certified in Europe and the testing will be performed by trained investigational site staff.

After signing treatment informed consent 68 subjects will undergo further screening procedures in order to determine baseline characteristics. Subjects failing these procedures will be replaced by screened subjects matching the genotype (normal, intermediate or poor *CYP2C19* activity).

All 68 subjects will then be included in the treatment phase of the trial and will receive during the first week cilostazol 100 mg twice daily for 1 week (trial period A), followed by a 1 week wash-out period (trial period B, return to baseline). Subjects who fail to return to baseline with respect to platelet function testing and bleeding time will be re-tested within a further week.

Thereafter subjects will be stratified and randomized into 4 treatment groups according to their *CYP2C19* genotype (normal or low *CYP2C19* activity).

- Treatment group 1 will consist of CYP2C19 wildtype
   (\*1/\*1) subjects and will receive standard doses of ASA
   100 mg/ day (Group 1, n=17) for 1 week (trial period
   C).
- Treatment group 2 will consist of *CYP2C19 wildtype* (\*1/\*1) subjects and will receive standard doses of clopidogrel 75 mg/ day (Group 2, n=17) for 1 week (trial period C).
- Treatment group 3 will consist of subjects identified as *CYP2C19 heterozygous* (\*1/\*2) subjects and will receive standard doses of clopidogrel 75 mg/ day (Group 3, n=17) for 1 week (trial period C).
- Treatment group 4 will consist of subjects identified as CYP2C19 homozygous (\*2/\*2) subjects and will receive

standard doses of clopidogrel 75 mg/ day (Group 4, n=17) for 1 week (trial period C).

In the following week subjects in all treatment groups will receive 100 mg cilostazol twice daily for 1 week on top as an add-on therapy (trial period D).

## **Subject Population:**

68 healthy male volunteers, 18-45 years.

Approximately 2000 subjects will be screened and their *CYP2C19* genotype will be determined in order to identify at least 19 (17 + 2 replacements) subjects each with *CYP2C19* heterozygous (\*1/\*2) (Group 3) and homozygous (\*2/\*2) isoforms (Group 4), respectively, and at least 38 (34 + 4 replacements) subjects with *CYP2C19* wildtype allele (\*1/\*1) (Group 1+2)

This number of approximately 2000 subjects in screening is based on the published ~30% prevalence of *CYP2C19* heterozygous (\*1/\*2) isoform and 2-5% of the CYP2C19 homozygous (\*2/\*2) isoform in Caucasian population, with frequency of the \*2 genotype in the German population at the lower end of this range.

Sample Size of 17 healthy subjects per treatment arm is based on the following considerations:

The primary variable of the trial is ex-vivo inhibition of platelet aggregation. Comparisons of the inhibition of platelet aggregation are made between subjects during treatment of reference medication alone (Reference) and during the concomitant treatment of reference medication and cilostazol (Test). When assuming that the expected platelet aggregation treatment mean ratio is 1 with a standard deviation of 27% (Angiolillo et al, 2011) <sup>19</sup>, for showing equivalence of a single parameter, a sample size of 17 patients per group would be required to provide a 90% power. That is, with the crossover

| Investigational Medicinal Product, | design, 17 subjects yield a probability of 0.95 to reject the null hypotheses that the platelet aggregation with treatment of cilostazol along with reference medication versus reference medication along is below 0.70 or above 1.43, ie, the 95% confidence interval (CI) is contained within the equivalence limit [0.70,1.43]. Study hypothesis and sample size estimation has been based on the primary end-point platelet aggregation. Similar considerations apply to the assessment of bleeding time which therefore will be treated according to the same principles, however, the estimates for statistical power do not apply for this response variable. Therefore, as well as due to a higher level of intra- as well as interindividual variability and an additional tissue dependent variability bleeding time is evaluated as a key secondary parameter. Cilostazol (Pletal®) 100 mg oral tablets Clopidogrel (Plavix®) 75 mg oral tablets |
|---|---|
| Dose, Formulation,<br>Mode of | Acetylsalicylic Acid (Aspirin® protect) 100 mg oral tablets |
| Administration: | |
| Criteria for<br>Evaluation: | Primary Outcome Variable: Primary efficacy parameters: • Ex-vivo Platelet function: primary parameters to be determined in citrated platelet rich plasma (PRP) by • Light transmission aggregometry (5 µM |
| | ADP, residual aggregation at 5 minutes) Light transmission aggregometry (Arachidonic acid 500 mg/L, residual aggregation at 5 minutes) |
| | Secondary efficacy parameters: • Skin bleeding time: to be determined with Ivy method utilizing standardized bleeding with |

## Surgicutt<sup>®</sup> device

- Ex-vivo Platelet function as determined by
  - Light transmission aggregometry in PRP (20 μM ADP, collagen 1mg/L and 2.5 mg/L, TRAP 25 μM, residual aggregation at 5 minutes)
  - Multiple electrode impedance aggregometry in hirudine-anticoagulated blood (Multiplate®) (ASPItest, ADPtest, ADP/PGEtest, TRAP-test)
  - o VerifyNow<sup>TM</sup> (P2Y12 and Aspirin test)
  - Vasodilator-stimulated phosphoprotein (VASP) by flow cytometry
  - o P-Selectin expression by flow cytometry

Secondary Outcome Variables:

## Safety:

- Vital signs
- Physical examination
- ECG
- Safety lab
- Adverse events

Trial Duration: August 2015 to May 2018

The total study duration for a subject who completes all study procedures will be approximately 120 days at the longest, from the screening visit until End of trial procedures.

## **Table of Contents**

| Sign | atures of Sponsor Representatives | 2 |
|-------|--------------------------------------------------|----|
| Prot | ocol Synopsis | 3 |
| Tabl | le of Contents | 9 |
| List | of In-text Tables | 13 |
| List | of In-text Figures | 14 |
| | of Appendices | |
| | of Abbreviations and Definitions of Terms | |
| 1 | Introduction | |
| 1.1 | Nonclinical Data | |
| 1.2 | Clinical Data | |
| Other | indications (outside Europe) | 25 |
| 1.3 | Pharmacokinetics | 25 |
| 1.3.1 | Cilostazol | 25 |
| 1.3.2 | Clopidogrel | 26 |
| 1.3.3 | Acetylsalicylic Acid (ASA) | 27 |
| 1.4 | Known and Potential Risks and Benefits | 28 |
| 2 | Trial Rationale and Objectives | 28 |
| 2.1 | Trial Rationale | 28 |
| 2.2 | Dosing Rationale | 29 |
| 2.3 | Trial Objectives | 29 |
| 3 | Trial Design | 30 |
| 3.1 | Type/ Design of Trial | 30 |
| 3.2 | Trial Treatments | 32 |
| 3.3 | Trial Population | 34 |
| 3.3.1 | Number of Subjects and Description of Population | 34 |
| 3.3.2 | Subject Selection and Numbering | 34 |
| 3.4 | Eligibility Criteria | 35 |
| 3.4.1 | Informed Consent | 35 |
| 3.4.2 | Inclusion Criteria | 35 |

| 3.4.3 | Exclusion Criteria | 36 |
|---|---|---|
| 3.5 | Primary and Secondary Outcome Variables | 38 |
| 3.5.1 | Primary Outcome Variables | 38 |
| 3.5.2 | Secondary Outcome Variables | 39 |
| 3.6 | Measures to Minimize/ Avoid Bias | 40 |
| 3.7 | Trial Procedures | 40 |
| 3.7.1 | General Inpatient Procedures | 45 |
| 3.7.2 | Dietary Requirements | 45 |
| 3.7.3 | Schedule of Assessments | 45 |
| 3.7.3.1 | Visit 1 (Screening/ Baseline) | 45 |
| 3.7.3.2 | Visit 2 – Trial period A – Day 1 - 7 | 46 |
| 3.7.3.3 | Visit 3 – Trial period B – Day 8 – 14 (21) | 47 |
| 3.7.3.4 | Visit 3 unscheduled – Trial period B – Day 15 - 21 | 47 |
| 3.7.3.5 | Randomization/ Stratification | 48 |
| 3.7.3.6 | Visit 4 – Trial period C – Day 15 – 21 (22 - 28) | 48 |
| 3.7.3.7 | Visit 5 – Trial period D – Day 22 – 29 (29 - 36) | 48 |
| 3.7.3.8 | Time of Withdrawal | 49 |
| 3.7.4 | Safety Assessments | 49 |
| 3.7.4.1 | Clinical Laboratory Tests | 50 |
| 3.7.4.2 | Physical Examination and Vital Sign Assessments | 52 |
| 3.7.4.3 | ECG Assessments | 52 |
| 3.7.5 | End of Trial | 53 |
| 3.8 | Stopping Rules, Withdrawal Criteria and Procedures, and Subject Replacement | 53 |
| 3.8.1 | Entire Trial or Treatment Arm(s) | 53 |
| 3.8.2 | Individual Site | 53 |
| 3.8.3 | Individual Subject | 53 |
| 3.9 | Screen Failures | 54 |
| 3.10 | Definition of Completed Subjects | 54 |
| 3.11 | Subject Compliance | 54 |
| 3.12 | Protocol Deviations | 54 |
| 4 R | lestrictions | 55 |


| 4.1 | Prohibited Medications | 55 |
|---|---|---|
| 5 | Reporting of Adverse Events | 55 |
| 5.1 | Definitions | 55 |
| 5.2 | Eliciting and Reporting Adverse Events | 57 |
| 5.3 | Immediately Reportable Events (IRE) | 58 |
| 5.4 | Potential Hy's Law Cases | 58 |
| 5.5 | Pregnancy | 59 |
| 5.6 | Fathering | 59 |
| 5.7 | Overdose, Misuse, Abuse | 59 |
| 5.8 | Procedure for Breaking the Blind | 60 |
| 5.9 | Follow-up of Adverse Events | 60 |
| 5.9.1 | Follow- up of Adverse Events | 60 |
| 5.9.2 | Follow- up of Post Trial Serious Adverse Events | 60 |
| 5.9.3 | Follow-up and Reporting of Serious Adverse Events Occurring after Last Scheduled Contact | 60 |
| 6 | Pharmacokinetic/ Pharmacodynamic Analysis | 61 |
| 7 | Statistical Analysis | 61 |
| <b>7</b> 7.1 | Sample Size | |
| - | • | 61 |
| 7.1 | Sample Size | 61<br>61 |
| 7.1<br>7.1.1 | Sample Size Sensitivity analysis | 61<br>61 |
| 7.1<br>7.1.1<br>7.2 | Sample Size Sensitivity analysis Analysis of Demographic and Baseline Characteristics | 61<br>61<br>62 |
| 7.1<br>7.1.1<br>7.2<br>7.2.1 | Sample Size | 61<br>62<br>62 |
| 7.1<br>7.1.1<br>7.2<br>7.2.1<br>7.3 | Sample Size Sensitivity analysis Analysis of Demographic and Baseline Characteristics Datasets for Analysis Safety Analysis | 61<br>62<br>62<br>62 |
| 7.1<br>7.1.1<br>7.2<br>7.2.1<br>7.3<br>7.3.1 | Sample Size Sensitivity analysis Analysis of Demographic and Baseline Characteristics Datasets for Analysis Safety Analysis Adverse Events | 61<br>62<br>62<br>62<br>62 |
| 7.1<br>7.1.1<br>7.2<br>7.2.1<br>7.3<br>7.3.1<br>7.3.2 | Sample Size Sensitivity analysis Analysis of Demographic and Baseline Characteristics Datasets for Analysis Safety Analysis Adverse Events Clinical Laboratory Data | 61<br>62<br>62<br>62<br>63 |
| 7.1<br>7.1.1<br>7.2<br>7.2.1<br>7.3<br>7.3.1<br>7.3.2<br>7.3.3 | Sample Size Sensitivity analysis Analysis of Demographic and Baseline Characteristics Datasets for Analysis Safety Analysis Adverse Events Clinical Laboratory Data Physical Examination and Vital Signs Data | 61<br>62<br>62<br>63<br>63 |
| 7.1<br>7.1.1<br>7.2<br>7.2.1<br>7.3<br>7.3.1<br>7.3.2<br>7.3.3<br>7.3.4 | Sample Size Sensitivity analysis Analysis of Demographic and Baseline Characteristics Datasets for Analysis Safety Analysis Adverse Events Clinical Laboratory Data Physical Examination and Vital Signs Data ECG Data | 61<br>62<br>62<br>63<br>63 |
| 7.1<br>7.1.1<br>7.2<br>7.2.1<br>7.3<br>7.3.1<br>7.3.2<br>7.3.3<br>7.3.4<br>7.4 | Sample Size Sensitivity analysis Analysis of Demographic and Baseline Characteristics Datasets for Analysis Safety Analysis Adverse Events Clinical Laboratory Data Physical Examination and Vital Signs Data ECG Data Pharmacokinetic Comparisons | 61<br>62<br>62<br>63<br>63<br>63 |
| 7.1<br>7.1.1<br>7.2<br>7.2.1<br>7.3<br>7.3.1<br>7.3.2<br>7.3.3<br>7.3.4<br>7.4<br>7.5 | Sample Size Sensitivity analysis Analysis of Demographic and Baseline Characteristics Datasets for Analysis Safety Analysis Adverse Events Clinical Laboratory Data Physical Examination and Vital Signs Data ECG Data Pharmacokinetic Comparisons Pharmacodynamic Comparisons | 61<br>62<br>62<br>63<br>63<br>63<br>63 |
| 7.1<br>7.1.1<br>7.2<br>7.2.1<br>7.3<br>7.3.1<br>7.3.2<br>7.3.3<br>7.3.4<br>7.5<br>7.5.1 | Sample Size Sensitivity analysis Analysis of Demographic and Baseline Characteristics Datasets for Analysis Safety Analysis Adverse Events Clinical Laboratory Data Physical Examination and Vital Signs Data ECG Data Pharmacokinetic Comparisons Pharmacodynamic Comparisons Primary analysis | 61<br>62<br>62<br>63<br>63<br>63<br>63 |


| 8.3 | Accountability | 65 |
|-------|----------------------------------------------------|-----------------|
| 8.4 | Returns and Destruction | |
| 8.5 | Reporting of Product Quality Complaints | 66 |
| 8.5.1 | Eliciting and Reporting Product Quality Complaints | |
| 8.5.2 | | |
| 8.5.3 | Return Process | 67 |
| 8.5.4 | Assessment/Evaluation | 67 |
| 9 | Records Management | 67 |
| 9.1 | Source Documents | |
| 9.2 | Data Collection | 68 |
| 9.3 | File Management at the Trial Site | 68 |
| 9.4 | Records Retention at the Trial Site | 69 |
| 10 | Quality Control and Quality Assurance | 69 |
| 10.1 | Monitoring | |
| 10.2 | Auditing | 69 |
| 11 | Ethics and Responsibility | <mark>70</mark> |
| 11.1 | Ethical Conduct of the Trial | 70 |
| 11.2 | Investigator Obligations | 70 |
| 11.3 | Ethics Committee and Competent Authority | 70 |
| 12 | Confidentiality | <mark>71</mark> |
| 13 | Amendment Policy | <mark>71</mark> |
| 14 | References | |

13

| L | ist | of | In-to | ext <sup>-</sup> | Tab | les |
|---|-----|----|-------|------------------|-----|-----|

| Table 3.4.2-1 | Inclusion Criteria | 36 |
|-----------------|----------------------------------|----|
| Table 3.4.3-1 | Exclusion Criteria | 36 |
| Table 3.7-1 | Schedule of Assessments | 42 |
| Table 3.7.4.1-1 | Safety Clinical Laboratory Tests | 50 |

| Protocol | 21 | 1 1 | 12 | 1 ( | 12 |
|----------|----|-----|--------------|-----|----|
| Protocol | | - 1 | ۱ <b>۱</b> – | ı | 1/ |

| List of In-text Figure | Li | st | of | In-te | ext F | Fiaı | ıre | S |
|------------------------|----|----|----|-------|-------|------|-----|---|
|------------------------|----|----|----|-------|-------|------|-----|---|


| List of Appendice |
|-------------------|
|-------------------|

| Appendix 1 | Sponsor Drug Safety Contacts |
|------------|---------------------------------------|
| Appendix 2 | Institutions Concerned with the Trial |
| Appendix 3 | SmPCs7 |

## **List of Abbreviations and Definitions of Terms**

| <b>Abbreviation</b> | <b>Definition</b> |
|---------------------|------------------------------------------------|
| AE | Adverse event |
| AP | Alkaline phosphatase |
| ALT | Alanine transaminase |
| AMG | [Arzneimittelgesetz] German Drug Law |
| AST | Aspartate transaminase |
| BT | (Skin) Bleeding time |
| BUN/ UREA | Blood urea nitrogen |
| CA | Competent Authority |
| CTA | Clinical Trial Application |
| CRF | Case report form |
| EC | Ethics committee |
| ECG | Electrocardiogram |
| FDA | (United States) Food and Drug Administration |
| GCP | Good Clinical Practice |
| GGT | Gamma glutamyl transferase |
| HBsAg | Hepatitis B surface antigen |
| HCV Ab | Hepatitis C antibodies |
| HCT | Haematocrit |
| HGB | Haemoglobine |
| HIV | Human immunodeficiency virus |
| ICH | International Conference on Harmonisation |
| IMP | Investigational medicinal product |
| INR | International normalized ratio |
| IRB | Institutional review board |
| IRE | Immediately reportable event |
| LDH | Lactic dehydrogenase |
| PQC | Product quality complaint |
| PF | Platelet function |
| PRP | Platelet rich plasma |
| PT | Prothrombin time |
| PTT | Partial thromboplastin time |
| RBC | Red blood cell count |
| SAE | Serious adverse event |
| SUSAR | Suspected unexpected serious adverse reactions |
| TEAE | Treatment-emergent adverse event |
| TSH | Thyroid-stimulating hormone |
| WBC | White blood cells |

## 1 Introduction

Cilostazol is an inhibitor of PDE-3 and has several other pharmacological activities that are thought to contribute to its overall benefit in the treatment of Intermittent Claudication (IC). Peripheral arterial disease (PAD) is one presentation of advanced atherosclerosis. PAD patients generally require anti-platelet treatment to reduce their atherothrombotic risk, i.e. the elevated risk of myocardial infarction and stroke. Cilostazol has anti-platelet activity and may add to the effect of e.g. acetylsalicylic acid or clopidogrel which could potentially result in bleeding complications.

Cilostazol alone has not been shown to prolong bleeding time in healthy volunteers and was not associated with increased major haemorrhagic complications in comparison with clopidogrel in a recent stroke prevention trial <sup>1</sup>, as well as in a trial of aspirin and clopidogrel in patients with IC <sup>2</sup>. However, the potential risk for increased bleeding remains.

This trial will provide helpful information towards the understanding of the combined effect of cilostazol and another single antiplatelet agent, and the correlation between bleeding time measurement and platelet function.

#### 1.1 Nonclinical Data

The animal toxicity investigations included single- and repeated-dose toxicity studies. Oncogenicity studies, reproductive and genetic toxicity studies, as well as antigenicity studies and cardiotoxicity studies have been performed.<sup>3 4 5 6 7 8 9 10 11</sup>

| Key safety findings (from non-clinical studies) | Relevance to human usage |
|---|---|
| Toxicity including: | |
| Single and repeat dose toxicity | |
| By virtue of its inhibition of cGMP inhibited | Although compounds of this class |
| cAMP phosphodiesterase (PDE-3), high doses of | may have some potentially |
| cilostazol can be expected to have | undesirable cardiovascular effects at |
| pharmacological effects on the cardiovascular | higher doses than the MRHD, |
| system. The nature and extent of these effects in | including positive inotropy and |
| the species used for repeated-dose toxicity testing | chronotropy, studies conducted on |
| depend on both the level of systemic exposure and | cilostazol have provided clear |


## **Key safety findings (from non-clinical studies)** Relevance to human usage on the intrinsic sensitivity of the target organ. evidence to differentiate it from drugs such as milrinone. Cardiovascular changes were a prominent feature in many of the studies performed in dogs. Long-term exposure to cilostazol in Treatment-related microscopic changes were human also in controlled clinical found in the heart and coronary vessels of dogs in trials indicated that cilostazol did not the pivotal oral toxicity studies. The most frequent increase cardiac risks in the targeted lesions were recent or old endocardial IC population in comparison with placebo. haemorrhages in the left ventricle ('jet lesions'), right atrial lesions and arteriopathy in the coronary vessels ranging from simple intimal However, because of the proliferation to coronary arteritis. chronotropic and dromotropic Comparable haemorrhagic lesions were recorded effects of cilostazol, arrhythmic in the cynomolgus monkey heart but, in contrast events are expected to occur in to the dog, no coronary arteritis or periarteritis association with administration of was found in male cynomolgus monkeys given cilostazol and accordingly cardiac daily oral doses of cilostazol at 300, 900 or arrhythmic events including 1800 mg/kg/day for 13 weeks or daily i.v. doses palpitation, tachycardia etc. are of 3, 5 or 10 mg/kg/day for one week. identified as safety concerns and Establishing NOAEL levels for coronary artery stated in the CCSI/SmPC. lesions is difficult because of spontaneous background pathology, but in summary: 5-week oral: treatment-related endocardial and arterial lesions at 750 mg/kg/day, NOAEL 150 mg/kg/day. 13-week oral: treatment-related endocardial ('jet') and arterial lesions at 150 and 750 mg/kg/day, NOAEL 30 mg/kg/day. 52-week oral: endocardial ('jet') lesions at 30 and 150 mg/kg/day, NOAEL 12 mg/kg/day. No clear treatment-related arterial lesions, but a minor increase of spontaneous intimal thickening and coronary arteritis.

Hence, the various lesions of the heart in dogs are

| Key safety findings (from non-clinical studies) | Relevance to human usage |
|---|---|
| only seen at dosages of 30 mg/kg/day and above | |
| in the 52-week trial. Cardiac lesions were not | |
| observed when cilostazol was administered to | |
| dogs for 5 weeks at a dose of 150 mg/kg/day | |
| (approximately 24 times the Maximum | |
| Recommended Human Dose (MRHD) on a | |
| mg/m2 basis), for 13 weeks at a dose of 30 | |
| mg/kg/day (approximately 4.9 times the MRHD | |
| on a mg/m2 basis) or for 52 weeks at a dose of 12 | |
| mg/kg/day (approximately twice the MRHD on a | |
| mg/m2 basis). | |
| Such lesions were not seen in rats or monkeys and | |
| are considered species specific. | |
| Investigation of QTc in dogs and monkeys | |
| showed no prolongation after administration of | |
| cilostazol or its metabolites.31 | |
| Reproductive toxicity | |
| Body weight in the females treated at 150 | Cilostazol may be used in women of |
| mg/kg/day and above (1000 mg/kg/day) tended to | child-bearing potential provided |
| be higher during treatment in the gestation period. | adequate contraception is practiced |
| Cilostazol did not cause any changes in the | in order to prevent inadvertent |
| reproductive performance of male or female | pregnancy due to the reported |
| animals or in the foetal development. | developmental toxicity in seen in |
| Dosages of 30, 150 and 1,000 mg/kg/day | rats. |
| administered orally were investigated in pregnant | As no adequate data are available, |
| female rats and offspring. The transfer of | cilostazol must not be used during |
| cilostazol to breast milk has been observed in | pregnancy. It is not recommended to |
| animal studies. | use cilostazol during breast feeding. |
| Cilostazol did not alter fertility in animal studies. | |
| Developmental toxicity | |
| Dosages of 30, 150 and 1,000 mg/kg/day | As no adequate data are available, |


| Key safety findings (from non-clinical studies) | Relevance to human usage |
|---|---|
| administered orally were investigated in pregnant | cilostazol must not be used during |
| female rats and offspring. It was observed that | pregnancy. It is not recommended to |
| foetal weight was decreased; and there were an | use cilostazol during breast feeding. |
| increased number of external, visceral and | |
| skeletal abnormalities in foetuses from dams | |
| treated at 1,000 mg/kg/day. Retardation of | |
| ossification was seen in foetuses from dams | |
| treated at 150 mg/kg/day. | |
| • Nephrotoxicity | |
| Cilostazol may produce morphological changes in | No relevance to human usage |
| the kidney of SD rats at 1500 mg/kg/day by | |
| gavage. A clear cut NOAEL was not established | |
| for increased progressive nephropathy when | |
| cilostazol was administered to F344 rats by the | |
| dietary route for 2 years at dose levels of 50-500 | |
| mg/kg/day. As no renal effects were seen in other | |
| species, there is little or no risk to man at | |
| therapeutic dose levels. | |
| Hepatotoxicity | |
| The liver weight was increased at all dose levels | No relevance to human usage |
| and associated microscopically with dose-related | |
| hepatocytic hypertrophy. A NOAEL was not | |
| established for most of these findings, which were | |
| mainly physiological adaptive changes of no | |
| toxicological significance to humans at the | |
| intended therapeutic dose levels. | |
| • Genotoxicity | |
| A series of studies were conducted to evaluate the | No relevance to human usage |
| genotoxic potential of cilostazol. Genotoxic | |
| potential was evaluated in mutation and | |
| chromosome aberration test systems. In addition, | |
| cilostazol's DNA damaging potential was | |
| evaluated in bacterial DNA repair and SOS | |


| Key safety findings (from non-clinical studies) | Relevance to human usage |
|---|---|
| induction test systems. These mutagenic tests showed no mutation or DNA damage. Cilostazol produced a weak but significant increase in chromosome aberration frequency at 140 p g/mL and higher in an in vitro CHO cell assay. However, cilostazol did not produce chromosome aberration in an in vivo mouse (BDF, male) bone marrow aberration assay at 6000 mg/kg. | |
| Carcinogenicity | |
| There were no increased tumour incidences in rats and mice. Although there were higher incidences of adrenal medullary tumours in F344 rats and liver tumours in B6C3F1 mice, it was concluded that these findings were non-specific rather than drug related responses. There were no unusual neoplastic outcomes in the 2-year rat and mouse bioassays to indicate any potential carcinogenic risk to humans at the intended therapeutic dose levels. In addition there were no unusual findings suggestive of any unexpected target organ toxicity due to repeated administration of cilostazol to laboratory animals. | No clinical significance. |
| General safety pharmacology: | |
| Cardiovascular (including potential for QT interval prolongation) | |
| The cardiovascular pharmacology studies in dogs indicated significant decreases in blood pressure and increases in heart rate at doses of 30 and 100 mg/kg. Cardiac lesions have been observed in a 52-week toxicity trial with dogs in doses of 30 mg/kg/day | Although compounds of this class may have some potentially undesirable cardiovascular effects at higher doses than the MRHD, including positive inotropy and chronotropy, studies conducted on cilostazol have provided clear |

## **Key safety findings (from non-clinical studies)**

and above (approximately 4.9 times the Maximum Recommended Human Dose (MRHD) on a mg/m2 basis).

Cardiac lesions could not be observed when cilostazol was administered to dogs

for 5 weeks at a dose of 150 mg/kg/day (approximately 24 times the MRHD on a mg/m2 basis),

for 13 weeks at a dose of 30 mg/kg/day (approximately 4.9 times the MRHD on a mg/m2 basis) or

for 52 weeks at a dose of 12 mg/kg/day (approximately twice the MRHD on a mg/m2 basis) (Dossier Module 2.4.6).



Hence, cardiac lesions were only observed with 30 mg/kg/day when cilostazol was administered for a longer period (52 weeks) - grey shaded in picture above - but not for a shorter period (13 weeks); subsequently, higher doses of cilostazol (150 mg/kg/day) but shorter administration periods (5 weeks) did not lead to cardiac lesions.

Such lesions were not seen in rats or monkeys and are considered species specific.

Investigation of QTc in dogs and monkeys

#### Relevance to human usage

evidence to differentiate it from drugs such as milrinone.

Long-term exposure to cilostazol in human also in controlled clinical trials indicated that cilostazol did not increase cardiac risks in the targeted IC population in comparison with placebo.

However, because of the chronotropic and dromotropic effects of cilostazol, arrhythmic events are expected to occur in association with administration of cilostazol and accordingly cardiac arrhythmic events including palpitation, tachycardia etc. are identified as safety concerns and stated in the CCSI/SmPC.

| Key safety findings (from non-clinical studies) | Relevance to human usage |
|-------------------------------------------------|--------------------------|
| showed no prolongation after administration of | |
| cilostazol or its metabolites. | |

Available non-clinical data provide adequate non-clinical evidence for the use of cilostazol in the indicated population; given the extensive clinical and post-marketing experience, no additional non-clinical data are proposed for investigation of possible effects in special populations at this time.

## 1.2 Clinical Data

In Europe, cilostazol-containing medicinal products are indicated for the improvement of the maximal and pain-free walking distances in patients with IC, who do not have rest pain and who do not have evidence of peripheral tissue necrosis (peripheral arterial disease Fontaine stage II).

Cilostazol-containing medicinal products are for second-line use, in patients in whom lifestyle modifications (including stopping smoking and [supervised] exercise programs) and other appropriate interventions have failed to sufficiently improve their intermittent claudication symptoms.

A total of 14 clinical trials were performed enrolling more than 4,000 IC patients, including 8 double-blind, controlled Phase III trials. All Phase III trials included treatment arms with the approved dose of cilostazol 100 mg bid and placebo; two of the 8 trials had an additional arm of 50 mg cilostazol bid and one trial an arm with 150 mg bid. Two Phase III trials compared efficacy of cilostazol to standard therapy (pentoxifylline) and placebo over a period of 24 weeks.

After the approval in the US in 1999 and in the UK in 2000, two further trials were initiated. In August 1999, the PACE trial, a double-blind, placebo-controlled Phase IV trial with pentoxifylline as active comparator was initiated to corroborate efficacy data of previous trials. Secondly, in March 2001, the CASTLE trial, a double-blind, placebo-controlled Phase IV trial, was initiated in the US to evaluate safety in long-term treatment of the IC population. At the time when cilostazol was approved in the US and UK, no long-term controlled safety data were available except post-authorisation data from Japan, where cilostazol had been marketed since 1988.

In 9 efficacy trials (8 Phase III trials, plus the phase IV PACE trial) a total of 3,482 patients were randomised and received at least one dose of the investigational product.

The safety dataset of the original European MAA in 2000 was derived from 8 placebo-controlled Phase III (7 in the USA, 1 in UK) trials, all including treatment arms of the approved dose cilostazol 100 mg bid. Similarities can be seen in the trial population, trial design and duration of treatment between these 8 Phase III trials and a Phase IV trial, PACE (21-98-213). In August 1999, the PACE trial, a double-blind, placebo-controlled Phase IV trial with pentoxifylline as active comparator was initiated to corroborate efficacy data of previous trials. <sup>12</sup>

These trials are hereinafter referred to as "mid-term trials" (treatment duration between 12 and 24 weeks). Another Phase IV placebo controlled trial (CASTLE) was designed to compare long-term treatment of cilostazol with placebo for the same IC population with regard to all-cause mortality; the trial design and duration of exposure were different. This trial is hereinafter referred to as a "long-term trial" (duration up to three years).

The CASTLE trial was conducted to evaluate the long-term effects of cilostazol and was intended primarily to provide an estimate of the relative risk of death in patients taking cilostazol versus placebo with long-term use. 13 The primary outcome variable in this trial was a time-to-event variable where the event of interest was death due to any cause. Due to a low mortality rate with a relatively high drop-out rate, feasibility of completion of the trial had been evaluated. CASTLE was terminated after 3 years trial duration and before reaching the originally intended number of events. At that time 1,899 patients had been screened, and a total of 1,435 patients (the original targeted number) had been randomised to treatment with either cilostazol or placebo. The decision to prematurely terminate the trial was made under blinded conditions and in agreement with the FDA. The available data from the trial provides an extensive data base for understanding the long-term risk for treatment with cilostazol. Neither the statistical integrity nor the double-blind status was broken through the whole trial period and the conclusion from this trial remains unbiased and fully interpretable. CASTLE trial provides extensive, valid data on the safety of cilostazol and demonstrates no evidence of increased mortality associated with the long-term use of cilostazol.

25

## Other indications (outside Europe)

In regions outside Europe, cilostazol has been developed for additional indication other than IC, e.g. cilostazol is approved in Japan for the recurrence of stroke.

From the clinical development program for this indication the two main studies are listed below:

CSPS I: The objective of trial CSPS I was to assess the long-term safety and efficacy of cilostazol in preventing recurrence of cerebral infarction in patients who had suffered a cerebral infarction 1 to 6 months prior to entering the trial.

Trial CSPS I was started in April 1991 and for each patient enrolled from this point onward trial medication was to be continued for as long as possible until the final day of the trial (31 Mar 1997).

CSPS II: The Japanese trial CSPS II compared cilostazol (200 mg/day) with Aspirin<sup>®</sup> (81 mg/day) in patients receiving treatment for secondary prevention of stroke. All patients had a medical history of cerebral infarction. A total of 1,356 patients in the cilostazol and 1,360 patients in the Aspirin<sup>®</sup> group received trial medication. Patients were on treatment for varying durations until the date of the overall trial completion. Those who were on medication at the time of trial completion were observed until a 38-day follow-up visit after stopping of trial medication.

Other indication under investigation or development (e.g. the drug was also investigated in the indications of juvenile primary and secondary Raynaud's phenomenon in paediatric population) play a minor role in the overall development program and are not described in detail.

#### 1.3 Pharmacokinetics

#### 1.3.1 Cilostazol

Cilostazol is absorbed after oral administration. A high fat meal increases absorption, with an approximately 90% increase in  $C_{max}$  and a 25% increase in AUC. Absolute bioavailability is not known. Cilostazol is extensively metabolized by hepatic cytochrome P-450 enzymes, mainly 3A4, and to a lesser extent, 2C19, with metabolites largely excreted in urine. Two metabolites are active, with one metabolite appearing to account for at least 50% of the pharmacologic (PDE III inhibition) activity after administration of

cilostazol. Pharmacokinetics are approximately dose proportional. Cilostazol and its active metabolites have apparent elimination half-lives of about 11-13 hours. Cilostazol and its active metabolites accumulate about 2-fold with chronic administration and reach steady state blood levels within a few days. The pharmacokinetics of cilostazol and its two major active metabolites were similar in healthy subjects and patients with intermittent claudication due to peripheral arterial disease (PAD).

## 1.3.2 Clopidogrel

After single and repeated oral doses of 75 mg per day, clopidogrel is rapidly absorbed. Mean peak plasma levels of unchanged clopidogrel (approximately 2.2 - 2.5 ng/ ml after a single 75 mg oral dose) occurred approximately 45 minutes after dosing. Absorption is at least 50%, based on urinary excretion of clopidogrel metabolites.

Clopidogrel is extensively metabolised by the liver. In vivo, clopidogrel is metabolised according to two main metabolic pathways: one mediated by esterases and leading to hydrolysis into its inactive carboxylic acid derivative (85% of circulating metabolites), and one mediated by multiple cytochromes P450 with formation of the active metabolite exerting antiplatelet effects. Clopidogrel is first metabolised to a 2-oxo-clopidogrel intermediate metabolite. Subsequent metabolism of the 2-oxo-clopidogrel intermediate metabolite results in formation of the active metabolite, a thiol derivative of clopidogrel. In vitro experiments with incubation of clopidogrel and either liver microsomes or isolated cytochrome P450 enzymes indicate that this metabolic pathway is mediated by *CYP3A4*, *CYP2C19*, *CYP1A2* and *CYP2B6*. The active thiol metabolite which has been isolated in vitro, binds rapidly and irreversibly to platelet P2Y<sub>12</sub> receptors, thus inhibiting platelet aggregation. The C<sub>max</sub> of the active metabolite is twice as high following a single 300-mg clopidogrel loading dose as it is after four days of 75-mg maintenance dose. C<sub>max</sub> occurs approximately 30 to 60 minutes after dosing.

CYP2C19 is involved in the formation of both the active metabolite and the 2-oxoclopidogrel intermediate metabolite. Clopidogrel active metabolite pharmacokinetics and antiplatelet effects, as measured by ex vivo platelet aggregation assays, differ according to CYP2C19 genotype. The CYP2C19\*1 allele corresponds to fully functional metabolism while the CYP2C19\*2 and CYP2C19\*3 alleles are nonfunctional. The CYP2C19\*2 and CYP2C19\*3 alleles account for the majority of reduced function alleles

in the Caucasian (85%) and the Asian (99%) population and are the major reason for genetically fixed clopidogrel "resistance" <sup>14</sup>.

Other alleles associated with absent or reduced metabolism are less frequent and include *CYP2C19\*4*, \*5, \*6, \*7, and \*8. A patient with poor metaboliser status will carry two loss-of-function alleles as defined above. Published frequencies for the poor *CYP2C19* metaboliser genotypes are approximately 2% for Caucasians, 4% for Blacks and 14% for Chinese.

In addition to the alleles associated with impaired CYP2C19 function the *CYP2C19\*17* allele exists, which is associated with ultra-rapid metabolizer phenotypes due to an increased gene expression. The *CYP2C19\*17* allele is found in approximately 21% of Caucasians, 27% of Africans and less than 2% of Asians. Some studies indicate that this allele results in enhanced platelet inhibition and clopidogrel response<sup>15,16</sup>.

Tests are available to determine a patient's CYP2C19 genotype.

## 1.3.3 Acetylsalicylic Acid (ASA)

Following oral administration, absorption of non-ionised aspirin occurs mainly in the upper intestine. Some aspirin is hydrolysed to salicylate in the gut wall. After absorption aspirin is rapidly converted to salicylate but during the first twenty minutes following oral administration, aspirin is the predominant form of the drug in the plasma. Aspirin is bound to plasma proteins and is widely distributed. Plasma-aspirin concentrations decline rapidly (half-life 15-20 minutes) as plasma salicylate concentrations increase. Salicylates are extensively bound to plasma proteins and are rapidly distributed to all body parts. Salicylates appear in breast milk and cross the placenta. Salicylate is mainly eliminated by renal excretion in form of glucuronidated or free salicylic acid metabolites. Following a 100 mg aspirin dose, elimination is a first-order process and the serum-salicylate half-life is about two to three hours; at high aspirin doses, the half-life increases to fifteen to thirty hours. Salicylate is also excreted unchanged in the urine; the amount excreted by this route increases with increasing dose and also depends on urinary pH, about 30% of a dose being excreted in alkaline urine compared with 2% of a dose in acidic urine.

Similar to clopidogrel, the antiplatelet effect of aspirin is also irreversible and apparently complete after about 3 days administration of 100 mg/ day orally.

## 1.4 Known and Potential Risks and Benefits

This is a clinical trial in healthy volunteers and in consequence no therapeutic benefit can be expected.

Potential risks of Cilostazol, Clopidogrel or Acetylsalicylic Acid are described in the currently approved versions of the Summary of Product Characteristics (SmPC) and are filed as Appendices to this trial protocol.

## 2 Trial Rationale and Objectives

## 2.1 Trial Rationale

Platelets contribute to the pathogenesis of a variety of different vascular syndromes, including myocardial infarction, ischemic stroke and peripheral artery disease. Antiplatelet therapy is commonly used for the prevention of these events. The current therapeutic strategies for inhibiting platelets include the inhibition of phosphodiesterase III (e.g. by Cilostazol), inhibition of cyclooxygenase (e.g. by ASA) or blockage of the platelet P2Y12 receptor (e.g. by Clopidogrel).

Due to their different mechanisms of action, a dual combination is likely to have an additive effect and therefore can result in a more effective way to reduce vascular events. However, dual therapy can also pose the risk of excess bleeding.

The aim of this trial is to evaluate and compare the effects on platelet function and skin bleeding time during the administration of Cilostazol, ASA or Clopidogrel alone or in combination of ASA/ Cilostazol or Clopidogrel/ Cilostazol in healthy subjects.

In addition, loss-of-function mutations in the hepatic cytochrome P450 *CYP2C19* gene have been shown repeatedly to have an important influence on the responses to Clopidogrel. <sup>14 17 18</sup>

Although Cilostazol is mainly converted into the active metabolite by the hepatic cytochrome *CYP3A4* system, platelet inhibition by adjunctive cilostazol intake is also expected to be influenced to a lesser extent by the *CYP2C19* loss-of-function variants, which is present in about 30 % of the Caucasians. To evaluate the impact of the heterozygous or homozygous loss-of-function alleles on the effect of bleeding time after administration of Cilostazol alone or in combination of Cilostazol and Clopidogrel,

subjects will be screened for their respective genotype prior to enrolment. Stratification into three groups will be done for those subjects receiving the combination of Cilostazol and Clopidogrel: one sub-group will consist of subjects carrying the wildtype alleles of *CYP2C19* (\*1/\*1) - (normal *CYP2C19* activity), the second sub-group will consist of subjects carrying the heterozygous (\*1/\*2) isoform (intermediate *CYP2C19* activity) and the third group the homozygous (\*2/\*2) isoform (poor *CYP2C19* activity).

This setting will allow us to evaluate the impact of the respective genotypes on platelet function and bleeding time after administration of Cilostazol alone or in combination of Cilostazol and Clopidogrel.

## 2.2 Dosing Rationale

Dosing, dosage form and dosing regimen for Cilostazol, ASA and Clopidogrel will be done according to the recommendations laid down in the SmPCs for each drug.

## 2.3 Trial Objectives

The primary objective of this trial is to determine the effects of orally administered Cilostazol 100 mg twice daily, Acetylsalicylic acid 100 mg once daily or Clopidogrel 75mg once daily alone as well as in combination of Cilostazol 100 mg twice daily/ Clopidogrel 75 mg once daily or Cilostazol 100 mg twice daily/ Acetylsalicylic acid 100 mg once daily on ex-vivo platelet function testing.

A key secondary objective is the effect of orally administered Cilostazol 100 mg twice daily, Acetylsalicylic acid 100 mg once daily or Clopidogrel 75mg once daily alone as well as in combination of Cilostazol 100 mg twice daily/ Clopidogrel 75 mg once daily or Cilostazol 100 mg twice daily/ Acetylsalicylic acid 100 mg once daily on bleeding time in healthy subjects. While bleeding time is an important parameter in this regard it also does exhibit a higher level of intra- as well as interindividual variability and an additional tissue dependent variability. Therefore, bleeding time is evaluated as a key secondary parameter.

In addition, the effects of a combined administration of Cilostazol 100 mg twice daily/ Clopidogrel 75 mg once daily in subjects with a homozygous wildtype allele of CYP2C19 (\*1/\*1) showing normal CYP2C19 activity will be compared with the effects of subjects carrying either the heterozygous CYP2C19 (\*1/\*2) isoform and with subjects carrying the homozygous CYP2C19 (\*2/\*2) isoforms, displaying a intermediate and poor CYP2C19 activity, respectively.

A further secondary objective is to assess the safety variables after the orally administration of Cilostazol 100 mg twice daily, Acetylsalicylic acid 100 mg once daily or Clopidogrel 75 mg once daily alone as well as a combination of Cilostazol 100mg twice daily/ Clopidogrel 75mg once daily or Cilostazol 100mg twice daily/ Acetylsalicylic acid 100 mg once daily.

## 3 Trial Design

## 3.1 Type/ Design of Trial

An Open-label, single centre, parallel group trial in healthy volunteers.

The trial will be conducted at one (1) investigational site in Germany.



Figure 3.1-1 Trial Design Schematic

#### 3.2 Trial Treatments

After signing screening informed consent, approximately 2000 subjects will be screened to evaluate inclusion/exclusion criteria and to determine subjects CYP2C19 genotype.

Screening will be performed until:

at least 38 (34+ 4 = replacements) subjects with CYP2C19 wildtype allele (\*1/\*1) (normal CYP2C19 activity)

and

at least 19 (17+2 = replacements) subjects with CYP2C19 heterozygous (\*1/\*2) isoform (intermediate CYP2C19 activity)

and

at least 19 (17+2 = replacements) subjects with CYP2C19 homozygous (\*2/\*2) isoform (poor CYP2C19 activity) have been identified and screened.

For the purpose of statistical analyses 34 evaluable subjects with normal *CYP2C19* activity, 17 evaluable subjects with intermediate and 17 evaluable subjects with low *CYP2C19* activity, respectively, are required. Subjects who will be considered not evaluable during course of the trial (e.g. early termination, protocol violators) will be replaced. Any replacement subjects must begin the trial at the start of the protocol.

The stated number of replacements for the individual study groups are estimates and may become higher in the case that data of unexpectedly high numbers of subjects are found to be of not evaluable in the course of the study.

All subjects suitable for enrolment/randomization are required to meet all inclusion criteria and no exclusion criterion.

The *CYP2C19* genotype will be determined by commercially-available technology. The Spartan RX<sup>®</sup> System will be used, allowing determination of the *CYP2C19* phenotype within 60 minutes in the patient's saliva. The assay allows to discriminate between the *CYP2C19 wildtype allele (\*1/\*1*, normal *CYP2C19* activity), *heterozygous (\*1/\*2*, low *CYP2C19* activity) and *homozygous (\*2/\*2*, low *CYP2C19* activity) alleles.

The assay directly detects the *CYP2C19\*2*, \*3, and \*17 alleles. Besides the \*1 allele these are the alleles with the highest frequency in Caucasian populations. The system reports for each allele whether none, one or two copies of it are detected. Detection of one or two \*2 alleles, for example, allows to determine whether the test subject has a *CYP2C19\*1/\*2* or *CYP2C19\*2/\*2* genotype. If no copy of the \*2, \*3 or \*17 alleles is detected it can be concluded that the test subject has a \*1/\*1 genotype.

The Spartan RX<sup>®</sup> *CYP2C19* system is certified in Europe and the testing will be performed by trained investigational site staff.

After signing treatment informed consent, 68 subjects will undergo further screening procedures in order to determine baseline characteristics. Subjects failing these procedures will be replaced by screened subjects matching the genotype (normal, intermediate or poor *CYP2C19* activity).

All 68 subjects will then be included in the treatment phase of the trial and will receive during the first week cilostazol 100 mg twice daily for 1 week (trial period A), followed by a 1 week wash-out period (trial period B, return to baseline). Subjects who fail to return to baseline with respect to platelet function testing and skin bleeding time will be re-tested within a further week.

Thereafter subjects will be stratified and randomized into 4 treatment groups according to their *CYP2C19* genotype (normal or low *CYP2C19* activity).

- Treatment group 1 will consist of subjects with CYP2C19 wildtype allele (\*1/\*1) and will receive standard doses of ASA 100 mg/ day (Group 1, n=17) for 1 week (trial period C).
- Treatment group 2 will consist of subjects with CYP2C19 wildtype allele (\*1/\*1) and will receive standard doses of clopidogrel 75 mg/ day (Group 2, n=17) for 1 week (trial period C).
- Treatment group 3 will consist of subjects with *CYP2C19 heterozygous* (\*1/\*2) isoform and will receive standard doses of clopidogrel 75 mg/ day (Group 3, n=17) for 1 week (trial period C).
- Treatment group 4 will consist of subjects with *CYP2C19 homozygous* (\*2/\*2) isoform and will receive standard doses of clopidogrel 75 mg/ day (Group 3, n=17) for 1 week (trial period C).

In the following week subjects in all treatment groups will receive 100 mg cilostazol twice daily for 1 week on top as an add-on therapy (trial period D).

Drug intake of ASA and clopidogrel will be in the morning hours, for cilostazol drug intake will be twice daily: once in the morning and once in the evening.

## 3.3 Trial Population

## 3.3.1 Number of Subjects and Description of Population

Approximately 2000 subjects will be screened and their *CYP2C19* genotype will be determined in order to identify at least 17 + 2 subjects with *CYP2C19 heterozygous* (\*1/\*2) isoform (Group 3) and 17 + 2 subjects with *CYP2C19 homozygous* (\*2/\*2) isoforms (Group 4) and at least 34 + 4 subjects with *CYP2C19 wildtype allele* (\*1/\*1) (Group 1+2)

This number of approximately 2000 subjects in screening is based on the published  $\sim$ 30% prevalence of *CYP2C19 heterozygous* (\*1/\*2) and 2-5% of *CYP2C19 homozygous* (\*2/\*2) isoforms in the Caucasian population and under consideration of the fact that the \*2 isoform is closer to the lower end of probability in the German population.

A total of 68 healthy male volunteers, aged 18-45 years, will be dosed with trial medication and complete all trial procedures and periods. Trial participants who will early terminate their trial participation will be replaced. If the scheduled evaluation of the primary efficacy parameter (outlined in Section 3.5.1) cannot be performed (e.g. for technical reasons), additional subjects may be enrolled at the sponsor's discretion in agreement with the principal investigator. Any replacement subjects must begin the trial at the start of the protocol.

## 3.3.2 Subject Selection and Numbering

The investigational site will identify potential trial participants and perform screening procedures. Screened subjects will be assigned a unique identification number. The investigational site will maintain a confidential list identifying all subjects.
# 3.4 Eligibility Criteria

#### 3.4.1 Informed Consent

Written informed consent will be obtained from all subjects. Consent will be documented on a written informed consent form (ICF). The ICF will be approved by the same ethics committee (EC) that approves this protocol. Each ICF will comply with the EU Clinical Trials Directive (2001/20/EC), FDA regulations in 21 CFR Part 50, ICH Good Clinical Practice (GCP) Guideline and local regulatory requirements. The investigator agrees to obtain sponsor approval of any written ICF used in the trial, prior to submission to the EC.

Investigators may discuss trial availability and the possibility for entry with a potential subject without first obtaining consent. However, informed consent must be obtained and documented prior to initiation of any procedures that are performed solely for the purpose of determining eligibility.

Once appropriate essential information has been provided and fully explained in layman's language to the subject by the investigator (or a qualified designee), two versions of the EC -approved written ICF will be signed and dated by both the subject and the person obtaining consent (investigator or designee). The subject will receive one version of the signed ICF; the other version shall be kept on confidential file by the investigator.

## 3.4.2 Inclusion Criteria

Subjects are required to meet the following inclusion criteria:

36

#### Table 3.4.2-1 Inclusion Criteria

- 1. Healthy Caucasian male subjects
- 2. Aged 18 to 45 years, inclusive
- 3. Able to read, to write and to fully understand German language
- 4. Provision of written informed consent before screening and baseline
- 5. BMI between 19.0 and 30.0 kg/m<sup>2</sup>, inclusive and body weight between 50.0 and 100.0 kg, inclusive
- 6. Good general health as determined by the investigator by medical history, physical examination, vital signs, electrocardiogram, baseline and safety lab

#### 3.4.3 Exclusion Criteria

Subjects will be excluded if they meet any of the following exclusion criteria:

#### Table 3.4.3-1 Exclusion Criteria

- 1. Personal or family history of bleeding disorders, or reasonable suspicion of vascular malformations, including aneurysms
- 2. Known predisposition to bleeding (e.g. active peptic ulceration, recent (within 6 month prior to screening) haemorrhagic stroke, proliferative diabetic retinopathy, poorly controlled hypertension)
- 3. Participation in a clinical investigation within the last thirty (30) days prior to screening or during this trial
- 4. Acute illness, surgical procedure or trauma from thirty (30) days before screening and until baseline visit
- 5. Use of antibiotics within thirty (30) days prior to baseline visit
- 6. Clinically significant abnormalities in medical history, physical examination, vital signs, electrocardiogram, baseline and safety lab
- 7. History of severe tachyarrhythmia (of any type)
- 8. Unstable angina, myocardial infarction within the last 6 months prior to screening or a coronary intervention within the last 6 months prior to screening
- 9. Positive results in HIV, HBV and HCV tests during baseline
- 10. Positive drug screen during baseline

- 11. Smokers
- 12. Supine pulse rate > 100 beats/min or <50 beats/min
- 13. Systolic blood pressure <100 or >140 mmHg
- 14. Diastolic blood pressure <50 or >90 mmHg
- 15. Prolongation of QTc interval > 450 ms
- Known impaired glucose tolerance, known galactose intolerance, total lactase deficiency or glucose-galactose malabsorption or known or suspected Gilbert's syndrome
- 17. Clinically relevant allergy (except for untreated, asymptomatic, seasonal allergies at time of dosing) drug hypersensitivity
- 18. Known hypersensitivity to one of the IMP substances
- 19. Severe digestive disorder or surgery of the digestive tract (except for appendectomy)
- 20. Clinically relevant renal disorders
- 21. Clinically relevant hepatic disorders
- 22. Clinically relevant respiratory disorders
- 23. Clinically relevant cardiovascular disorders, especially any history of ventricular tachycardia, ventricular fibrillation or multifocal ventricular ectopics, or a history of additional risk factors for torsades de pointes (TdP) (e.g. heart failure, hypokalaemia, congenital long QT-syndrome)
- 24. Thyroid dysfunction or other endocrine disorders
- 25. Malignancy
- 26. Substance abuse or addiction (alcohol, illicit drugs) in the past 3 years
- 27. Neurologic or psychiatric illness
- 28. Concomitant use of any other medication including over-the-counter preparations
- 29. Consumption of more than 600 mg of caffeine/day (1 cup of coffee contains approximately 100 mg of caffeine, 1 cup of tea approximately 30 mg and 1 glass of coke approximately 20 mg)
- 30. Consumption of more than 40 g of alcohol/day (amount corresponds to 1 l of beer/day or 0.5 l of wine/day or 6 glasses (à 2 cl) of liquor/day
- 31. A diet which deviates notably from the "normal" amounts of protein, carbohydrate and fat, as judged by the investigator (e.g. vegetarians)
- 32. Donation of blood, plasma or platelets within ninety (90) days prior to baseline visit, or

planned donation of blood, plasma or platelets during trial participation or within ninety (90) days after trial completion

Subjects excluded for positive drug/ alcohol/ infections screen at baseline are not eligible to be re-screened for participation in the trial.

However subjects excluded for any other reasons may be re-screened at a later stage if the individual exclusion characteristic has changed.

In the event that the subject is re-screened, a new ICF must be signed and a new screening number needs to be assigned. All screening procedures need to be repeated with the exemption of Genotyping.

# 3.5 Primary and Secondary Outcome Variables

## 3.5.1 Primary Outcome Variables

Primary efficacy parameters:

- Ex-vivo Platelet function: primary parameters to be determined in citrated platelet rich plasma (PRP) by
  - Light transmission aggregometry (5 μM ADP, residual aggregation at 5 minutes)
  - Light transmission aggregometry (Arachidonic acid 500 mg/L, residual aggregation at 5 minutes)

Primary efficacy parameter (PFT) will be tested at trough (i.e. 24 hours after last administration of ASA/ clopidogrel, 12 hours after last administration of cilostazol) in the morning hours after 7 days treatment (i.e. on the 1st day of the next study period) and prior to intake of next study medication. Appropriate controls will be performed in accordance with the instructions provided by the manufacturers of test equipment each time any of the platelet tests is run.

Secondary efficacy parameters:

 Skin bleeding time: to be determined with Ivy method utilizing standardized bleeding with Surgicutt<sup>®</sup> device


- Ex-vivo Platelet function as determined by
  - Light transmission aggregometry in PRP (20 μM ADP, collagen
     1mg/L and 2.5 mg/L, TRAP 25 μM residual aggregation at 5 minutes)
  - Multiple electrode impedance aggregometry in hirudineanticoagulated blood (Multiplate®) (ASPItest, ADPtest, ADP/PGEtest, TRAP-test)
  - VerifyNowTM (P2Y12 and Aspirin test)
  - o Vasodilator-stimulated phosphoprotein (VASP) by flow cytometry
  - o P-Selectin expression by flow cytometry

Secondary efficacy parameters (BT and PFT) will be tested at trough (i.e. 24 hours after last administration of ASA/ clopidogrel, 12 hours after last administration of cilostazol) in the morning hours after 7 days treatment (i.e. on the 1st day of the next study period) and prior to intake of next study medication. Appropriate controls will be performed in accordance with the instructions provided by the manufacturers of test equipment each time any of the platelet tests is run.

Remaining plasma will be stored frozen for further biochemical assessments yet to be specified.

#### Skin bleeding time

The investigator will place a sphygmomanometer cuff on the upper arm of the subject and will inflate the cuff to 40 mm Hg. The investigator will immediately make an incision (6 mm long and 1 mm deep) on the volar surface of the forearm parallel to the antecubital crease using a Surgicutt<sup>®</sup> device. The flow of blood from the incision will be blotted gently with filter paper every 30 seconds. The time from the start of bleeding from the incision until blood no longer stained the filter paper is defined as the bleeding time (in seconds). The procedure will be performed safely in reference to the package insert for Surgicutt<sup>®</sup> device.

# 3.5.2 Secondary Outcome Variables

#### Safety:

- Vital signs
- Physical examination


- ECG
- Safety lab
- Adverse events

#### 3.6 Measures to Minimize/ Avoid Bias

Not applicable for this trial.

## 3.7 Trial Procedures

This is a single-centre, open-label, randomized, stratified, clinical trial in three parallel treatment groups to evaluate the effects of Cilostazol 100 mg oral twice daily, Acetylsalicylic acid (ASA) 100 mg oral once daily and Clopidogrel 75 mg once daily alone as well as combinations of Cilostazol 100 mg oral twice daily/ASA 100 mg oral once daily and Cilostazol 100 mg oral twice daily /Clopidogrel 75 mg once daily on the ex-vivo Platelet Function testing and Skin Bleeding Time. The trial will be performed with 68 healthy male subjects, aged between 18 and 45 years.

After signing screening informed consent, subjects will be tested for their *CYP2C19* genotype. Screening will be performed until at least 38 (34 + 4 replacements) subjects with the *CYP2C19* wild type allele (\*1/\*1), who show normal *CYP2C19* activity, and at least 19 (17 + 2 replacements) subjects with *CYP2C19* heterozygous (\*1/\*2), who show intermediate *CYP2C19* activity as well as at least 19 (17 + 2 replacements) subjects with *CYP2C19* homozygous (\*2/\*2) isoforms, who show poor *CYP2C19* activity, have been identified.

After signing treatment informed consent 68 subjects will undergo further screening procedures in order to determine baseline characteristics. Subjects failing these procedures will be replaced by screened subjects matching the genotype (normal, intermediate or low *CYP2C19* activity).

All 68 subjects will then be included in the treatment phase of the trial and will receive during the first week cilostazol 100 mg twice daily for 1 week (trial period A), followed by a 1 week wash-out period (trial period B, return to baseline). Subjects who fail to return to baseline with respect to platelet function testing and skin bleeding time will be re-tested within a further week.

After return to baseline, patients will be randomized into the four different treatment groups:


#### Protocol 21-13-102

#### Trial period C:

Treatment group 1 will consist of 17 subjects carrying the *CYP2C19 wild type allele* (\*I/\*I). This group will receive Acetylsalicylic acid 100 mg oral once daily for 7 consecutive days.

Treatment group 2 will consist of 17 subjects also carrying the CYP2C19 wild type allele (\*1/\*1). This group will receive Clopidogrel 75 mg once daily for 7 consecutive days.

Treatment group 3 will consist of 17 subjects carrying the CYP2C19 heterozygous (\*1/\*2) isoform. This group will receive Clopidogrel 75mg once daily for 7 consecutive days.

Treatment group 4 will consist of 17 subjects carrying the *CYP2C19 homozygous* (\*2/\*2) isoform. This group will receive Clopidogrel 75mg once daily for 7 consecutive days.

Following this treatment, group 1 will receive a combination of Cilostazol 100 mg oral twice daily and Acetylsalicylic acid 100mg oral once daily for 1 week (trial period D).

Treatment group 2, 3 and 4 will receive a combination of Cilostazol100 mg oral twice daily and Clopidogrel 75 mg once daily for 1 week (trial period D)..

Trial assessments are summarized in Table 3.7-1.

| Table 3.7-1 Schedule | of Assessme | ents | | | | | |
|---|---|---|---|---|---|---|---|
| Period | Screening | Baseline | Trial period<br>A<br>Cilostazol | Trial period B Wash-out, return to baseline | Trial period C ASA/ Clopidogrel | Trial period D Add-on of Cilostazol to ASA/ Clopidogrel | End of Trial /<br>Withdrawal of<br>study subjects |
| Visit(s) | 1 | 1 | 2 | 3 | 4 | 5 | 5 |
| Day(s) | - 90 to 0 | -14 to 0 | 1 to 7 | 8 to 14<br>(8 to 21) <sup>5</sup> | 15-21<br>(22 to 28) <sup>5</sup> | 22-29<br>(29 to 36) <sup>5</sup> | 29<br>(36) <sup>5</sup> |
| Assessments | | | | | | | |
| Screening informed consent | X | | | | | | |
| Genotyping | X | | | | | | |
| Inclusion/exclusion criteria | $X^{10}$ | $X^{10}$ | | | | | |
| Treatment informed consent | | $X^1$ | | | | | |
| Demographic data | | X | | | | | |
| Medical history | | X | | | | | |


| Concomitant medication | X | X | X | X | X | X |
|---|---|---|---|---|---|---|
| Platelet function testing <sup>9</sup> | X | | X <sup>8,11</sup> | | X <sup>8</sup> | |
| Skin Bleeding time | X | | X <sup>8, 11</sup> | | X <sup>8</sup> | |
| Physical examination | X | X | X | X | X | |
| Vital signs | X | X | X | X | X | |
| ECG | X | X | X | X | X | |
| Clinical laboratory assessments • Safety | X | X | X | X | X | |
| Clinical laboratory assessments • Baseline | X | | | | | |
| Randomization/<br>Stratification | | | | X | | |
| Drug Accountability | | X <sup>6</sup> | | X <sup>6</sup> | X <sup>6</sup> | $X^6$ |
| Deviations | | $X^7$ | $X^7$ | $X^7$ | $X^7$ | X <sup>7</sup> |
| IMP-Dispensing | | $X^{2,3}$ | | X | X | |
| IMP-Intake | | X <sup>4</sup> | | X <sup>4</sup> | X <sup>4</sup> | |


| Adverse Events | X | X | X | X | X | X |
|----------------|---|---|---|---|---|---|

- Patients can proceed with the treatment informed consent after a positive result of the genotyping is available
- The results of the baseline and safety laboratory assessments must be available before administration of IMP
- <sup>3</sup> IMP-administration will begin at least one day after the treatment informed consent was signed
- <sup>4</sup> IMP-intake will take place at the investigational site under supervision at the 1<sup>st</sup>, 4<sup>th</sup>, 6<sup>th</sup>, and 7<sup>th</sup> day (trial period A, C and D). Drug intake of ASA and clopidogrel will be in the morning hours, for cilostazol drug intake will be twice daily: once in the morning and once in the evening. Date and time of study drug administration are recorded.
- If a subject does not reach baseline values after the 7 day wash-out phase, the wash-out phase will be extended for additional 7 days
- <sup>6</sup> Drug Accountability: Documentation of drug dispense, intake and return
- Deviations: Documentation of non-compliance with trial procedures and violations from the trial protocol
- Primary and secondary efficacy parameters will be tested at trough (i.e. 24 hours after last administration of ASA/ clopidogrel, 12 hours after last administration of cilostazol) in the morning hours after 7 days treatment (i.e. on the 1st day of the next study period) and prior to intake of next study medication.
- The validity of test results will be assured by the use of calibrated equipment and/ or the use of internal controls. Controls will be carried out each time (day) the corresponding parameter is measured.
- The subjects who meet all the inclusion criteria will be selected. If the investigator discovers that the subjects fall under any of the exclusion criteria, the subjects should be excluded from the trial.
- During Period B platelet function testing and skin bleeding time measurements will be performed on the first and the last day of the period (days 8 and 14). If the results of these tests during this period indicate that a subject failed to return to baseline and that an extension of the wash-out period is required, platelet function testing and skin bleeding time measurements will be performed again on the last day of the extension week (unscheduled visit, day 21).

## 3.7.1 General Inpatient Procedures

Subjects will not be required to stay overnight at the investigational site. IMP-intake will take place at the investigational site under supervision at the 1<sup>st</sup>, 4<sup>th</sup>, 6<sup>th</sup>, and 7<sup>th</sup> day (trial period A, C and D). Drug intake of ASA or Clopidogrel will be in the morning hours, for Cilostazol drug intake will be twice daily: once in the morning and once in the evening. All measurements of PFT and BT will be at trough in the morning hours after 7 days treatment (1st day of next study period) and prior to intake of next study medication.

# 3.7.2 Dietary Requirements

During the course of the trial, subjects should consume "normal" amounts of protein, carbohydrate and fat (no special dietary requirements), as judged by the investigator. Not to be included in the trial are subjects that are on a strictly vegetarian or vegan diet.

#### 3.7.3 Schedule of Assessments

All subjects participating in the trial must be evaluated according to the assessment schedule of the trial outlined in Table 3.7.1.

## 3.7.3.1 Visit 1 (Screening/ Baseline)

For all subjects the following procedures will be conducted and/or recorded in the subject's CRF:

**Screening Procedures** 

(Screening procedures are required to be performed within 90 days prior to Day 1):

- Written informed consent for screening
- Review of inclusion/ exclusion criteria
- Genotyping

The subjects who meet all the inclusion criteria 1 to 4 will be selected. If the investigator discovers that the subjects fall under any of the exclusion criteria, the subjects should be excluded from the trial

**Baseline Procedures** 

(baseline procedures are required to be performed within 14 days prior to Day 1 and


might be carried out on the same day as screening procedures after positive result of genotyping):

The following procedures will be performed and subjects who meet all the inclusion criteria and do not fall under any of the exclusion criteria will be selected.

- Written informed consent for treatment
- Demographic data
- Medical history
- Review of inclusion/ exclusion criteria
- Concomitant medication
- Platelet function testing
- Measurement of bleeding time
- Physical examination including weight and height
- Vital signs (Systolic blood pressure, diastolic blood pressure, pulse rate, body temperature)
- Standard 12-lead ECG
- Laboratory tests safety (haematology, clinical chemistry, coagulation, urine)
- Laboratory tests baseline (TSH in serum, urine drug screening, breath alcohol, and infectious diseases)
- Adverse events

#### 3.7.3.2 Visit 2 – Trial period A – Day 1 - 7

- IMP dispense and controlled administration of IMP at the site at day 1.
   IMP (cilostazol) will be taken for 7 consecutive days.
   The results of the baseline and safety laboratory assessments must be available before administration of IMP. IMP-administration will begin at least one day after the treatment informed consent was signed.
- Controlled IMP intake will take place at the investigational site under supervision at the 1<sup>st</sup>, 4<sup>th</sup>, 6<sup>th</sup>, and 7<sup>th</sup> day. Cilostazol drug intake will be twice daily: once in the morning and once in the evening. Date and time of study drug administration are recorded.
- Concomitant medication
- Adverse events
- Vital signs (Systolic blood pressure, diastolic blood pressure, pulse rate, body temperature) at day 7

- Comprehensive physical examination including weight at day 7
- Standard 12-lead ECG at day 7
- Laboratory tests safety (haematology, clinical chemistry, coagulation, urine) at day 7
- Deviations

## 3.7.3.3 Visit 3 – Trial period B – Day 8 – 14 (21)

- IMP return and drug accountability at day 8
- Platelet function testing at day 8. Platelet function will be tested at trough i.e. 12 hours after last administration of cilostazol
- Measurement of bleeding time at day 8
- Concomitant medication
- Adverse events
- Vital signs (Systolic blood pressure, diastolic blood pressure, pulse rate, body temperature) at day 14
- Physical examination including weight at day 14
- Standard 12-lead ECG at day 14
- Platelet function testing at day 14 in the morning hours
- Measurement of bleeding time at day 14 in the morning hours
- Laboratory tests safety (haematology, clinical chemistry, coagulation, urine) at day 14
- Deviations

This wash-out period will lead to a return to baseline in relation to platelet function testing and bleeding time. Subjects who fail to return to baseline with respect to platelet function testing and bleeding time will be re-tested within a further week.

#### 3.7.3.4 Visit 3 unscheduled – Trial period B – Day 15 - 21

Visit 3 unscheduled for subjects to be re-tested within a further week from Visit 3.

- Concomitant medication
- Adverse events
- Platelet function testing at day 21 in the morning hours


- Measurement of bleeding time at day 21 in the morning hours
- Deviations

#### 3.7.3.5 Randomization/ Stratification

Subjects with normal *CYP2C19* activity will be randomized to either Group 1 (ASA oral tablets) or Group 2 (Clopidogrel oral tablets). Randomization will be done on Visit 4.

### 3.7.3.6 Visit 4 – Trial period C – Day 15 – 21 (22 - 28)

- IMP dispense and controlled administration of IMP at the site at day 1
- IMP (ASA or clopidogrel) will be taken for 7 consecutive days
- Controlled IMP intake will take place at the investigational site under supervision at the 1<sup>st</sup>, 4<sup>th</sup>, 6<sup>th</sup>, and 7<sup>th</sup> day of this visit. Drug intake of ASA and clopidogrel will be in the morning hours. Date and time of study drug administration are recorded.
- Concomitant medication
- Adverse events
- Vital signs (Systolic blood pressure, diastolic blood pressure, pulse rate, body temperature) at day 21 (28)
- Physical examination including weight at day 21 (28)
- Standard 12-lead ECG at day 21 (28)
- Laboratory tests safety (haematology, clinical chemistry, coagulation, urine) at day 21 (28)
- Deviations

# 3.7.3.7 Visit 5 – Trial period D – Day 22 – 29 (29 - 36)

- IMP return and drug accountability at day 22 (29)
- Platelet function testing at day 22 (29). Platelet function will be tested at trough i.e. 24 hours after last administration of ASA/ clopidogrel respective 12 hours after last administration of cilostazol and prior to intake of next study medication
- Measurement of bleeding time at day 22 (29) and prior to intake of next study medication
- IMP dispense and controlled administration of IMP at the site at day 1

- IMP (ASA/ cilostazol or clopidogrel/ cilostazol) will be taken for 7 consecutive days.
- Controlled IMP intake will take place at the investigational site under supervision at the 1<sup>st</sup>, 4<sup>th</sup>, 6<sup>th</sup>, and 7<sup>th</sup> day of this visit. Drug intake of ASA and clopidogrel will be in the morning hours, for cilostazol drug intake will be twice daily: once in the morning and once in the evening. Date and time of study drug administration are recorded.
- Concomitant medication
- Adverse events
- Vital signs (Systolic blood pressure, diastolic blood pressure, pulse rate, body temperature) at day 28 (35)
- Physical examination including weight at day 28 (35)
- Standard 12-lead ECG at day 28 (35)
- Laboratory tests safety (haematology, clinical chemistry, coagulation, urine) at day 28 (35)
- IMP return and drug accountability at day 28 (35)
- Platelet function testing at day 29 (36). Platelet function will be tested at trough
  i.e. 24 hours after last administration of ASA/clopidogrel respective 12 hours after
  last administration of cilostazol
- Measurement of bleeding time at day 29 (36)
- End of trial procedures at day 29 (36):
  - o Trial summary
  - o Concomitant medication
  - Adverse events
  - Deviations
  - Comments

#### 3.7.3.8 Time of Withdrawal

If the study subject is withdrawn from the trial after the start of IMP administration, the End of trial procedures as described in Section 3.7.3.7 will be performed.

# 3.7.4 Safety Assessments

Safety will be assessed by investigation of:

Vital signs


- o Pulse rate in beats/ min.
- o Diastolic and systolic blood pressure in mmHg
- o Body temperature in °C
- Physical examination
  - Complete physical examination of organ systems in relation to findings and abnormalities
  - o Height in cm
  - o Weight in kg
- ECG
  - 12-lead ECG in relation to rhythm, frequency, clinical significant abnormalities
- Safety lab
  - o Haematology, clinical chemistry, coagulation, urine
- Adverse events
  - o Documentation of all reported AEs

# 3.7.4.1 Clinical Laboratory Tests

The tests listed in Table 3.7.4.1-1 will be collected at the times presented in the schedule of assessments, Table 3.7-1, and processed in accordance with directions from the clinical chemistry laboratory.

| <b>Table 3.7.4.1-1</b> | Cable 3.7.4.1-1 Safety Clinical Laboratory Tests | |
|---|---|---|
| Hematology: | <u>C</u> | Clinical Chemistry: |
| HGB | A | Albumin |
| HCT | T | Total Protein |
| RBC | A | AP |
| WBC | A | ALT |
| Platelets | A | AST |
| Basophils | G | GGT |
| Eosinophils | L | LDH |
| Lymphocytes | В | Bili |
| Monocytes | P | Potassium |
| Neutrophils | S | Sodium |
| Abs. Basophils | C | Chloride |
| Abs. Eosinophils | C | Creatinine |
| Abs. Lymphocytes | U | Jrea |
| Abs. Monocytes | U | Jric acid |
| Abs. Neutrophils | G | Glucose |

#### Protocol 21-13-102

| Coagulation: | Urine: |
|---|---|
| Congulation. | Offic. |
| PT | Blood |
| INR | Clarity |
| PTT | Colour |
| Fibrinogen | Glucose |
| | Ketones |
| | Nitrite |
| | рН |
| | Protein |
| | RBC |
| | WBC |
| | Specific Gravity |
| In addition to these safety laboratory parameters, the following investigations will be performed at base | |
| Drug Screen Urine: | Infectious diseases: |
| Amphetamines | HIV 1&2 EIA Ab |
| Barbiturates | HBs Ag |
| Benzodiazepines | HCV Ab |
| Cannabinoids | |
| Cocaine | |
| Opiates | |
| Phencyclidine | |
| Propoxyphene | |
| D 0 D 4 | |
| Drug Screen Breath: | |
| Ethanol | |
| Clinical Chemistry: | |
| TSH in serum | |

Blood collection for platelet function testing will be performed at trough i.e. 24 hours after last administration of ASA/ clopidogrel respective 12 hours after last administration of cilostazol and prior to intake of next study medication.

Measurement of skin bleeding time will be performed in a timely relation to the collection for platelet function testing.

Platelet function testing and skin bleeding time measurements will be performed locally at the site. Validity of measurements regarding platelet function will be assured by the use of calibrated equipment and/or the use of test specific controls in accordance with the manufacturers' instructions and the technical report Thrombocyte diagnostics (DIN SPEC 58961:2013-04).

Appropriate controls will be used at each time any of the platelet tests is run as foreseen by the device manufacturer and/or the technical report. For this purpose commercially

available PFT devices (LTA PAP4, Multiplate, VerifyNow P2Y12) will be used. Control samples for verification of measurements are available for all devices.

Blood and urine analysis for baseline and safety assessments will be performed locally at the site. Ethanol will be determined as breath alcohol employing a CE certified breathalyzer.

A laboratory manual will be developed and provide detailed instructions for handling of platelet function testing and bleeding time measurements as well as for blood and urine analysis for baseline and safety assessments.

## 3.7.4.2 Physical Examination and Vital Sign Assessments

Physical examination will be performed by a physician. It is preferred that the same investigator is performing all physical examinations for any individual subject throughout the course of the trial.

Abnormalities and findings will be documented in the respective CRF section. Newly identified clinically significant findings and abnormalities need to be documented as an Adverse Event.

Vital signs will be performed by trial staff experienced in these aspects of clinical research.

Height will be measured and documented in cm, weight will be measured and documented in kg. Body temperature will be measured and documented in °C.

Pulse rate will be measured and documented in beats/ min. Diastolic and systolic blood pressure will be measured and documented in mmHg. Pulse rate and blood pressure will be obtained after subjects having had 10 minutes rest in supine position.

#### 3.7.4.3 ECG Assessments

12-lead ECG will be performed throughout the trial. Findings in relation to rhythm, frequency, clinical significant abnormalities will be captured in the CRF. Each ECG record needs to be reviewed and signed by a physician. ECG will be obtained after subjects having had 10 minutes rest in supine position.

#### 3.7.5 End of Trial

The End of Trial date is defined as the last date of contact or the date of the final contact attempt of the last subject completing (last patient last visit) or withdrawing from the trial.

# 3.8 Stopping Rules, Withdrawal Criteria and Procedures, and Subject Replacement

#### 3.8.1 Entire Trial or Treatment Arm(s)

If the sponsor terminates or suspends the trial for safety or unanticipated other reasons, prompt notification will be given to investigators, ECs, and regulatory authorities in accordance with regulatory requirements.

#### 3.8.2 Individual Site

The investigator will notify the sponsor promptly if the trial is terminated by the investigator or the EC at the site.

#### 3.8.3 Individual Subject

If a subject discontinues from the trial prematurely, the reason must be fully evaluated and recorded appropriately in source documents and the CRF. If the subject is being withdrawn because of an adverse event (AE), that AE must be indicated as the reason for withdrawal.

All subjects have the right to withdraw at any point during treatment without prejudice. The investigator can discontinue a subject's participation in the trial at any time if medically necessary. In addition, subjects meeting the following criteria must be withdrawn from the trial:

- a) occurrence of any AE, intercurrent illness or abnormality in a laboratory assessment which, in the opinion of the investigator, warrants the subject's permanent withdrawal from the trial;
- b) treatment with a prohibited concomitant medication other than the use of appropriate medications for the treatment of adverse events under direction of the investigator;

- c) subject noncompliance, defined as refusal or inability to adhere to the trial schedule or procedures;
- d) at the request of the subject, investigator, sponsor or regulatory authority;
- e) subject is lost to follow-up.

The investigator will notify the sponsor promptly when a subject is withdrawn.

#### 3.9 Screen Failures

A screen failure subject is one from whom informed consent is obtained and is documented in writing (ie, subject signs an informed consent form), but who is not started on treatment.

# 3.10 Definition of Completed Subjects

The treatment period is defined as the time period during which subjects are evaluated for primary and/ or secondary objectives of the trial. Subjects who are evaluated at the last scheduled visit during the treatment period will be defined as trial completers. For purposes of this trial, subjects who complete all of the 4 trial periods will be defined as completers

#### 3.11 Subject Compliance

Inappropriate taking of IMP and lack of adherence to visit schedule will be considered as non-compliance of subjects and the investigator or designee will contact the sponsor at the earliest possible time by telephone or e-mail. Investigator and sponsor will come as quickly as possible to a joint decision regarding the subject's continuation in the trial. This decision will be documented by the investigator and the sponsor, and reviewed by the site monitor.

## 3.12 Protocol Deviations

In the event of a significant deviation from the protocol due to an emergency, accident, or mistake (e.g. violation of informed consent process, IMP dispensing or subject dosing error, treatment assignment error, subject enrolled in violation of eligibility criteria or concomitant medication criteria), the investigator or designee will contact the sponsor at

the earliest possible time by telephone or e-mail. Investigator and sponsor will come as quickly as possible to a joint decision regarding the subject's continuation in the trial. This decision will be documented by the investigator and the sponsor, and reviewed by the site monitor.

#### 4 Restrictions

#### 4.1 Prohibited Medications

No concomitant medication is allowed from screening to end of trial. Subjects taking other concomitant medication apart from allowed rescue medication need to be discussed with the sponsor's medical team and may be replaced by screened subjects matching the genotype.

Single doses of acetaminophen 500 mg orally for the treatment of headache are acceptable as a rescue. The maximum dose of 3 g per day for more than 2 consecutive days must not be exceeded. In that case subject may be excluded from trial and other treatment options will be considered by the investigator.

For treatment of diarrhoea single doses of loperamide are accepted.

# 5 Reporting of Adverse Events

#### 5.1 Definitions

An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.

A suspected adverse reaction means any AE for which there is a reasonable possibility that the drug caused the AE. For the purpose of IND safety reporting, "reasonable possibility" means there is evidence to suggest a causal relationship between the drug and the AE. Suspected adverse reaction implies a lesser degree of certainty about causality.

A serious adverse event (SAE) includes any event that results in any of the following outcomes:

- 1) Results in death
- 2) Is life-threatening, ie, the subject was, in the opinion of the investigator, at <u>immediate</u> risk of death from the event as it occurred. It does not include an event that, had it occurred in a more severe form, might have caused death.


- 3) Results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
- Requires in-patient hospitalization or prolongs hospitalization
   NOTE: A pre-scheduled hospitalization is not considered an SAE.
- 5) Is a congenital anomaly or birth defect
- 6) Is considered a medically significant event as, based upon appropriate medical judgment, it may jeopardize the subject or may require medical or surgical intervention to prevent one of the outcomes listed above. Example are a allergic bronchospasm requiring intensive treatment in an emergency room or home, blood dyscrasias or convulsions that do not result in hospitalization, or the development of drug dependency or drug abuse.

Non-serious adverse events are all adverse events that do not meet the criteria for a "serious" adverse event.

#### Immediately Reportable Event (IRE) (also see Section 5.3):

- Any serious adverse event
- Any adverse event that necessitates discontinuation of IMP
- Potential Hy's Law cases (Any increase of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 3 times the upper normal limit or screening value with an increase in total bilirubin ≥ 2 times the upper normal limit or screening value)
- Fathering is also defined as IREs. Although fathering is not an adverse event, it
  will mandate drug discontinuation and must be reported to the sponsor or
  designee as an IRE. Pregnancy of female partner will only be documented on the
  AE-section if there is an abnormality or complication
- All events involving overdose, misuse, and abuse.
   This includes accidental overdose by investigator or patient. It also includes all such events, whether the course is symptomless, or whether an AE or SAE results.
   These events may involve cilostazol or any other medicinal products or illicit drugs (See also Section 5.7)

<u>Clinical Laboratory Changes</u>: It is the investigator's responsibility to review the results of all laboratory tests as they become available. This review will be documented by the

investigator's dated signature on the laboratory report. For each abnormal laboratory test result, the investigator needs to ascertain if this is an abnormal (ie, clinically significant) change from baseline for that individual subject. (This determination, however, does not necessarily need to be made the first time an abnormal value is observed. The investigator may repeat the laboratory test or request additional tests to verify the results of the original laboratory tests). If this laboratory value is determined by the investigator to be an abnormal change from baseline for that subject, this is considered an AE.

<u>Severity:</u> Adverse events will be graded on a 3-point scale and reported as indicated on the CRF. The intensity of an adverse experience is defined as follows:

**1 = Mild:** Discomfort noticed, but no disruption to daily activity.

**2 = Moderate:** Discomfort sufficient to reduce or affect normal daily activity.

**3 = Severe:** Inability to work or perform normal daily activity.

IMP Causality: Assessment of causal relationship of an AE to the use of IMP:

**Related**: There is a reasonable possibility of a causal relationship.

**Possibly related**: There is a reasonable causal relationship between the IMP and the

AE. Dechallenge is lacking or unclear.

**Unlikely related**: There is a temporal relationship to IMP administration, but there is

not a reasonable causal relationship between the IMP and the AE.

**Not Related**: There is no temporal or reasonable relationship to IMP

administration.

## 5.2 Eliciting and Reporting Adverse Events

The investigator will periodically assess subjects for the occurrence of AEs. In order to avoid bias in eliciting AEs, subjects should be asked the following non-leading question: "How are you feeling, and how have you felt since the last visit?" All AEs (serious and non-serious) reported by the subject must be recorded on the source documents and CRFs provided by the sponsor or designee.

In addition, the sponsor or designee must be notified immediately by telephone or fax of any <u>immediately reportable events</u> according to the procedure outlined below in Section 5.3. Special attention should be paid to recording hospitalization and concomitant medications.

## 5.3 Immediately Reportable Events (IRE)

The investigator must report immediately and not later than 24 hours after either the investigator or site personnel become aware of any IRE as defined in section 5.1 by telephone or by fax to the sponsor or designee as outlined in Appendix 1. An Immediately Reportable Event (IRE) form should be completed and sent by fax or overnight courier to the sponsor or designee. The investigator should sign the IRE form personally.

(Please note that the IRE form is NOT the adverse event CRF.)

If the IRE cannot be sent successfully electronically or on time (eg, due to technical difficulties) using the contact information above, the report should be made by fax or, if not possible, via phone to the contact person above.

Receipt of the IRE by the sponsor will be confirmed as soon as possible, usually within 24 hours. If further information is required, the sponsor will contact the investigator (usually via the Clinical Research Associate [CRA] responsible for the site). The investigator is responsible for promptly providing any further information requested.

<u>Non-serious events</u> that require discontinuation of IMP (including laboratory abnormalities) should be reported to the sponsor within 3 working days. The IRE form must be completed and sent by fax or overnight courier to the sponsor or designee.

Subjects experiencing serious adverse events should be followed clinically until their health has returned to baseline status or until all parameters have returned to normal, or have otherwise been explained. It is expected that the investigator will provide or arrange appropriate supportive care for the subject.

## 5.4 Potential Hy's Law Cases

For a subject that experiences an elevation in AST or ALT that is  $\geq 3$  times the upper normal limit or whose levels increase  $\geq 3$  times their initial screening value, a total bilirubin level should also be evaluated. If the total bilirubin is  $\geq 2$  times the upper

normal limit or  $\geq 2$  times their screening value, complete an IRE form with all values listed and also report as an AE on the CRFs.

## 5.5 Pregnancy

Not applicable for this trial.

## 5.6 Fathering

Male subjects who are sexually active must avoid fathering a child for 30 weeks after the last dose of cilostazol by abstain from sex or use of effective contraceptive method during the clinical trial and 30 weeks after. The investigator must immediately notify the sponsor of any reported pregnancy of the female partner associated with cilostazol exposure, including a period of 30 weeks for after the last dose of cilostazol and record the event on the IRE form and forward it to the sponsor. The sponsor will forward Pregnancy Surveillance Form(s) for monitoring the outcome of the pregnancy.

Pregnancy of female partner is an IRE and must be reported immediately as such using the IRE Form. Pregnancy of female partner will only be documented on the AE-section in the CRF if there is an abnormality or complication.

Upon receipt of an IRE concerning pregnancy, the safety contact of the sponsor will inform the investigator of the further information required. The investigator must report to the sponsor, on appropriate Pregnancy Surveillance form(s), follow-up information regarding the course of the pregnancy, including perinatal and neonatal outcome. Infants will be followed for a minimum of 6 months. Any congenital anomaly or birth defect constitutes an SAE and must be entered as follow-up information on the IRE Form and on the AEs eCRF.

#### 5.7 Overdose, Misuse, Abuse

Overdose, misuse, or abuse of cilostazol or any other medication or illicit drug constitute IREs, and must be reported and recorded as such.

If such an event fulfils the definition of an AE or an SAE, they must be documented as such on the AEs CRF, as well.

## 5.8 Procedure for Breaking the Blind

Not applicable for this trial.

# 5.9 Follow-up of Adverse Events

## 5.9.1 Follow- up of Adverse Events

Adverse events that are identified on the last scheduled contact (End of trial procedures on day 29 or the day of withdrawal examination) must be recorded on the AE CRF with the current status noted. All adverse events that are ongoing at this time will be recorded as ongoing on the CRF.

The investigator will follow the adverse events until the events are resolved, or the subject is lost to follow-up. Resolution means the subject has returned to the baseline state of health, or the investigator does not expect any further improvement or worsening of the subject's condition. The investigator will continue to report any significant follow-up information to sponsor or designee up to the point the event has been resolved.

### 5.9.2 Follow- up of Post Trial Serious Adverse Events

Serious adverse events that are **identified on the last scheduled contact** (End of trial procedures on day 29 or the day of withdrawal examination) must be reported to the Sponsor or designee as named in Appendix 1 according to the reporting procedures outlined in Section 5.3. This may include **unresolved previously reported** serious adverse events, or **new serious adverse events**. The investigator will follow serious adverse events according to the procedures outlined in Section 5.9.1.

This trial requires that subjects be actively monitored for serious adverse events up to 90 days after discharge from the trial.

# 5.9.3 Follow-up and Reporting of Serious Adverse Events Occurring after Last Scheduled Contact

Any new serious adverse events reported by the subject to the investigator that occur after the last scheduled contact, and are determined by the investigator to be reasonably associated with the use of the IMP, should be reported to sponsor or designee. This may include serious adverse events that are captured on follow-up telephone contact or at any other time point after the defined trial period (ie, up to last scheduled contact). The investigator should follow serious related adverse events identified after the last scheduled contact until the events are resolved, or the subject is lost to follow-up. The

investigator should continue to report any significant follow-up information to up to the point the event has been resolved.

# 6 Pharmacokinetic/ Pharmacodynamic Analysis

Not applicable for this trial.

# 7 Statistical Analysis

#### 7.1 Sample Size

The primary variable of the trial is ex-vivo inhibition of platelet aggregation. Comparisons of the inhibition of platelet aggregation are made between subjects during treatment of reference medication alone (Reference) and during the concomitant treatment of reference medication and cilostazol (Test). When assuming that the expected platelet aggregation treatment mean ratio is 1 with a standard deviation of 27% (Angiolillo *et al*, 2011) <sup>19</sup>, for showing equivalence of a single parameter, a sample size of 17 patients per group would be required to provide a 90% power. That is, with the crossover design, 17 subjects yield a probability of 0.95 to reject the null hypotheses that the platelet aggregation with treatment of cilostazol along with reference medication versus reference medication along is below 0.70 or above 1.43, ie, the 95% confidence interval (CI) is contained within the equivalence limit [0.70,1.43].

Ex-vivo inhibition of platelet aggregation is the primary endpoint of the study and accordingly study hypothesis and sample size estimation has been based on the primary end-point. Similar considerations apply to the assessment of bleeding time, for which the biological variation is considered to be greater than for platelet aggregation, as it is affected additionally by tissue- or organ-dependent differences in the physiology of the vascular bed. The hypothesis tested for bleeding time will be analogue to these tested for platelet aggregation, however, the statistical power of treatment effects estimated for platelet aggregation does not apply to bleeding time.

## 7.1.1 Sensitivity analysis

If a substantial number of patients drop out of the analysis before finishing the third period, an analysis of covariance (ANCOVA) will be provided to assess the impact of missing data on the method chosen to analyse the data.

## 7.2 Analysis of Demographic and Baseline Characteristics

Summary statistics for age, race, body weight, height, and BMI will be summarized.

## 7.2.1 Datasets for Analysis

The safety dataset includes all subjects that were administered at least one dose of IMP. Full Analysis Set: All subjects who completed both periods of treatment with reference medication alone and treatment with reference medication and cilostazol.

Safety Analysis Data Set: All subjects who received at least one dose of trial medication are included in the safety, demographic, and baseline characteristic analyses.

## 7.3 Safety Analysis

Safety analysis will be conducted based upon the safety population, which is defined as all subjects who take at least one dose of trial medication. Safety variables to be analysed include clinical laboratory tests, vital signs, electrocardiograms, and adverse events. In general, summary statistics of changes from baseline will be provided for safety variables based upon all available data.

#### 7.3.1 Adverse Events

All AEs will coded by Medical Dictionary for Regulatory Activities system organ class and preferred term. The incidence of the following events will be summarized by each cohort and by treatment regimen:

- TEAEs by severity
- Potentially drug-related TEAEs
- TEAEs with an outcome of death
- Serious TEAEs
- Discontinuations due to TEAEs

# 7.3.2 Clinical Laboratory Data

Laboratory data will be listed and changes in clinical laboratory test values from baseline will be summarized by each cohort using descriptive statistics.

## 7.3.3 Physical Examination and Vital Signs Data

Physical examination findings will be listed by subject and by each cohort. Vital sign data will be listed and changes in vital sign test values from baseline will be summarized by cohort and treatment regimen using descriptive statistics.

#### **7.3.4 ECG Data**

Electrocardiogram data will be listed and changes in ECG values from baseline will be summarized by each cohort and treatment regimen using descriptive statistics.

## 7.4 Pharmacokinetic Comparisons

Not applicable for this trial.

## 7.5 Pharmacodynamic Comparisons

#### 7.5.1 Primary analysis

The primary analysis variables is the effect on the ex-vivo inhibition of platelet aggregation. Platelet aggregation is assessed after stimulation of aggregation by

Primary efficacy parameters:

- Ex-vivo Platelet function: primary parameters to be determined in citrated platelet rich plasma (PRP) by
  - $\circ$  Light transmission aggregometry (5  $\mu$ M ADP, residual aggregation at 5 minutes)
  - Light transmission aggregometry (Arachidonic acid 500 mg/L, residual aggregation at 5 minutes)

Secondary efficacy parameters:

- Skin bleeding time: to be determined with Ivy method utilizing standardized bleeding with Surgicutt® device
- Ex-vivo Platelet functionas determined by
  - Light transmission aggregometry in PRP (20 μM ADP, collagen 1mg/L and 2.5 mg/L, TRAP 25 μM, residual aggregation at 5 minutes)
  - Multiple electrode impedance aggregometry in hirudine-anticoagulated blood (Multiplate<sup>®</sup>) (ASPItest, ADPtest, ADP/PGEtest, TRAP-test)
  - o VerifyNow<sup>TM</sup> (P2Y12 and Aspirin test)
  - o Vasodilator-stimulated phosphoprotein (VASP) by flow cytometry
  - P-Selectin expression by flow cytometry

For individual subjects, inhibition of platelet aggregation (IPA) is defined as the percentage decrease of platelet aggregation of stimulated plasma before and after treatments with trial medications.

To rule out of a 30% inhibition and establish equivalence of inhibition of platelet aggregation, each parameter of inhibition of platelet aggregation will be compared in subjects during treatment with reference medication along and during treatment with reference medication and cilostazol.

Equivalence will be indicated if the 95% confidence interval (CI) for the ratio (T/R) of the inhibition of platelet aggregation, based on the analysis of the log-transformed data, is contained within the equivalence limits of 0.7 0 to 1.43 for each parameter of platelet aggregation. Due to the nature of the normal-theory CIs, this comparison of the 95% CI to the equivalence limits is equivalent to carrying out two 1-sided tests of hypotheses, each at the 5% level of significance for each parameter.

Analysis of variance (ANOVA) will be performed on the natural-log transformed inhibition of platelet aggregation using the MIXED procedure in SAS<sup>®</sup>. The mixed-effects linear model for each parameter will include terms for period and treatment as fixed effects, and a term for subjects as a random effect. From each analysis, we obtain the least squares treatment means and difference (T - R) and the 95% CI for the treatment difference. Then, the antilogs of the difference and the confidence limits provide the estimate and 95% CI for the ratio (T/R) of the geometric means of platelet aggregation parameters of the test and reference.

This method will be used to compare all drugs/ combinations i.e. cilostazol vs. baseline; clopidogrel vs. baseline; clopidogrel vs. clopidogrel alone; cilostazol/ASA vs. ASA alone, as well as the different genotype combinations.

Bleeding time at baseline, after monotherapy with cilostazol, aspirin or clopidogrel as well as concomitant treatment of cilostazol plus aspirin and cilostazol plus clopidogrel will also be analysed using the methodology specified in section 7.5.1. Natural log-transformation will be applied to bleeding time to fit a mixed effect ANOVA model.

# 8 Trial Drug Management

## 8.1 Packaging and Labelling

Trial drugs will be provided to the investigator(s) by the sponsor (or designated agent). The IMP will be labelled to clearly disclose the compound ID, protocol number, the sponsor's name and address, instructions for use, route of administration, and appropriate precautionary statements.

## 8.2 Storage

Trial drugs will be stored in a securely locked cabinet or enclosure. Access should be strictly limited to the investigators and their designees. Neither the investigators nor any designees may provide trial drugs to any subject not participating in this protocol.

The IMP will be stored at 15° - 25 °C. The clinical site staff will maintain a temperature log in the drug storage area recording the temperature at least once each working day.

#### 8.3 Accountability

The investigator, or designee, must maintain an inventory record of trial drug(s) (including IMP, active control, or placebo) received, dispensed, administered and returned.

#### 8.4 Returns and Destruction

Upon completion or termination of the trial, all unused and/or partially used IMP must be returned the sponsor or a designated agent.


All IMP returned to the sponsor must be accompanied by the appropriate documentation and be clearly identified by protocol number and trial site number on the outermost shipping container. Returned supplies should be in the original containers (eg, subject kits). The assigned trial monitor will facilitate the return of unused and/or partially used IMP.

## 8.5 Reporting of Product Quality Complaints

The following describes the methods and timing for reporting Product Quality Complaints (PQCs).

A PQC is any written, electronic, or verbal communication by a healthcare professional, consumer, subject, medical representative, Competent Authority, regulatory agency, partner, affiliate or other third party that alleges deficiencies or dissatisfaction related to identity, quality, labelling, packaging, reliability, safety, durability, tampering, counterfeiting, theft, effectiveness or performance of a drug product or medical device after it is released for distribution. Examples include, but are not limited to, communications involving:

- Failure/malfunction of a product to meet any of its specifications
- Incorrect or missing labelling
- Packaging issues (eg, damaged, dirty, crushed, missing product)
- Blister defects (eg, missing, empty blisters)
- Bottle defects (eg, under/over-fill, no safety seal)
- Vial defects
- Product defect (eg, odour, chipped, broken, embossing illegible)
- Loss or theft of product

#### 8.5.1 Eliciting and Reporting Product Quality Complaints

The investigator or designee must record all Product Quality Complaints identified through any means from the receipt of the IMP from sponsor through and including reconciliation and up to destruction, including subject dosing. The investigator or designee must notify the sponsor (or sponsor's designee) within 24 hours of becoming aware of the PQC by e-mail or telephone and according to the procedure outlined below.

Identification of a PQC by the subject should be reported to the site investigator, who should then follow one of the reporting mechanisms above.

## 8.5.2 Information Required for Reporting Purposes

- Description of complaint
- Reporter identification (eg, subject, investigator, site, etc)
- Reporter contact information (eg, address, phone number, e-mail address.)
- ID of material (product/compound name, coding)
- Clinical protocol reference (number and/or trial name)
- Dosage form/strength (if known)
- Pictures (if available)
- Availability for return

#### 8.5.3 Return Process

Indicate during the report of the PQC if the complaint sample is available for return. If the complaint sample is available for return, return it in the product retrieval package, which will be provided by Sponsor.

It should be documented in the site accountability record that a complaint sample for a dispensed kit has been forwarded to Sponsor for complaint investigation.

#### 8.5.4 Assessment/Evaluation

Assessment and evaluation of Product Quality complaints will be handled by Sponsor Quality Management group.

# 9 Records Management

#### 9.1 Source Documents

Source documents are defined as the results of original observations and activities of a clinical investigation. Source documents will include, but are not limited to, progress notes, electronic data, screening logs, and recorded data from automated instruments. All source documents pertaining to this trial will be maintained by the investigators and made available for direct inspection by authorized persons. Investigator(s)/institution(s) will


permit trial-related monitoring, audits, EC review, and regulatory inspection(s) by providing direct access to source data/documents by authorized persons as defined in the ICF.

#### 9.2 Data Collection

During each subject's visit to the clinic, a clinician participating in the trial will record progress notes to document all significant observations. At a minimum, these notes will contain:

- Documentation of the informed consent process, including any revised consents;
- The date of the visit and the corresponding Visit or Day in the trial schedule;
- General subject status remarks, including any significant medical findings. The
  severity, frequency, and duration of any AEs and the investigator's assessment of
  relationship to IMP must also be recorded;
- Any changes in concomitant medications or dosages;
- A general reference to the procedures completed;
- The signature (or initials) and date of all clinicians who made an entry in the progress notes.

In addition, any contact with the subject via telephone or other means that provides significant clinical information will also be documented in the progress notes as described above. Any changes to information in the trial progress notes and other source documents will be <u>initialled and dated on the day the change is made</u> by a site trial staff member authorized to make the change. Changes will be made by striking a single line through erroneous data, and clearly entering the correct data (eg, wrong data right data). If the reason for the change is not apparent, a brief explanation for the change will be written adjacent to the change by the clinician.

Information from the trial progress notes and other source documents will be entered by investigative site personnel directly onto electronic CRFs in the sponsor's electronic data capture (EDC) system. Changes to the data will be captured by an automatic audit trail.

### 9.3 File Management at the Trial Site

The investigator will ensure that the trial centre file is maintained in accordance with Section 8 of the International Conference on Harmonization (ICH) GCP Guideline and as required by applicable local regulations. The investigator/institution will take measures to prevent accidental or premature destruction of these documents.

## 9.4 Records Retention at the Trial Site

International regulations require all investigators participating in clinical trials to maintain detailed clinical data.

The investigator must not dispose of any records relevant to this trial without either (1) written permission from the sponsor or (2) providing an opportunity for the sponsor to collect such records. The investigator shall take responsibility for maintaining adequate and accurate electronic or hard copy source documents of all observations and data generated during this trial. Such documentation is subject to inspection by the sponsor and relevant regulatory agencies. If the investigator withdraws from the trial (e.g., relocation or retirement), all trial related records should be transferred to a mutually agreed upon designee within a sponsor-specified timeframe. Notice of such transfer will be given to the sponsor in writing.

# 10 Quality Control and Quality Assurance

#### 10.1 Monitoring

Otsuka has ethical, legal and scientific obligations to follow this trial in a detailed and orderly manner in accordance with established research principles, the ICH GCP (CPMP/ICH/135/95 and CPMP768/97) guidelines and the principles of the Declaration of Helsinki. As part of a concerted effort to fulfil these obligations (maintain current personal knowledge of the progress of the trial), the monitors will visit the site during the trial, as well as communicate frequently via telephone and written communication(s).

# 10.2 Auditing

Otsuka's Management Unit (or representative) may conduct audits at the trial site. Audits will include, but are not be limited to, adherence to the protocol, drug supply, presence of required documents, the informed consent process, and comparison of CRFs with source documents. The investigator agrees to participate with audits.

Competent Authorities worldwide may inspect the trial site during or after the trial. The investigator should contact Otsuka immediately if this occurs and must fully cooperate with such inspections conducted at a reasonable time in a reasonable manner.

# 11 Ethics and Responsibility

#### 11.1 Ethical Conduct of the Trial

The trial will be conducted in accordance with the trial protocol, the International Conference on Harmonization (ICH) guideline for Good Clinical Practice (GCP) in its current version and the ethical principles laid down in the Declaration of Helsinki. Current national regulations and guidelines will also be followed.

# 11.2 Investigator Obligations

The Investigator agrees to conduct the trial in compliance with the protocol agreed by the Sponsor and, if required, by Competent Authorities (CAs), which was approved by an EC and for which a Clinical Trial Authorization (CTA) has been granted by the CA. The Investigator and the Sponsor should sign the protocol (and protocol amendments) to confirm this agreement.

The EC of the Investigator as well as the CA must review and give approval for the trial as described in this protocol to be conducted in human subjects.

#### 11.3 Ethics Committee and Competent Authority

The trial will be initiated only after written approval from the responsible EC and after obtaining CTA from the CA. The EC should operate according to ICH GCP guidelines and local law. The written EC approval and the names and qualifications of members of the EC must be made available to the Sponsor before the trial can be initiated. The Investigator is responsible for submission(s) to, and communications with, the EC.

This trial protocol (including all substantial amendments) together with the written Informed Consent Form (ICF) and updates thereof, subject recruitment procedures (e.g. advertisements), any other written information to be provided to subjects, and any other documents that the EC may need to fulfil its responsibilities will be submitted for approval to the EC.
The Investigator should submit written reports of the clinical trial status to the EC annually, or more frequently if requested by the EC. A final trial notification should be forwarded by the Sponsor to the EC within 90 days after the trial has been completed or in the event of premature termination of the trial within 15 days.

# 12 Confidentiality

All information generated in this trial will be considered highly confidential and will not be disclosed to any person not directly concerned with the trial without the sponsor's prior written permission. However, officials from Competent Authorities and sponsor personnel (or their representatives) will be allowed full access to inspect and copy the records.

All IMPs, subject bodily fluids, and/or other materials collected shall be used solely in accordance with this protocol, unless otherwise agreed to in writing by Otsuka.

All CRFs as well as all reports and communications relating trial participation will identify each participant only by the participant identification number. The investigator will maintain a current confidential Participant Identification Code List of full names of all participants in this trial. This list will allow the investigator to reveal the identity of the participants in the event that they need to be contacted for safety reasons. This information will be held in the strictest confidence and will only be used for emergency purposes, if needed. The CRF will be used to transmit the information collected in the performance of this trial to Otsuka and to Competent Authorities, as appropriate.

# 13 Amendment Policy

The investigator will not make any changes to this protocol without prior written consent from Otsuka and subsequent approval by the EC and CA. Any permanent change to the protocol, whether it is an overall change or a change for specific trial site(s), must be handled as a protocol amendment. Any amendment to the protocol will be fully discussed by Otsuka (or designee). If agreement is reached regarding the need for an amendment, it will be written by Otsuka (or designee). Each amendment will be submitted to the EC and CA. Except for non-substantial (ie, administrative) amendments, investigators will wait for EC and CA approval of the amended protocol before implementing the change(s). Administrative amendments are defined as having no effect on the safety or physical or mental integrity of the research subjects, the conduct or management of the trial, the scientific value of the trial or the quality or safety of IMP(s)


Version 11.0 2018-03-07

# Protocol 21-13-102

used in the trial. However, a protocol change intended to eliminate an apparent immediate hazard to subjects should be implemented immediately, followed by EC and CA notification within 5 working days. Otsuka or its designee will submit protocol amendments to the competent authorities or other regulatory agencies.

When the EC or CA, the investigators and/or the sponsor conclude that the protocol amendment substantially alters the trial design and/or increases the potential risk to the subject, the currently approved written ICF will require similar modification. In such cases, after the approval of the new ICF by the EC and CA, repeat informed consent will be obtained from subjects in a timely manner before expecting continued participation in the trial.

# 14 References

- 1 Kwon et al., Efficacy and Safety of Combination Antiplatelet Therapies in Patients With Symptomatic Intracranial Atherosclerotic Stenosis, Stroke. 2011; 42:2883-2890; originally published online July 28, 2011;
- 2 Hiatt et al., Long-term safety of cilostazol in patients with peripheral artery disease: The CASTLE trial (Cilostazol: A Trial in Long-term Effects) JOURNAL OF VASCULAR SURGERY Volume 47, Number 2
- 3 Report # 000737 Mutagenicity trial of OPC-13013 by the Ames test.
- 4 Mutagenicity trial of OPC-13013 by the Rec-assay.
- 5 Mutagenicity trial of OPC-13013 by biochemical induction Assay
- 6 Oncogenicity trial in mice.
- 7 OPC-21 Oncogenicity trial in rats.
- 8 Mutagenicity trial of OPC-13013 by bacterial reverse mutation test.
- 9 OPC-21: Mutation at the thymidine kinase (TK) locus of mouse lymphoma L5178Y cells using the microtitre fluctuation technique.
- 10 OPC-21 Induction of chromosome aberration in cultured Chinese hamster ovary (CHO) cells.
- 11 Reevaluation of the effects of OPC-13013 and its main metabolites, OPC-13015 and OPC-13213, on QTc values of dogs and cynomolgus monkeys corrected by various formulas.
- 12 21-98-213 Final Trial Report (FSR): Internal Report Otsuka ("PACE").
- 13 21-98-214 CASTLE trial a blinded, placebo-controlled phase IV trial.
- 14 Trenk D, Hochholzer W, Fromm MF, et al. Cytochrome P450 2C19 681G>A polymorphism and high on-clopidogrel platelet reactivity associated with adverse 1-year clinical outcome of elective percutaneous coronary intervention with drugeluting or bare-metal stents. J Am Coll Cardiol 2008; 51: 1925-34.
- 15 Sanford JC, Guo Y, Sadee W, et al. Regulatory polymorphisms in CYP2C19 affecting hepatic expression. Drug Metabol Drug Interact. 2013;28(1):23-30.
- 16 Scott SA, Sangkuhl K, Stein CM, et al. Clinical Pharmacogenetics Implementation Consortium guidelines for CYP2C19 genotype and clopidogrel therapy: 2013 update. Clin Pharmacol Ther. 2013 Sep;94(3):317-23.

- 17 Mega JL, Simon T, Collet JP, et al. Reduced-function CYP2C19 genotype and risk of adverse clinical outcomes among patients treated with clopidogrel predominantly for PCI: a meta-analysis. JAMA 2010; 304: 1821-30.
- 18 Siller-Matula et al., Thienopyridines in cardiovascular disease: Focus on clopidogrel resistance, Thromb Haemost 2007; 97: 385–393
- Angiolillo, D. J.; Piera Capranzano; Jose Luis Ferreiro; Masafumi Ueno; Davide Capodanno; Kodlipet Dharmashankar; Andrew Darlington; Sabrina Sumner; Bhaloo Desai; Ronald K. Charlton; Lyndon C. Box; Martin M. Zenni; Luis A. Guzman; Theodore A. Bass: Impact of adjunctive cilostazol therapy on platelet function profiles in patients with and without diabetes mellitus on aspirin and clopidogrel therapy. Thromb Haemost 2011; 106: 253–262

# **Appendix 1 Sponsor Drug Safety Contacts**

Report Immediately Reportable Events (serious adverse events, potential Hy's Law cases, pregnancies and adverse events requiring discontinuation of trial drug) to:

Otsuka Europe Development and Commercialisation Ltd. Zweigniederlassung Frankfurt am Main Pharmacovigilance Region Europe Europa-Allee 52 60327 Frankfurt am Main Germany

Phone: +49 69 955044 0

Fax: +49 69 955044 63

Email: Global Intake@otsuka-us.com

In case it is also not possible to submit a safety report by fax the reporter should report by phone.

SAE phone: + 49 172 61 44 932

# **Appendix 2** Institutions Concerned with the Trial

# **Sponsor**

Otsuka Pharmaceutical Co., Ltd. 2-9 Kanda-Tsukasamachi, Chiyoda-ku Tokyo Japan

# **Investigator**



# **Contract Research Organization**

ICON Clinical Research Ltd. South County Business Park Leopardstown Dublin 18 Ireland

# **Investigational Medicinal Product Supplier**



# Protocol 21-13-102

Appendix 3 SmPCs

Cilostazol: FACHINFORMATION - Pletal® 50 mg/100 mg Tabletten

ASA: FACHINFORMATION - Aspirin® protect 100 mg/- 300 mg

Clopidogrel: FACHINFORMATION - Plavix® 75 mg Filmtabletten

# **Investigator Agreement**

I, the undersigned investigator, have read and understand the protocol (including the SmPCs) and agree that it contains all the ethical, legal and scientific information necessary to conduct this trial in accordance with the principles of Good Clinical Practices and as described herein and in the sponsor's (or designee's) Clinical Research Agreement.

I will provide copies of the protocol to all physicians, nurses and other professional personnel to whom I delegate trial responsibilities. I will discuss the protocol with them to ensure that they are sufficiently informed regarding the clinical trial, the concurrent medications, the efficacy and safety parameters and the conduct of the trial in general. I am aware that this protocol must be approved by the Institutional Review Board (IRB) or Ethics Committee (EC) responsible for such matters in the clinical trial facility. I agree to adhere strictly to the attached protocol.

I understand that this IRB- or EC approved protocol will be submitted to the appropriate competent authority/ies by the sponsor. I agree that clinical data entered on case report forms by me and my staff will be utilized by the sponsor in various ways such as for submission to governmental regulatory authorities and/or in combination with clinical data gathered from other research sites, whenever applicable. I agree to allow sponsor monitors and auditors full access to all medical records at the research facility for subjects screened or enrolled in the trial.

I agree to await IRB/EC approval before implementation of any protocol amendments to this protocol. If, however, there is an immediate hazard to subjects, I will implement the amendment immediately, and provide the information to the IRB/EC within 5 working days. Administrative changes to the protocol will be transmitted to the IRB/EC for informational purposes only.

I agree to provide all subjects with informed consent forms, as required by the applicable regulations and by ICH guidelines. I agree to report to the sponsor any adverse events in accordance with the terms of the sponsor's Clinical Research Agreement and the relevant local regulation(s) and guideline(s). I further agree to provide all required information

# Protocol 21-13-102

regarding financial certification or disclosure to the sponsor for all investigators and sub-investigators in accordance with the terms of the relevant regulation(s).

I understand that participation in the protocol involves a commitment to publish the data from this trial in a cooperative publication prior to publication of efficacy and safety results on an individual basis.




Version 11.0 2018-03-07



Pletal<sup>®</sup> 50 mg Tabletten Pletal<sup>®</sup> 100 mg Tabletten

Dieses Arzneimittel unterliegt einer zusätzlichen Überwachung. Dies ermöglicht eine schnelle Identifizierung neuer Erkenntnisse über die Sicherheit. Angehörige von Gesundheitsberufen sind aufgefordert, jeden Verdachtsfall einer Nebenwirkung zu melden. Hinweise zur Meldung von Nebenwirkungen, siehe Abschnitt 4.8.

# 1. BEZEICHNUNG DER ARZNEIMITTEL

Pletal® 50 mg Tabletten Pletal® 100 mg Tabletten

# 2. QUALITATIVE UND QUANTITATIVE ZUSAMMENSETZUNG

- 1 Tablette Pletal® 50 mg enthält 50 mg
- 1 Tablette Pletal® 100 mg enthält 100 mg

Vollständige Auflistung der sonstigen Bestandteile siehe Abschnitt 6.1.

# 3. DARREICHUNGSFORM

Tablette

Pletal® 50 mg

Weiße, runde, abgeflachte Tabletten mit Prägung "OG31" auf einer Seite.

Pletal® 100 mg

Weiße, runde, abgeflachte Tabletten mit Prägung "OG30" auf einer Seite.

#### 4. KLINISCHE ANGABEN

# 4.1 Anwendungsgebiete

Pletal® ist indiziert zur Verlängerung der maximalen und schmerzfreien Gehstrecke bei Patienten mit Claudicatio intermittens, die keinen Ruheschmerz und keine Anzeichen von peripheren Gewebsnekrosen haben (periphere arterielle Verschlusskrankheit Fontaine-Stadium II).

Pletal® 50/100 mg ist zur Second-Line-Therapie bei Patienten indiziert, bei denen eine Lebensstilumstellung (einschließlich Einstellung des Rauchens und körperliches Training [unter Anleitung]) und andere geeignete Interventionen nicht zu einer ausreichenden Verbesserung der Symptome ihrer Claudicatio intermittens führten.

#### 4.2 Dosierung, Art und Dauer der Anwendung

Die empfohlene Dosis Cilostazol beträgt zweimal täglich 100 mg.

Cilostazol sollte jeweils 30 Minuten vor dem Frühstück und dem Abendessen eingenommen werden. Die Einnahme von Cilostazol mit Nahrungsmitteln zeigt einen Anstieg der maximalen Plasmakonzentration (C<sub>max</sub>) von Cilostazol, was mit einem erhöhten Auftreten von unerwünschten Reaktionen verbunden sein kann.

Die Therapie mit Cilostazol sollte von Ärzten eingeleitet werden, die Erfahrung haben mit der Behandlung von Claudicatio intermittens (siehe Abschnitt 4.4).

Der Arzt sollte den Patienten nach 3 Monaten Behandlung erneut untersuchen und die Behandlung mit Cilostazol abbrechen, falls Cilostazol keine angemessene Wirkung zeigt oder sich die Symptome nicht verbesserten.

Die Patienten, die mit Cilostazol behandelt werden, sollten ihre Lebensstilumstellung beibehalten (nicht rauchen und körperliches Training) sowie auch ihre medikamentöse Behandlung (z.B. Lipidsenker und Thrombozytenaggregationshemmer) fortführen, um das Risiko kardiovaskulärer Ereignisse zu reduzieren. Cilostazol ersetzt diese Behandlung nicht.

Eine Reduzierung der Dosis auf 50 mg zweimal täglich wird bei den Patienten empfohlen, die Medikamente mit starker CYP3A4-Hemmung einnehmen, wie z. B. einige Makrolide, Azol-Antimykotika, Protease-Inhibitoren oder Medikamente mit starker CYP2C19-Hemmung, wie z. B. Omeprazol (siehe Abschnitte 4.4 und 4.5).

#### Ältere Patienten

Es gibt keine spezielle Dosierungsanleitung für ältere Patienten.

# Pädiatrische Patienten

Bei Kindern wurden die Sicherheit und Wirksamkeit nicht ermittelt.

# Nierenfunktionsstörungen

Bei Patienten mit einer Kreatininclearance von > 25 ml/min ist keine Dosisanpassung erforderlich.

Cilostazol ist bei Patienten mit einer Kreatininclearance von  $\leq 25$  ml/min kontraindiziert.

# Leberfunktionsstörungen

Bei Patienten mit leichten Lebererkrankungen ist keine Dosisanpassung erforderlich. Es liegen keine Daten von Patienten mit mittelschweren bis schweren Leberfunktionsstörungen vor.

Da Cilostazol weitgehend durch Leberenzyme metabolisiert wird, ist es bei Patienten mit mittelschweren bis schweren Leberfunktionsstörungen kontraindiziert.

# 4.3 Gegenanzeigen

- Bekannte Überempfindlichkeit gegen Cilostazol oder einen der sonstigen Bestandteile,
- schwere Nierenfunktionsstörungen: Kreatininclearance ≤ 25 ml/min,
- mittelschwere oder schwere Leberfunktionsstörungen,
- · kongestive Herzinsuffizienz,
- Schwangerschaft,
- Patienten mit jeder bekannten Veranlagung für Blutungen (z. B. aktives peptisches Ulkus, kurz zurückliegender hämorrhagischer Schlaganfall [innerhalb der letzten 6 Monate], proliferative diabetische Retinopathie, schlecht eingestellte Hypertonie),
- Patienten mit anamnestisch bekannter ventrikulärer Tachykardie, Kammerfilmmern oder multifokalen ventrikulären Ektopien, unabhängig davon, ob adäquat behandelt oder nicht, sowie bei Patienten mit Verlängerung des QTc-Intervalls,
- Patienten mit anamnestisch bekannter schwerer Tachyarrhythmie,
- Patienten, die gleichzeitig zusätzlich mindestens zwei Thrombozytenaggregationshemmer oder Antikoagulanzien erhalten (z. B. Acetylsalicylsäure, Clopidogrel, Heparin, Warfarin, Acenocoumarol, Dabigatran, Rivaroxaban oder Apixaban),

 Patienten mit instabiler Angina pectoris, Myokardinfarkt in den letzten 6 Monaten oder Koronarintervention in den letzten 6 Monaten.

# 4.4 Besondere Warnhinweise und Vorsichtsmaßnahmen für die Anwendung

Ob Cilostazol zur Behandlung geeignet ist, sollte mit anderen Behandlungsoptionen, wie z. B. Revaskularisation, sorgfältig abgewogen werden.

Aufgrund seines Wirkmechanismus kann Cilostazol Tachykardie, Palpitation, Tachyarrhythmie und/oder Hypotonie hervorrufen. Die mit Cilostazol assoziierte Erhöhung der Herzfrequenz beträgt ca. 5 bis 7 bpm (beats per minute); bei Risikopatienten kann dies folglich zu Angina pectoris führen.

Patienten mit einem erhöhten Risiko für schwere unerwünschte kardiale Ereignisse als Folge einer erhöhten Herzfrequenz, z. B. Patienten mit stabiler koronarer Herzkrankheit, sollten während der Behandlung mit Cilostazol engmaschig überwacht werden; hingegen ist der Einsatz von Cilostazol bei Patienten mit instabiler Angina pectoris oder Myokardinfarkt/Koronarintervention in den letzten 6 Monaten oder einer anamnestisch bekannten Tachyarrhythmie kontraindiziert (siehe Abschnitt 4.3).

Vorsicht ist geboten, wenn Cilostazol bei Patienten mit atrialer oder ventrikulärer Ektopie sowie bei Patienten mit Vorhofflimmern oder -flattern verordnet wird.

Die Patienten sind ausdrücklich dazu anzuhalten, jeden Vorfall einer Blutung oder Neigung zu Hämatomen während der Behandlung zu melden. Im Fall einer Netzhatblutung ist die Einnahme von Cilostazol zu beenden. Siehe Abschnitte 4.3 und 4.5 für weitere Informationen bei Blutungen.

Aufgrund der thrombozytenaggregationshemmenden Wirkung von Cilostazol ist bei Operationen ein erhöhtes Blutungsrisiko möglich (auch bei kleineren Eingriffen wie z.B. einer Zahnextraktion). Falls beim Patienten eine Operation geplant ist und eine thrombozytenaggregationshemmende Wirkung nicht erforderlich ist, sollte Cilostazol 5 Tage vor dem Eingriff abgesetzt werden.

Es hat selten bzw. sehr selten Berichte über Blutbildveränderungen einschließlich Thrombozytopenie, Leukopenie, Agranulozytose, Panzytopenie und aplastischer Anämie gegeben (siehe Abschnitt 4.8). Die meisten Patienten erholten sich nach Absetzen von Cilostazol. Jedoch verliefen einige Fälle von Panzytopenie und aplastischer Anämie tödlich.

Die Patienten sind ausdrücklich darauf hinzuweisen, außer Blutungsereignissen und der Neigung zu Hämatomen auch sofort alle anderen Anzeichen zu melden, die auf erste Zeichen einer Blutdyskrasie hinweisen, z. B. Pyrexie oder Halsschmerzen. Ein großes Blutbild sollte erstellt werden, wenn Verdacht auf eine Infektion besteht oder ein anderer klinischer Nachweis einer Blutdyskrasie vorliegt. Cilostazol ist sofort abzusetzen, wenn es klinische oder laborchemische Nachweise für Blutbildveränderungen gibt.

ar 2017

012880-24499

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.

# Pletal<sup>®</sup> 50 mg Tabletten Pletal<sup>®</sup> 100 mg Tabletten



Bei Patienten, die starke CYP3A4- oder CYP2C19-Inhibitoren erhielten, war der Cilostazol-Plasmaspiegel erhöht. Für diesen Fall wird eine Cilostazol-Dosis von 50 mg zweimal täglich empfohlen (siehe Abschnitt 4.5 für weitere Informationen).

Vorsicht ist erforderlich, wenn Cilostazol zusammen mit anderen Substanzen mit Potenzial zur Blutdrucksenkung gegeben wird. Es besteht die Möglichkeit, dass dies einen additiven hypotensiven Effekt mit reflektorischer Tachykardie haben könnte. Siehe auch Abschnitt 4.8.

Vorsicht ist geboten, wenn Cilostazol zusammen mit anderen, die Thrombozytenaggregation hemmenden Substanzen, gegeben wird. Siehe Abschnitte 4.3 und 4.5.

#### 4.5 Wechselwirkungen mit anderen Arzneimitteln und sonstige Wechselwirkungen

Thrombozytenaggregationshemmer

Cilostazol ist ein PDE III-Hemmer mit thrombozytenaggregationshemmender Aktivität. In einer klinischen Studie mit gesunden Probanden führte die Einnahme von 150 mg Cilostazol b.i.d. über 5 Tage nicht zu einer Verlängerung der Blutungszeit.

# Acetylsalicylsäure (ASS)

Verglichen mit der alleinigen Gabe von ASS zeigte die kurzzeitige (≤ 4 Tage) gleichzeitige Anwendung von ASS und Cilostazol eine 23–25%ige Zunahme der Hemmung der ADP-induzierten ex-vivo-Thrombozytenaggegation.

Bei Patienten, die Cilostazol und ASS einnahmen, gab es keine offensichtlichen Trends in Richtung eines vermehrten Auftretens hämorrhagischer Nebenwirkungen im Vergleich zu Patienten, die Placebo und äquivalente Dosen von Aspirin einnahmen.

# Clopidogrel und andere thrombozytenaggregationshemmende Arzneimittel

Die gleichzeitige Gabe von Cilostazol und Clopidogrel hatte keinen Einfluss auf die Thrombozytenzahl, die Prothrombinzeit (PT) und die aktivierte partielle Thromboplastinzeit (aPTT). Alle gesunden Studienteilnehmer zeigten bei alleiniger Behandlung mit Clopidogrel eine verlängerte Blutungszeit. Die gleichzeitige Gabe von Cilostazol führte nicht zu einem signifikanten zusätzlichen Effekt auf die Blutungszeit. Vorsicht ist angeraten, wenn Cilostazol mit anderen Arzneimitteln, die die Thrombozytenaggregation hemmen, gleichzeitig gegeben wird. Eine regelmäßige Überwachung der Blutungszeit ist zu erwägen. Bei Patienten, die mit mindestens zwei Thrombozytenaggregationshemmern/Antikoagulantien behandelt werden, ist die Behandlung mit Cilostazol kontraindiziert (siehe Abschnitt 4.3).

Bei gleichzeitiger Einnahme von Clopidogrel, ASS und Cilostazol kam es in der CASTLE-Studie zu einer Erhöhung der Bluttungsrate.

Orale Antikoagulanzien wie Warfarin In einer klinischen Einzeldosis-Studie konnte keine Hemmung des Metabolismus von Warfarin oder ein Effekt auf die Gerinnungsparameter (PT, aPTT, Blutungszeit) beobachtet werden. Dennoch ist Vorsicht angeraten bei Patienten, die sowohl Cilostazol als auch andere Substanzen mit gerinnungshemmender Wirkung erhalten. Es sollten häufige Kontrollen durchgeführt werden, um die Blutungsgefahr zu reduzieren.

Cytochrom P-450-(CYP-) Enzyminhibitoren Cilostazol wird weitgehend durch CYP Enzyme metabolisiert, insbesondere durch CYP3A4 und CYP2C19, in geringerem Maße durch CYP1A2. Der Dehydro-Metabolit, der eine 4- bis 7-mal größere thrombozytenhemmende Wirkung als Cilostazol hat, scheint primär über CYP3A4 gebildet zu werden. Der 4'-trans-Hydroxy-Metabolit mit einem Fünftel der Potenz von Cilostazol wird anscheinend hauptsächlich über CYP2C19 gebildet. Daher erhöhen Arzneimittel mit Hemmwirkung auf CYP3A4 (z. B. manche Makrolide, Azol-Antimykotika, Protease-Inhibitoren) oder CYP2C19 (wie Protonenpumpenhemmer, PPI) die pharmakologische Gesamtaktivität von Cilostazol und können die unerwünschten Wirkungen vor Cilostazol verstärken. Aus diesem Grund beträgt die empfohlene Dosis für Patienten. die starke CYP3A4- oder CYP2C19-Inhibitoren einnehmen, 50 mg zweimal täglich (siehe Abschnitt 4.2).

Die Gabe von Cilostazol in Kombination mit Erythromycin (ein CYP3A4-Inhibitor) führte zu einem Anstieg der AUC von Cilostazol um 72%, begleitet von einem 6% igen Abfall der AUC des Dehydro-Metaboliten und einem 119%igen Anstieg der AUC des 4'-trans-Hydroxy-Metaboliten.

Auf der Basis der AUC steigt die pharmakologische Gesamtaktivität von Cilostazol um 34 %, wenn es in Kombination mit Erythromycin gegeben wird. Basierend auf diesen Daten beträgt die empfohlene Dosis von Cilostazol 50 mg zweimal täglich, wenn es in Kombination mit Erythromycin und ähnlichen Substanzen (z. B. Clarithromycin) gegeben wird.

Die gleichzeitige Gabe von Ketoconazol (ein Inhibitor von CYP3A4) und Cilostazol 100 mg führte zu einem Anstieg der AUC von Cilostazol um 117%, begleitet von einer Senkung der AUC des Dehydro-Metaboliten um 15% und einem Anstieg der AUC des 4'-trans-Hydroxy-Metaboliten um 87%. Auf der Basis der AUC steigt die pharmakologische Gesamtaktivität von Cilostazol um 35 %, wenn es in Kombination mit Ketoconazol gegeben wird. Basierend auf diesen Daten beträgt die empfohlene Dosis von Cilostazol 50 mg zweimal täglich, wenn es in Kombination mit Ketoconazol und ähnlichen Substanzen (z. B. Itraconazol) gegeben wird

Die Verabreichung von Cilostazol zusammen mit Diltiazem (einem schwachen CYP3A4-Inhibitor) führte zu einem Anstieg der AUC von Cilostazol von 44 %, begleitet von einem 4 %igen Anstieg in der AUC des Dehydro-Metaboliten und einem 43 %igen Anstieg der AUC des 4'-trans-Hydroxy-Metaboliten. Basierend auf diesen Daten ist keine Dosisanpassung erforderlich.

Die Einnahme einer Einzeldosis von 100 mg Cilostazol mit 240 ml Grapefruitsaft (ein Inhibitor des intestinalen CYP3A4) hatte keinen nennenswerten Einfluss auf die Pharmakokinetik von Cilostazol. Basierend auf diesen Daten ist keine Dosisanpassung erforderlich. Ein klinisch bedeutsamer Effekt auf Cilostazol ist jedoch bei größeren Mengen Grapefruitsaft durchaus möglich.

Die Einnahme von Cilostazol mit Omeprazol (ein CYP2C19-Inhibitor) vergrößerte die AUC von Cilostazol um 22%, begleitet von einer Vergrößerung der AUC des Dehydro-Metaboliten um 68% und einer Abnahme der AUC des 4'-trans-Hydroxy-Metaboliten um 36%. Auf der Basis der AUC steigt die pharmakologische Gesamtaktivität von Cilostazol um 47%, wenn es in Kombination mit Omeprazol gegeben wird. Basierend auf diesen Daten beträgt die empfohlene Dosis von Cilostazol 50 mg zweimal täglich, wenn es in Kombination mit Omeprazol gegeben wird.

# Cytochrom P-450-Enzymsubstrate

Es konnte gezeigt werden, dass Cilostazol die AUC für Lovastatin (für CYP3A4 empfindliches Substrat) und seiner β-Hydroxysäure um 70 % erhöht. Vorsicht ist geboten bei gleichzeitiger Gabe von Cilostazol und CYP3A4-Substraten mit enger therapeutischer Breite (z.B. Cisaprid, Halofantrin, Pimozid, Ergotderivate). Vorsicht ist geboten bei gleichzeitiger Gabe von Statinen, die von CYP3A4 metabolisiert werden, wie z.B. Simvastatin, Atorvastatin und Lovastatin

# Induktoren von Cytochrom P-450

Die Wirkung von CYP3A4- und CYP2C19-Induktoren (z. B. Carbamazepin, Phenytoin, Rifampicin und Johanniskraut) auf die Pharmakokinetik von Cilostazol wurde nicht untersucht. Da es theoretisch zu einer Änderung der thrombozytenaggregationshemmenden Wirkung kommen kann, sollte diese bei Gabe von Cilostazol zusammen mit CYP3A4- und CYP2C19-Induktoren sorgfältig überwacht werden.

In klinischen Prüfungen reduzierte Rauchen (CYP1A2 induzierend) die Plasmakonzentration von Cilostazol um 18 %.

Weitere potenzielle Wechselwirkungen Vorsicht ist geboten bei gleichzeitiger Gabe von Cilostazol und Substanzen, die blutdrucksenkend wirken können, weil es dadurch zu einem additiven hypotensiven Effekt mit reflektorischer Tachykardie kommen

### 4.6 Fertilität, Schwangerschaft und Stillzeit

# Schwangerschaft

Es liegen keine hinreichenden Daten für die Verwendung von Cilostazol bei Schwangeren vor. Tierexperimentelle Studien haben Reproduktionstoxizität gezeigt (siehe Abschnitt 5.3). Über das potenzielle Risiko beim Menschen liegen keine Erkenntnisse vor. Pletal® darf während der Schwangerschaft nicht angewendet werden (siehe Abschnitt 4.3).

# Stillzeit

In Tierstudien wurde gezeigt, dass Cilostazol in die Muttermilch übergeht. Es ist nicht bekannt, ob Cilostazol in die Muttermilch ausgeschieden wird. Aufgrund der potenziell schädigenden Effekte bei Neugeborenen, die von einer behandelten Mutter ge-

012880-24499



Pletal<sup>®</sup> 50 mg Tabletten Pletal<sup>®</sup> 100 mg Tabletten

stillt werden, wird die Anwendung von Pletal<sup>®</sup> während der Stillzeit nicht empfohlen.

#### Fertilität

Cilostazol hat die Fertilität weiblicher Mäuse reversibel beeinträchtigt, bei anderen Tierspezies trat dies aber nicht auf (siehe Abschnitt 5.3). Die klinische Signifikanz ist unbekannt.

#### 4.7 Auswirkungen auf die Verkehrstüchtigkeit und die Fähigkeit zum Bedienen von Maschinen

Cilostazol kann Schwindel verursachen. Patienten sollten daher gewarnt werden, Vorsicht walten zu lassen, ehe sie fahren oder Maschinen bedienen.

#### 4.8 Nebenwirkungen

Die in klinischen Studien am häufigsten berichteten Nebenwirkungen waren Kopfschmerzen (> 30 %), Diarrhoe und Stuhlweränderungen (jeweils > 15 %). Diese Reaktionen waren üblicherweise von leichter bis mittlerer Intensität und wurden durch Dosisreduktion gelegentlich abgemildert.

Die nebenstehende Tabelle enthält Nebenwirkungen, die in klinischen Prüfungen und nach der Markteinführung berichtet wurden.

Die Häufigkeitsangaben sind wie folgt definiert:

Sehr häufig (≥ 1/10)
Häufig (≥ 1/100, < 1/10)
Gelegentlich (≥ 1/1.000, < 1/100)
Selten (≥ 1/10.000, < 1/1.000)
Sehr selten (< 1/10.000)

Unbekannt (lässt sich anhand der vorhandenen Daten nicht abschätzbar)

Die Häufigkeit der nach der Markteinführung beobachteten Nebenwirkungen wird als unbekannt angegeben (Häufigkeit auf Grundlage der verfügbaren Daten nicht abschätzbar).

# Siehe Tabelle

Eine Zunahme der Häufigkeit von Palpitationen und peripheren Ödemen wurde beobachtet, wenn Cilostazol gleichzeitig mit anderen, eine reflektorische Tachykardie verursachenden Vasodilatatoren verabreicht wurde, zum Beispiel Calciumkanalblocker vom Dihydropyridin-Tyo.

Kopfschmerz war das einzige unerwünschte Ereignis, das bei ≥ 3 % der mit Cilostazol behandelten Patienten zum Therapieabruch führte. Andere häufige Gründe eines Therapieabbruchs beinhalteten Palpitationen und Diarrhoe (beide 1,1%).

Cilostazol per se kann zu einem erhöhten Blutungsrisiko führen. Dieses Risiko kann verstärkt werden, wenn Cilostazol zusammen mit einem anderen Wirkstoff mit einem solchen Potenzial eingenommen wird.

Das Risiko intraokulärer Blutungen kann bei Patienten mit Diabetes höher sein.

Eine Zunahme der Häufigkeit von Diarrhoe und Palpitationen wurde bei den über 70-jährigen Patienten beobachtet.

| 012880-24499 |
|--------------|

2017

| Erkrankungen des Blutes und<br>des Lymphsystems | Häufig:<br>Gelegentlich:<br>Selten:<br>Unbekannt: | Verlängerte Blutungszeit, Thrombozythämie |
|---|---|---|
| Erkrankungen des Immunsystems | Gelegentlich: | Allergische Reaktion |
| Stoffwechsel- und | Häufig: | Ödem (peripher, Gesicht), Anorexie |
| Ernährungsstörungen | | Hyperglykämie, Diabetes mellitus |
| Psychiatrische Erkrankungen | Gelegentlich: | Angstzustände |
| Erkrankungen des Nervensystems | Häufig: | Kopfschmerzen<br>Schwindel<br>Schlaflosigkeit, abnorme Träume |
| Augenerkrankungen | Unbekannt: | Konjunktivitis |
| Erkrankungen des Ohrs und des Labyrinths | Unbekannt: | Tinnitus |
| Herzerkrankungen | Häufig:<br>Gelegentlich: | Palpitationen, Tachykardie, Angina pectoris, Arrhythmien, ventrikuläre Extrasystole Myokardinfarkt, Vorhofflimmern, konges tive Herzinsuffizienz, supraventrikuläre Tachykardie, ventrikuläre Tachykardie, Synkope |
| Gefäßerkrankungen | Gelegentlich:<br>Unbekannt: | Augenblutung, Epistaxis, gastrointestinale<br>Blutung, unspezifische Blutung, orthosta-<br>tische Hypotonie<br>Hitzewallung, Hypertonie, Hypotonie,<br>zerebrale Blutung, Lungenblutung, Mus-<br>kelblutung, Atemwegsblutung, subkutane<br>Blutung |
| Erkrankungen der Atemwege,<br>des Brustraums und Mediastinums | Häufig:<br>Gelegentlich:<br>Unbekannt: | Rhinitis, Pharyngitis Dyspnoe, Pneumonie, Husten Interstitielle Pneumonie |
| Erkrankungen des<br>Gastrointestinaltrakts | Sehr häufig:<br>Häufig:<br>Gelegentlich: | Diarrhoe, Stuhlveränderungen<br>Übelkeit und Erbrechen, Dyspepsie, Flatu<br>lenz, abdominale Schmerzen<br>Gastritis |
| Leber- und Gallenerkrankungen | Unbekannt: | Hepatitis, abnorme Leberfunktion, Ikterus |
| Erkrankungen der Haut und<br>des Unterhautzellgewebes | Häufig:<br>Unbekannt: | Hautausschlag, Juckreiz<br>Ekzem, Hautausschläge, Stevens-John-<br>son-Syndrom, toxische epidermale Nekro<br>lyse, Urtikaria |
| Skelettmuskulatur-, Bindegewebs-<br>und Knochenerkrankungen | Gelegentlich: | Myalgie |
| Erkrankungen der Niere und<br>Harnwege | Selten: | Nierenversagen, Einschränkung der Nierenfunktion |
| | Unbekannt: | Hämaturie, erhöhte Miktionsfrequenz |
| Allgemeine Erkrankungen und<br>Beschwerden am Verabreichungsort | Häufig:<br>Gelegentlich:<br>Unbekannt: | Brustschmerzen, Asthenie<br>Schüttelfrost, Unwohlsein<br>Pyrexia, Schmerzen |
| Untersuchungen | Unbekannt: | Erhöhte Harnsäurespiegel, erhöhter BUN, erhöhtes Blutkreatinin |

# Meldung des Verdachts auf Nebenwirkungen

Die Meldung des Verdachts auf Nebenwirkungen nach der Zulassung ist von großer Wichtigkeit. Sie ermöglicht eine kontinuierliche Überwachung des Nutzen-Risiko-Verhältnisses des Arzneimittels. Angehörige von Gesundheitsberufen sind aufgefordert, jeden Verdachtsfall einer Nebenwirkung dem Bundesinstitut für Arzneimittel und Medizinprodukte, Abt. Pharmakovigilanz, Kurt-Georg-Kiesinger-Allee 3, D-53175 Bonn, Website: www.bfarm.de anzuzeigen.

# 4.9 Überdosierung

Informationen über eine akute Überdosierung beim Menschen sind begrenzt. Die zu erwartenden Anzeichen und Symptome sind voraussichtlich starke Kopfschmerzen, Diarrhoe, Tachykardie und möglicherweise kardiale Arrhythmien.

Die Patienten sollten beobachtet und mit einer unterstützenden Therapie behandelt werden. Der Magen sollte, soweit erforderlich, durch induziertes Erbrechen oder Magenspülung entleert werden.

3

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.

# Pletal<sup>®</sup> 50 mg Tabletten Pletal<sup>®</sup> 100 mg Tabletten



#### 5. PHARMAKOLOGISCHE EIGEN-SCHAFTEN

#### 5.1 Pharmakodynamische Eigenschaften

Pharmakotherapeutische Gruppe: Antithrombotische Mittel, Thrombozytenaggregationshemmer, exkl. Heparin; ATC-Code: B01AC

Daten aus neun Placebo-kontrollierten Studien (in denen 1634 Patienten Cilostazol erhielten) haben gezeigt, dass Cilostazol die Bewegungskapazität verbessert, gemessen anhand von Änderungen der Absolute Claudication Distance (ACD, oder maximale Gehstrecke) und der Initial Claudication Distance (ICD, oder schmerzfreie Gehstrecke) auf dem Laufband. Nach 24 Wochen Behandlung mit Cilostazol 100 mg zweimal täglich reichte die mittlere Zunahme der ACD von 60,4–129,1 Meter, während die mittlere ICD-Steigerung von 47,3–93,6 Metern reichte.

Eine auf gewichteten mittleren Unterschieden basierende Meta-Analyse der 9 Studien zeigte für Cilostazol 100 mg zweimal täglich eine signifikante, gegenüber dem Ausgangswert zu verzeichnende absolute Zunahme der maximalen Gehstrecke (ACD) von 42 m, bezogen auf die Zunahme unter Placebo. Dies entspricht einer relativen Verbesserung von 100 % gegenüber Placebo. Dieser Effekt war bei Diabetikern geringer als bei Nicht-Diabetikern.

Tierstudien haben gezeigt, dass Cilostazol vasodilatatorische Eigenschaften besitzt. Dies konnte in kleinen Studien beim Menschen belegt werden, in denen der Blutfluss am Knöchel mittels Strain-Gauge Plethysmographie gemessen wurde. Cilostazol hemmt auch die Proliferation der glatten Muskelzellen bei Ratten und die menschlichen glatten Muskelzellen in vitro. Des Weiteren wird die thrombozytäre Freisetzungsreaktion von Plättchenwachstumsfaktor (Platelet-Derived Growth Factor) und Plättchenfaktor 4 (PF-4) bei humanen Thrombozyten gehemmt.

Studien an Tieren und Menschen (in vivo und ex vivo) haben gezeigt, dass Cilostazol eine reversible Hemmung der Thrombozytenaggregation bewirkt. Die Hemmung ist wirksam gegen eine Reihe von Aggreganzien (einschließlich Scherkräfte, Arachidonsäure, Kollagen, ADP und Adrenalin). Beim Menschen dauert die Hemmung bis zu 12 Stunden an. Nach Beendigung der Cilostazolgabe erfolgte innerhalb von 48-96 Stunden die Wiederherstellung der Aggregation ohne Rebound-Hyperaggregabilität. Bei Patienten wurden während der Anwendung von Pletal® die Auswirkungen auf zirkulierende Plasmalipide untersucht. Nach 12 Wochen bewirkte Pletal® 100 mg zweimal täglich im Vergleich zu Placebo eine Reduzierung der Triglyceride um 0,33 mmol/l (15%) und einen Anstieg des HDL-Cholesterins um 0,10 mmol/l (10%).

Zur Untersuchung der Langzeitwirkung von Cilostazol wurde eine randomisierte doppelblinde Placebo-kontrollierte Phase IV-Studie durchgeführt, deren Fokus Sterblichkeit und Sicherheit waren. Insgesamt wurden 1439 Patienten mit Claudicatio intermittens und ohne Herzschwäche bis zu

3 Jahren mit Cilostazol oder Placebo behandelt. Bezogen auf die Sterblichkeit betrug die über 36 Monate beobachtete Ereignisrate (Kaplan-Meier) für Todesfälle unter der Studienmedikation mit einer medianen Behandlungsdauer von 18 Monaten für Cilostazol 5,6 % (95 % Konfidenzintervall 2,8 bis 8,4 %) und für Placebo 6,8 % (95 % Konfidenzintervall 1,9 bis 11,5 %). Langzeitbehandlung mit Cilostazol führte nicht zu Sicherheitsbedenken.

# 5.2 Pharmakokinetische Eigenschaften

Bei Patienten mit peripheren Durchblutungsstörungen wurde nach Mehrfachgabe von Cilostazol 100 mg zweimal täglich innerhalb von 4 Tagen ein Steady State erreicht.

Mit steigenden Dosierungen nimmt die C<sub>max</sub> von Cilostazol und seinen zirkulierenden Primärmetaboliten unterproportional zu. Die AUC von Cilostazol und seinen Metaboliten jedoch nimmt ungefähr proportional mit der Dosis zu

Die sichtbare Eliminations-Halbwertszeit von Gilostazol beträgt 10,5 Stunden. Es gibt zwei Hauptmetaboliten, ein Dehydro-Cilostazol und ein 4'-trans-Hydroxy-Gilostazol, die beide ähnliche sichtbare Eliminations-Halbwertszeiten haben. Der Dehydro-Metabolit ist ein 4- bis 7-mal wirksamerer Blutplättchenaggregationshemmer als die Ausgangssubstanz, der 4'-trans-Hydroxy-Metabolit ist ein Fünftel so wirksam. Die Plasmakonzentrationen (gemessen über die AUC) der Dehydro- und 4'-trans-Hydroxy-Metaboliten betragen etwa 41 % bzw. 12 % der Gilostazol-Konzentration.

Cilostazol wird hauptsächlich durch Metabolismus eliminiert und die Metaboliten werden anschließend im Urin ausgeschieden. Die in den Metabolismus involvierten primären Isoenzyme sind Cytochrom P-450 CYP3A4, in geringerem Ausmaß CYP2C19 und in einem noch geringeren Ausmaß CYP1A2.

Die Elimination erfolgt hauptsächlich über den Urin (74%), der Rest wird über die Fäzes ausgeschieden. Eine nicht messbare Menge von unverändertem Cilostazol wird mit dem Urin ausgeschieden und weniger als 2% der Dosis wird als Metabolit Dehydro-Cilostazol ausgeschieden. Ungefähr 30% der Dosis wird als 4'-trans-Hydroxy-Metabolit im Urin ausgeschieden. Der Rest wird als Metaboliten ausgeschieden, von denen keiner mehr als 5% der ausgeschiedenen Gesamtmenge ausmacht.

Cilostazol ist zu 95–98% proteingebunden, überwiegend an Albumin. Der Dehydro-Metabolit und der 4'-trans-Hydroxy-Metabolit sind zu 97,4% beziehungsweise 66% proteingebunden.

Es gibt keinen Beleg, dass Cilostazol hepatische mikrosomale Enzyme induziert.

Alter und Geschlecht hatten keinen signifikanten Einfluss auf die Pharmakokinetik von Cilostazol und seine Metaboliten bei gesunden Probanden zwischen 50–80 Jahren.

Bei Patienten mit schweren Nierenfunktionsstörungen war der freie Anteil von Cilostazol 27 % höher und  $C_{\text{max}}$  und AUC waren 29 % beziehungsweise 39 % nied-

riger als bei Patienten mit normaler Nierenfunktion. C<sub>max</sub> und AUC des Dehydro-Metaboliten waren bei Patienten mit schweren Nierenfunktionsstörungen um 41 % beziehungsweise 47 % niedriger als bei Patienten mit normaler Nierenfunktion. C<sub>max</sub> und AUC des 4'-trans-Hydroxy-Metaboliten waren bei Patienten mit schweren Nierenfunktionsstörungen um 173 % beziehungsweise um 209 % höher. Das Arzneimittel darf bei Patienten mit einer Kreatininclearance < 25 ml/min nicht angewendet werden (siehe Abschnitt 4.3).

Es gibt keine Daten von Patienten mit mittelschwerer bis schwerer Leberfunktionsstörung. Da Cilostazol weitgehend von Leberenzymen metabolisiert wird, darf dieses Arzneimittel nicht von diesen Patienten eingenommen werden (siehe Abschnitt 4.3).

#### 5.3 Präklinische Daten zur Sicherheit

Cilostazol und mehrere seiner Metaboliten sind Phosphodiesterase 3-Inhibitoren, die den Abbau des zyklischen AMP hemmen, was zu einer Erhöhung des cAMP-Spiegels in verschiedenen Geweben, einschliesslich Thrombozyten und Blutgefässe, führt. Wie andere positiv inotrope und vasodilatatorische Substanzen produziert Cilostazol bei Hunden kardiovaskuläre Läsionen. Diese Läsionen wurden bei Ratten oder Affen nicht gesehen und werden als speziesspezifisch angesehen. Die Untersuchung des QTc-Intervalls bei Hunden und Affen zeigte nach Verabreichung von Cilostazol oder seiner Metaboliten keine Verlängerung.

Mutagenitätsstudien waren negativ bei Genmutationen von Bakterien, bakterieller DNS Reparatur, Genmutation von Säugetierzellen und *in-vivo*-Chromosomenaberrationstests am Knochenmark der Maus. Bei *in-vitro*-Tests an Keimzellen des chinesischen Hamsters führte Cilostazol zu einem schwachen aber signifikanten Anstieg der Häufigkeit einer Chromosomenaberration. 2-Jahres-Kanzerogenitätsstudien mit oraler Gabe (über Nahrung) wurden bei Ratten mit Dosen bis zu 500 mg/kg/Tag und bei Mäusen mit Dosen von bis zu 1000 mg/kg/Tag durchgeführt. Es gab keine ungewöhnlichen neoplastischen Befunde in diesen Studien.

Feten von Ratten, die während der Tragezeit Cilostazol erhielten, hatten ein vermindertes Gewicht. Zusätzlich wurde im Hochdosisbereich ein Anstieg an äußerlichen, viszeralen und skeletalen Missbildungen bei den Föten beobachtet. Bei niedrigeren Dosierungen wurde eine Verzögerung der Ossiffikation beobachtet. Die Exposition in der Spätschwangerschaft führte zu einem erhöhten Auftretensraten an Totgeburten und einem geringerem Gewicht der Nachkommen. Bei Kaninchen wurde vermehrt eine verzögerte Ossifikation des Brustbeins beobachtet.

Cilostazol inhibiert in vitro die Reifung der Oozyten von Mäusen und löste bei weiblichen Mäusen eine Beeinträchtigung der Fertilität aus. Bei Ratten oder nicht-menschlichen Primaten wurden keine Auswirkungen auf die Fertilität festgestellt. Die Relevanz für Menschen ist unbekannt.

012880-24499



Pletal® 50 mg Tabletten Pletal® 100 mg Tabletten

#### 6. PHARMAZEUTISCHE ANGABEN

# 6.1 Liste der sonstigen Bestandteile

Maisstärke, mikrokristalline Cellulose, Carmellose-Calcium, Hypromellose, Magnesiumstearat.

### 6.2 Inkompatibilitäten

Nicht zutreffend.

# 6.3 Dauer der Haltbarkeit

3 Jahre

#### 6.4 Besondere Vorsichtsmaßnahmen für die Aufbewahrung

Für dieses Arzneimittel sind keine besonderen Lagerungsbedingungen erforderlich.

# 6.5 Art und Inhalt des Behältnisses

Packungen mit 14, 20, 28, 30, 50, 56, 98, 100, 112 oder 168 Tabletten und Klinikpackungen mit 70 (5 x 14) Tabletten in PVC/Aluminium-Blisterpackungen.

Es werden möglicherweise nicht alle Packungsgrößen in Verkehr gebracht.

# 6.6 Besondere Vorsichtsmaßnahmen für die Beseitigung

Keine besonderen Anforderungen.

# 7. INHABER DER ZULASSUNGEN

Otsuka Pharmaceutical Europe Ltd. Gallions, Wexham Springs Framewood Road Wexham SL3 6PJ Vereinigtes Königreich

Mitvertrieb

Otsuka Pharma GmbH Friedrichstr. 2-6 60323 Frankfurt am Main Deutschland

Telefon: 069 170086-0 Telefax: 069 170086-50

# 8. ZULASSUNGSNUMMERN

Pletal® 50 mg: 66599.00.00 Pletal® 100 mg: 66599.01.00

### 9. DATUM DER ERTEILUNG DER ZULASSUNGEN/VERLÄNGERUNG DER ZULASSUNGEN

05.12.2006

# 10. STAND DER INFORMATION

Januar 2017

# 11. VERKAUFSABGRENZUNG

Verschreibungspflichtig

Zentrale Anforderung an:

Rote Liste Service GmbH

Fachinfo-Service

Mainzer Landstraße 55 60329 Frankfurt

012880-24499

2017

5

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.



# Aspirin® protect 100 mg/- 300 mg

#### 1. BEZEICHNUNG DES ARZNEIMITTELS

### Aspirin® protect 100 mg Aspirin® protect 300 mg

Magensaftresistente Tablette Acetylsalicyl-

#### 2. QUALITATIVE UND QUANTITATIVE ZUSAMMENSETZUNG

1 magensaftresistente Tablette enthält: 100 mg Acetylsalicylsäure (Ph. Eur.) 1 magensaftresistente Tablette enthält: 300 mg Acetylsalicylsäure (Ph. Eur.)

Vollständige Auflistung der sonstigen Bestandteile siehe Abschnitt 6.1.

#### 3. DARREICHUNGSFORM

Magensaftresistente Tablette

# 4. KLINISCHE ANGABEN

# 4.1 Anwendungsgebiete

### Aspirin protect 100 mg

- instabile Angina pectoris als Teil der Standardtherapie
- akuter Myokardinfarkt als Teil der Stan-
- Reinfarktprophylaxe
- nach arteriellen gefäßchirurgischen oder interventionellen Eingriffen (z.B. nach ACVB, bei PTCA),
- zur Vorbeugung von transitorischen ischämischen Attacken (TIA) und
- Hirninfarkten, nachdem Vorläuferstadien aufgetreten sind.
- Kawasaki-Syndrom:
  - zur Entzündungshemmung für die Dauer der febrilen Phase
- zur prophylaktischen Thrombozytenaggregationshemmung bei koronararteriellen Aneurysmen

# Hinweis:

Aspirin protect 100 mg eignet sich auf Grund seines Wirkstoffgehaltes nicht zur Behandlung von Schmerzzuständen.

# Aspirin protect 300 mg

Zur Reinfarktprophylaxe.

Aspirin protect 300 mg ist nicht zur Behandlung von Schmerzzuständen vorgese-

# 4.2 Dosierung und Art der Anwendung

# Dosierung

# Bei instabiler Angina Pectoris

Es wird eine Tagesdosis von 1 magensaftresistenten Tablette Aspirin protect 100 mg (entsprechend 100 mg Acetylsalicylsäure pro Tag) empfohlen.

# Bei akutem Myokardinfarkt

Es wird eine Tagesdosis von 1 magensaftresistenten Tablette Aspirin protect 100 mg (entsprechend 100 mg Acetylsalicylsäure pro Tag) empfohlen.

# Zur Reinfarktprophylaxe

Es wird eine Tagesdosis von 3 magensaftresistenten Tabletten Aspirin protect 100 mg (entsprechend 300 mg Acetylsalicylsäure pro Tag) empfohlen.

001915-27444

#### Nach arteriellen gefäßchirurgischen oder interventionellen Eingriffen (z.B. nach ACVB, bei PTCA)

Es wird eine Tagesdosis von 1 magensaftresistenten Tablette Aspirin protect 100 mg (entsprechend 100 mg Acetylsalicylsäure pro Tag) empfohlen.

Der günstigste Zeitpunkt für den Beginn der Behandlung mit Aspirin protect 100 mg nach aortokoronarem Venen-Bypass (ACVB) scheint 24 Stunden nach der Operation zu

Zur Vorbeugung von transitorischen ischämischen Attacken (TIA) und Hirninfarkten, nachdem Vorläuferstadien aufgetreten sind

Es wird eine Tagesdosis von 1 magensaftresistenten Tablette Aspirin protect 100 mg (entsprechend 100 mg Acetylsalicylsäure pro Tag) empfohlen.

# Kawasaki-Syndrom

# Hemmung der Entzündung für die Dauer der febrilen Phase:

Die Behandlung sollte initial mit Acetylsalicylsäure in einer Dosierung von 80-100 mg/kg KG /Tag, verteilt auf 4 Einzeldosen, kombiniert mit Immunglobulinen, begonnen werden.

### Prophylaktische Hemmung der Thrombozytenaggregation bei koronararteriellen Aneurysmen:

Später (ab der 2.-3. Krankheitswoche) sollte die Behandlung mit Acetylsalicylsäure in einer Dosierung von 3-5 mg/kg KG/Tag fortgesetzt werden.

# Aspirin protect 300 mg:

# Zur Reinfarktprophylaxe

Es wird eine Tagesdosis von 1 magensaftresistenten Tablette Aspirin protect 300 mg (entsprechend 300 mg Acetylsalicylsäure pro Tag) empfohlen.

# Art der Anwendung

Die magensaftresistenten Tabletten sollen möglichst mindestens 30 min vor der Mahlzeit mit reichlich Wasser) eingenommen werden

Magensaftresistente Tabletten sollten nicht zerkleinert, zerbrochen oder gekaut werden, um die Freisetzung im alkalischen Milieu des Darms zu gewährleisten.

Zur Behandlung bei akutem Myokardinfarkt sollte die 1. Tablette zerbissen oder zerkaut

Aspirin protect 100 mg/-300 mg ist zur längerfristigen Anwendung vorgesehen. Über die Dauer der Anwendung entscheidet der behandelnde Arzt.

# 4.3 Gegenanzeigen

Aspirin protect 100 mg/-300 mg darf nicht angewendet werden:

- bei Überempfindlichkeit gegen Acetylsalicylsäure, andere Salicylate oder einen der in Abschnitt 6.1 genannten sonstigen Bestandteile
- bei Asthmaanfällen in der Vergangenheit, die durch die Verabreichung von Salicylaten oder Substanzen mit ähnlicher Wirkung, insbesondere nichtsteroidalen Antiphlogistika ausgelöst wurden
- bei akuten gastrointestinalen Ulzera
- bei hämorrhagischer Diathese

- bei Leber- und Nierenversagen
- bei schwerer, nicht eingestellter Herzinsuffizienz
- in Kombination mit Methotrexat in einer Dosierung von 15 mg oder mehr pro Woche (siehe Abschnitt 4.5)
- im letzten Trimenon der Schwangerschaft in einer Dosierung oberhalb von 150 mg Acetylsalicylsäure/Tag (siehe Abschnitt 4.6).

# 4.4 Besondere Warnhinweise und Vorsichtsmaßnahmen für die Anwendung

Eine besonders sorgfältige ärztliche Überwachung ist erforderlich:

- bei Überempfindlichkeit gegen andere Analgetika/Antiphlogistika/Antirheumatika oder gegen andere allergene Stoffe (siehe Abschnitt 4 3)
- bei der gleichzeitigen Einnahme von einigen nichtsteroidalen Antirheumatika (NSARs). wie zum Beispiel Ibuprofen und Naproxen. Diese können den plättchenhemmenden Effekt der Acetylsalicylsäure abschwächen. Patienten sollte angeraten werden, mit Ihrem Arzt zu sprechen, falls sie Acetylsalicylsäure einnehmen und vorhaben NSARs einzunehmen (siehe Abschnitt 4.5)
- bei Bestehen von anderen Allergien (z. B. mit Hautreaktionen, Juckreiz, Nesselfieber)
- bei Asthma bronchiale. Heuschnupfen. Nasenschleimhautschwellungen (Nasenpolypen) oder chronischen Atemwegserkrankungen
- bei gleichzeitiger Therapie mit Antikoagulantien
- bei gastrointestinalen Ulzera oder -Blutungen in der Anamnese
- bei Patienten mit eingeschränkter Leber-
- bei Patienten mit eingeschränkter Nierenfunktion oder mit verminderter kardiovaskulärer Durchblutung (z.B. renale Gefäßerkrankung, kongestive Herzinsuffizienz, Volumenverlust, größere Operationen, Sepsis oder schwere Blutungsereignisse): Acetylsalicylsäure kann das Risiko einer Nierenfunktionsstörung und eines akuten Nierenversagens weiter erhöhen
- vor Operationen (auch bei kleineren Eingriffen wie z.B. Zahnextraktionen): es kann zu verstärkter Blutungsneigung kommen
- bei Patienten mit schwerem Glukose-6-Phosphat-Dehydrogenasemangel: Acetylsalicylsäure kann eine Hämolyse oder eine hämolytische Anämie induzieren. Das Risiko einer Hämolyse kann durch Faktoren wie z.B. hohe Dosierung, Fieber oder akute Infektionen erhöht werden.

# Worauf müssen Sie noch achten?

Acetylsalicylsäure vermindert in niedriger Dosierung die Harnsäureausscheidung. Bei entsprechend gefährdeten Patienten kann dies unter Umständen einen Gichtanfall auslösen

# Kinder und Jugendliche

Aspirin protect 100 mg/-300 mg soll bei Kindern und Jugendlichen mit fieberhaften Erkrankungen nur auf ärztliche Anweisung und nur dann angewendet werden, wenn andere Maßnahmen nicht wirken. Sollte es bei diesen Erkrankungen zu lang anhaltendem Erbrechen kommen, so kann dies ein

G656

# Aspirin® protect 100 mg/- 300 mg



Zeichen des Reye-Syndroms, einer sehr seltenen, aber lebensbedrohlichen Krankheit sein, die unbedingt sofortiger ärztlicher Behandlung bedarf.

Acetylsalicylsäure-haltige Arzneimittel sollen längere Zeit oder in höheren Dosen nicht ohne Befragen des Arztes angewendet werden.

#### 4.5 Wechselwirkungen mit anderen Arzneimitteln und sonstige Wechselwirkungen

Verstärkung der Wirkung bis hin zu erhöhtem Nebenwirkungsrisiko:

- Antikoagulantien/Thrombolytika: Acetylsallicylsäure kann das Blutungsrisiko erhöhen, wenn es vor einer Thrombolysetherapie eingenommen wurde. Daher muss bei Patienten, bei denen eine Thrombolysebehandlung durchgeführt werden soll, auf Zeichen äußerer oder innerer Blutungen (z. B. blaue Flecken) aufmerksam geachtet werden.
- Thrombozytenaggregationshemmer, z. B. Ticlopidin, Clopidogrel: Es kann zu einer Verlängerung der Blutungszeit kommen.
- Andere nichtsteroidale Analgetika/Antiphlogistika sowie Antirheumatika allgemein: erhöhtes Risiko für gastrointestinale Ulzera und -Blutungen.
- Systemische Glukokortikoide (mit Ausnahme von Hydrocortison als Ersatztherapie bei Morbus Addison): erhöhtes Risiko für gastrointestinale Nebenwirkungen.
- Alkohol: erhöhtes Risiko für gastrointestinale Ulzera und -Blutungen.
- Digoxin: Erhöhung der Plasmakonzentration.
- Antidiabetika: der Blutzuckerspiegel kann sinken.
- Methotrexat: Verminderung der Ausscheidung und Verdrängung aus der Plasmaproteinbindung durch Salicylate.
- Valproinsäure: Verdrängung aus der Plasmaproteinbindung durch Salicylate.
- Selektive-Serotonin-Wiederaufnahme-Hemmer (SSRIs): erhöhtes Risiko für gastrointestinale Blutungen aufgrund synergistischer Effekte.

# Abschwächung der Wirkung:

- Aldosteronantagonisten (Spironolacton und Canrenoat).
- Schleifendiuretika (z. B. Furosemid).
- Antihypertonika (insbesondere ACE-Hemmer).
- Urikosurika (z.B. Probenecid, Benzbromaron).
- NSARs: Die gleichzeitige Anwendung (am gleichen Tag) von manchen NSARs (Acetylsalicylsäure ausgenommen), wie zum Beispiel Ibuprofen und Naproxen, kann den irreversiblen plättchenhemmemden Effekt der Acetylsalicylsäure abschwächen. Die klinische Relevanz dieser Wechselwirkung ist nicht bekannt. Die Behandlung von Patienten mit einem erhöhten kardiovaskulären Risiko mit manchen NSARs, wie zum Beispiel Ibuprofen oder Naproxen, kann die kardioprotektive Wirkung der Acetylsalicylsäure einschränken (siehe Abschnitt 4.4).

Aspirin protect 100 mg/-300 mg sollte daher nicht zusammen mit einem der o.g. Stoffe

angewendet werden, ohne dass der Arzt ausdrücklich die Anweisung gegeben hat.

# 4.6 Schwangerschaft und Stillzeit

#### Schwangerschaft

Eine Hemmung der Prostaglandinsynthese kann die Schwangerschaft und/oder die embryonale/fetale Entwicklung ungünstig beeinflussen.

Daten aus epidemiologischen Studien weisen auf ein erhöhtes Risiko für Fehlgeburten sowie kardiale Missbildungen und Gastroschisis nach der Anwendung eines Prostaglandinsynthesehemmers in der Frühschwangerschaft hin. Es wird angenommen, dass das Risiko mit der Dosis und der Dauer der Therapie steigt.

Bisherige Erfahrungen bei Schwangeren mit der Anwendung von ASS in Tagesdosen zwischen 50 und 150 mg im zweiten und dritten Trimenon haben keine Hinweise auf eine Wehenhemmung, eine erhöhte Blutungsneigung oder einen vorzeitigen Verschluss des Ductus arteriosus ergeben.

Für Tagesdosen zwischen 150 und 300 mg liegen keine Erkenntnisse vor. Analgetisch wirkende ASS-Dosierungen können bei der Einnahme im letzten Trimenon der Schwangerschaft durch eine Hemmung der Prostaglandinsynthese zu einer Verlängerung der Gestationsdauer, einer Wehenhemmung und ab der 28.–30. Schwangerschaftswoche zu einem vorzeitigen Verschluss des Ductus arteriosus führen. In diesen Dosierungen ist außerdem mit einer erhöhten Blutungsneigung bei Mutter und Kind sowie bei einer Einnahme kurz vor der Geburt vermehrt mit intracranialen Blutungen bei Frühgeborenen zu rechnen.

# 1. und 2. Trimenon:

Aspirin protect 100 mg/-300 mg sollte in Tagesdosen bis zu 300 mg ASS im ersten und zweiten Trimenon nur nach strenger Indikationsstellung verordnet werden.

# 3. Trimenon

Die Einnahme einer Tagesdosis von bis zu 150 mg ASS im dritten Trimenon sollte ebenfalls nur bei zwingender Indikation erfolgen. Eine Einnahme von Aspirin protect 100 mg/-300 mg in Tagesdosen oberhalb von 150 mg ASS ist im letzten Trimenon kontraindiziert (siehe Abschnitt 4.3).

# Stillzeit

Der Wirkstoff Acetylsalicylsäure und seine Abbauprodukte gehen in geringen Mengen in die Muttermilch über. Da nachteilige Folgen für den Säugling bisher nicht bekannt geworden sind, wird bei Anwendung einer Tagesdosis von bis zu 150 mg eine Unterbrechung des Stillens in der Regel nicht erforderlich sein. Bei Einnahmen höherer Dosen (über 150 mg Tagesdosis) sollte abgestillt werden.

# 4.7 Auswirkungen auf die Verkehrstüchtigkeit und die Fähigkeit zum Bedienen von Maschinen

Acetylsalicylsäure hat keinen Einfluss auf die Verkehrstüchtigkeit und die Fähigkeit zum Bedienen von Maschinen.

#### 4.8 Nebenwirkungen

Bei der Bewertung von Nebenwirkungen werden folgende Häufigkeiten zugrunde gelegt:

| Sehr häufig: | ≥ 1/10 |
|---|---|
| Häufig: | ≥ 1/100, < 1/10 |
| Gelegentlich: | ≥ 1/1.000, < 1/100 |
| Selten: | ≥ 1/10.000, < 1/1.000 |
| Sehr selten: | < 1/10.000 |
| Nicht bekannt: | Häufigkeit auf Grundlage<br>der verfügbaren Daten<br>nicht abschätzbar |

#### Erkrankungen des Blutes und des Lymphsystems:

Selten bis sehr selten sind auch schwerwiegende Blutungen wie z.B. cerebrale Blutungen, besonders bei Patienten mit nicht eingestelltem Bluthochdruck und/oder gleichzeitiger Behandlung mit Antikoagulantien berichtet worden, die in Einzelfällen möglicherweise lebensbedrohlich sein können. Hämolyse und hämolytische Anämie wurden bei Patienten mit schwerem Glukose-6-Phosphat-Dehydrogenasemangel berichtet. Blutungen wie z.B. Nasenbluten, Zahnfleischbluten, Hautblutungen oder Blutungen des Urogenitaltraktes mit einer möglichen Verlängerung der Blutungszeit (siehe Abschnitt 4.4). Diese Wirkung kann über 4 bis 8 Tage nach der Einnahme anhalten.

# Erkrankungen des Immunsystems: Selten:

 Überempfindlichkeitsreaktionen der Haut, des Respirationstrakts, des Gastrointestinaltrakts und des kardiovaskulären Systems, vor allem bei Asthmatikern. Symptome können sein: Blutdruckabfall, Anfälle von Atemnot, Rhinitis, verstopfte Nase, anaphylaktischer Schock oder Quincke-Ödem.

# **Stoffwechsel- und Ernährungsstörungen:** Sehr selten:

- Hypoglykämie.
- Acetylsalicylsäure vermindert in niedriger Dosierung die Harnsäureausscheidung. Bei hierfür gefährdeten Patienten kann dies unter Umständen einen Gichtanfall auslösen.

# Erkrankungen des Nervensystems:

Kopfschmerzen, Schwindel, gestörtes Hörvermögen, Ohrensausen (Tinnitus) und mentale Verwirrung können Anzeichen einer Überdosierung sein (siehe Abschnitt 4.9).

# Erkrankungen des Gastrointestinaltrakts: Häufig:

- Gastrointestinale Beschwerden wie Sodbrennen, Übelkeit, Erbrechen, Bauchschmerzen und Durchfälle.
- Geringfügige Blutverluste aus dem Gastrointestinaltrakt (Mikroblutungen).

# Gelegentlich:

- Gastrointestinale Ulzera, die sehr selten zur Perforation führen können.
- Gastrointestinale Blutungen.
   Nach längerer Anwendung von Aspirin protect 100 mg/-300 mg kann eine Eisenmangelanämie durch verborgene Blutverluste aus dem Gastrointestinaltrakt auftreten.
- Gastrointestinale Entzündungen.

001915-27444

2

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.



# Aspirin® protect 100 mg/- 300 mg

Bei Auftreten von schwarzem Stuhl oder blutigem Erbrechen (Zeichen einer schweren Magenblutung) ist sofort der Arzt zu benachrichtigen.

#### Leber- und Gallenerkrankungen: Sehr selten:

Erhöhungen der Leberwerte

# Erkrankungen der Haut und des Unterhautzellgewebes:

Gelegentlich:

Hautreaktionen (sehr selten bis hin zu Erythema exsudativum multiforme)

### Erkrankungen der Nieren und Harnwege: Sehr selten:

Nierenfunktionsstörungen und akutes Nierenversagen wurden berichtet.

# Meldung des Verdachts auf Nebenwir-

Die Meldung des Verdachts auf Nebenwirkungen nach der Zulassung ist von großer Wichtigkeit. Sie ermöglicht eine kontinuierliche Überwachung des Nutzen-Risiko Verhältnisses des Arzneimittels. Angehörige von Gesundheitsberufen sind aufgefordert, jeden Verdachtsfall einer Nebenwirkung

Bundesinstitut für Arzneimittel und Medizinprodukte Abt. Pharmakovigilanz Kurt-Georg-Kiesinger Allee 3 D-53175 Bonn Website: http://www.bfarm.de anzuzeigen

# 4.9 Überdosierung

Unterschieden werden die chronische Überdosierung von Acetylsalicylsäure mit überwiegend zentralnervösen Störungen wie Benommenheit, Schwindel, Verwirrtheit oder Übelkeit ("Salicylismus") und die akute Into-

Im Vordergrund einer akuten Acetylsalicylsäure-Vergiftung steht eine schwere Störung des Säure-Basen-Gleichgewichtes Bereits im therapeutischen Dosisbereich kommt es zu einer respiratorischen Alkalose infolge gesteigerter Atmung. Sie wird durch eine erhöhte renale Ausscheidung von Hydrogencarbonat kompensiert, so dass der pH-Wert des Blutes normal ist. Bei toxischen Dosen reicht diese Kompensation nicht mehr aus und der pH-Wert sowie die Hydrogencarbonatkonzentration im Blut sinken ab. Der PCO2-Wert des Plasmas kann zeitweilig normal sein. Es liegt scheinbal das Bild einer metabolischen Azidose vor. Tatsächlich aber handelt es sich um eine Kombination von respiratorischer und metabolischer Azidose. Die Ursachen hierfür sind: Einschränkung der Atmung durch toxische Dosen, Anhäufung von Säure, zum Teil durch verminderte renale Ausscheidung (Schwefel- und Phosphorsäure sowie Salicylsäure, Milchsäure, Acetessigsäure u.a.) infolge einer Störung des Kohlenhydrat-Stoffwechsels. Hierzu tritt eine Störung des Flektrolythaushaltes auf. Es kommt zu grö-Beren Kaliumverlusten.

Symptome der akuten Intoxikation

Die Symptome bei leichteren Graden einer akuten Vergiftung (200-400 µg/ml): Neben Störungen des Säure-Basen-Gleichgewichtes, des Elektrolythaushaltes (z. B.

Kaliumverluste), Hypoglykämie, Hautausschlägen sowie gastrointestinalen Blutungen werden Hyperventilation, Ohrensausen, Übelkeit, Erbrechen, Beeinträchtigung von Sehen und Hören, Kopfschmerzen, Schwindel. Verwirrtheitszustände beobachtet

Bei schweren Vergiftungen (über 400  $\mu g/ml$ ) können Delirien, Tremor, Atemnot, Schweißausbrüche, Exsikkose, Hyperthermie und Koma auftreten.

Bei Intoxikationen mit letalem Ausgang tritt der Tod in der Regel durch Versagen der Atemfunktion ein.

# Therapie der Intoxikation

Die Therapiemöglichkeiten zur Behandlung einer Acetylsalicylsäureintoxikation richten sich nach Ausmaß, Stadium und klinischen Symptomen der Intoxikation. Sie entsprechen den üblichen Maßnahmen zur Verminderung der Resorption des Wirkstoffs, Kontrolle des Wasser- und Elektrolythaushaltes sowie der gestörten Temperaturregulation und Atmung.

Im Vordergrund stehen Maßnahmen, die der Beschleunigung der Ausscheidung und der Normalisierung des Säure-Basen- und Elektrolythaushaltes dienen. Neben Infusionslösungen mit Natriumhydrogencarbonat und Kaliumchlorid werden auch Diuretika verabreicht. Die Reaktion des Harns soll basisch sein, damit der Ionisationsgrad der Salicylate zu- und damit die Rückdiffusionsrate in den Tubuli abnimmt.

Eine Kontrolle der Blut-Werte (pH, PCO2, Hydrogencarbonat, Kalium u. a.) ist sehr zu empfehlen. In schweren Fällen kann eine Hämodialyse notwendig sein.

# 5. PHARMAKOLOGISCHE EIGEN-**SCHAFTEN**

# 5.1 Pharmakodynamische Eigenschaften

Pharmakotherapeutische Gruppe: Antithrombotische Mittel, Thrombozytenaggregationshemmer, Acetylsalicylsäure ATC-Code: B01AC06

Acetylsalicylsäure hat eine irreversible thrombozytenaggregationshemmende Wirkung. Diese Wirkung auf die Thrombozyten wird über eine Acetylierung der Cyclooxygenase erreicht. Dadurch wird irreversibel die Bildung von Thromboxan A2 (einem die Thrombozytenaggregation fördernden und vasokonstringierend wirkenden Prostaglandin) in den Thrombozyten gehemmt. Dieser Effekt ist dauerhaft und hält gewöhnlich für die gesamte achttägige Lebensdauer eines Thrombozyten an.

Paradoxerweise hemmt die Acetylsalicylsäure auch die Bildung von Prostacyclin (einem thrombozytenaggregationshemmenden aber vasodilatorisch wirksamen Prostaglandin) in den Endothelzellen der Gefäßwände. Dieser Effekt ist vorübergehend. Sobald die Acetylsalicylsäure aus dem Blut ausgewaschen ist, produzieren die kernhaltigen Endothelzellen wieder Prostacyclin.

Infolge dessen bewirkt Acetylsalicylsäure bei einmal täglicher Gabe in niedriger Dosierung (< 300 mg /Tag) eine Blockade von Thromboxan A2 in den Thrombozyten ohne ausgeprägte Beeinträchtigung der Prostacyclinbildung.

Acetylsalicylsäure gehört außerdem zur Gruppe der säurebildenden nichtsteroidalen

Antiphlogistika mit analgetischen, antipyretischen und antiphlogistischen Eigenschaften. Ihr Wirkungsmechanismus beruht auf der irreversiblen Hemmung von Cyclooxygenase-Enzymen, die an der Prostaglandinsynthese beteiligt sind.

Acetylsalicylsäure wird in höheren oralen Dosierungen zur Behandlung von leichten bis mäßig starken Schmerzen, bei erhöhter Temperatur und zur Behandlung akuter und chronisch entzündlicher Erkrankungen (z. B. rheumatoide Arthritis) angewendet.

Experimentelle Daten deuten darauf hin, dass Ibuprofen bei gleichzeitiger Anwendung mit Acetylsalicylsäure die Wirkung von niedrig dosierter Acetylsalicylsäure auf die Blutplättchenaggregation hemmen kann. In einer Studie, in der 400 mg Ibuprofen als Einzeldosis 8 Stunden vor bzw. 30 Minuten nach der Gabe eines schnell freisetzenden Acetylsalicylsäure-Präparats (81 mg) eingenommen wurde, kam es zu einer verminderten Wirkung von Acetylsalicylsäure auf die Bildung von Thromboxan bzw. die Blutplättchenaggregation. Jedoch lassen sich wegen der begrenzten Datenlage sowie der Unsicherheiten bei einer Extrapolation von ex vivo Daten auf die klinische Situation keine sicheren Schlussfolgerungen bezüglich der regelmäßigen Anwendung von Ibuprofen treffen. Bei gelegentlicher Anwendung von Ibuprofen ist eine klinisch relevante Wechselwirkung nicht wahrscheinlich.

# 5.2 Pharmakokinetische Eigenschaften

Acetylsalicylsäure wird vor. während und nach der Resorption in ihren aktiven Hauptmetaboliten SalicvIsäure umgewandelt. Die Metaboliten werden überwiegend über die Niere ausgeschieden.

Hauptmetaboliten der Acetylsalicylsäure sind neben der Salicylsäure das Glycinkonjugat der Salicylsäure (Salicylursäure), das Ether- und das Esterglukuronid der Salicylsäure (Salicylphenolglukuronid und Salicylacetylglukuronid) sowie die durch Oxidation von Salicylsäure entstehende Gentisinsäure und deren Glycinkonjugat.

Die Resorption nach oraler Gabe von Acetylsalicylsäure erfolgt, abhängig von der galenischen Formulierung, schnell und vollständig. Der Acetylrest der Acetylsalicylsäure wird teilweise bereits während der Passage durch die Mukosa des Gastrointestinaltraktes hydrolytisch gespalten.

Maximale Plasmaspiegel werden nach 10-20 min (Acetylsalicylsäure) bzw. 0,3-2 h (Gesamtsalicylat) erreicht

Die Eliminationskinetik von Salicvlsäure ist in starkem Maße von der Dosis abhängig. da die Metabolisierung von Salicylsäure kapazitätslimitiert ist (fluktuelle Eliminationshalbwertszeit zwischen 2 und 30 h).

Die Eliminationshalbwertszeit von Acetylsalicylsäure beträgt nur einige Minuten, die Eliminationshalbwertszeit der Salicylsäure beträgt nach Einnahme einer Dosis von

Acetylsalicylsäure 2 h, nach Applikation von 1 g 4 h, nach Einnahme einer Einzeldosis von 5 g verlängert sie sich auf 20 h.

Die Plasmaeiweißbindung beim Menschen ist konzentrationsabhängig; Werte von  $49\,\%$ bis über 70 % (Acetylsalicylsäure) bzw. 66 % bis 98 % (Salicylsäure) wurden gefunden.

001915-27444

G656

# Aspirin® protect 100 mg/- 300 mg



Im Liquor und in der Synovialflüssigkeit ist Salicylsäure nach Einnahme von Acetylsalicylsäure nachweisbar.

Salicylsäure ist placentagängig und geht in die Muttermilch über.

# 5.3 Präklinische Daten zur Sicherheit

Das präklinische Sicherheitsprofil von Acetylsalicylsäure ist gut dokumentiert. Salicylate haben in tierexperimentellen Untersuchungen Nierenschädigungen und gastrointestinale Ulzera hervorgerufen. Acetylsalicylsäure wurde angemessen auf Mutagenität und Kanzerogenität untersucht; es wurden keine relevanten Hinweise auf mutagenes oder karzinogenes Potenzial festgestellt.

Salicylate haben bei einer Reihe von Tierspezies teratogene Wirkungen gezeigt. Es wurden Implantationsstörungen, embryotoxische- und fetotoxische Wirkungen sowie Störungen der Lernfähigkeit der Jungtiere nach pränataler Exposition angegeben.

#### 6. PHARMAZEUTISCHE ANGABEN

# 6.1 Liste der sonstige Bestandteile

Maisstärke

Cellulosepulver

Methacrylsäure-Ethylacrylat-Copolymer

1:1-Dispersion 30%

Polysorbat 80

Natriumdodecylsulfat

Talkum

Triethylcitrat

# 6.2 Inkompatibilitäten

keine

# 6.3 Dauer der Haltbarkeit

Aspirin protect 100 mg: 5 Jahre Aspirin protect 300 mg: 5 Jahre

#### 6.4 Besondere Vorsichtsmaßnahmen für die Aufbewahrung

Nicht über 25°C lagern!

# 6.5 Art und Inhalt des Behältnisses

# Aspirin protect 100 mg

PP-Aluminium-Blister:

Packung mit 42 magensaftresistenten Tabletten

Packung mit 98 magensaftresistenten Ta-

Klinikpackung mit 240 (10 x 24) magen-

# Aspirin protect 300 mg

PP-Aluminium-Blister:

Packungen mit 42 magensaftresistenten Tabletten Packungen mit 98 magensaftresistenten

Tabletten

Es werden möglicherweise nicht alle Packungsgrößen in den Verkehr gebracht.

# 6.6 Besondere Vorsichtsmaßnahmen für die Beseitigung

Keine besonderen Anforderungen.

# 7. INHABER DER ZULASSUNG

Bayer Vital GmbH 51368 Leverkusen Deutschland

#### 8. ZULASSUNGSNUMMERN

# Aspirin protect 100 mg

16854.01.01/30828.01.01/33171.00.00

<u>Aspirin protect 300 mg</u> 16854.00.01/30828.00.01/33171.01.00

### 9. DATUM DER ERTEILUNG DER ZULASSUNG/VERLÄNGERUNG **DER ZULASSUNG**

# Aspirin protect 100 mg

16854.01.01: 28.12.1993/30.03.2009 30828.01.01: 28.12.1993/18.11.2013 33171.00.00: 09.10.1995/19.08.2013

Aspirin protect 300 mg 16854.00.01: 28.12.1993/12.09.2007 30828.00.01: 28.12.1993/25.07.2007 33171.01.00: 09.10.1995/18.11.2013

# 10. STAND DER INFORMATION

März 2017

# 11. VERKAUFSABGRENZUNG

Apothekenpflichtig

Zentrale Anforderung an:

Rote Liste Service GmbH

Fachinfo-Service

Mainzer Landstraße 55 60329 Frankfurt

001915-27444



# Plavix® 75 mg Filmtabletten Plavix® 300 mg Filmtabletten

#### 1. BEZEICHNUNG DER ARZNEIMITTEL

Plavix 75 mg Filmtabletten Plavix 300 mg Filmtabletten

#### 2. QUALITATIVE UND QUANTITATIVE ZUSAMMENSETZUNG

Plavix 75 mg Filmtabletten

Jede Filmtablette enthält 75 mg Clopidogrel (als Hydrogensulfat).

Sonstige Bestandteile mit bekannter Wir-

Jede Filmtablette enthält 3 mg Lactose und 3,3 mg hydriertes Rizinusöl.

Plavix 300 mg Filmtabletten

Jede Filmtablette enthält 300 mg Clopidogrel (als Hydrogensulfat).

Sonstige Bestandteile mit bekannter Wirkung:

Jede Filmtablette enthält 12 mg Lactose und 13,2 mg hydriertes Rizinusöl.

Vollständige Auflistung der sonstigen Bestandteile siehe Abschnitt 6.1.

#### 3. DARREICHUNGSFORM

Filmtablette.

Plavix 75 mg Filmtabletten

Rosafarben, rund, bikonvex, mit Prägung "75" auf der einen Seite und "1171" auf der anderen Seite

Plavix 300 mg Filmtabletten

Rosafarben, länglich, mit Prägung "300" auf der einen Seite und "1332" auf der anderen Seite.

# 4. KLINISCHE ANGABEN

# 4.1 Anwendungsgebiete

Sekundärprävention atherothrombotischer Ereignisse

Clopidogrel ist indiziert bei:

- erwachsenen Patienten mit Herzinfarkt (wenige Tage bis weniger als 35 Tage mit ischämischem zurückliegend), Schlaganfall (7 Tage bis weniger als 6 Monate zurückliegend) oder mit nachgewiesener peripherer arterieller Verschlusskrankheit,
- erwachsenen Patienten mit akutem Koronarsyndrom:
- akutes Koronarsyndrom ohne ST-Strecken-Hebung (instabile Angina Pectoris oder Non-Q-Wave-Myokardinfarkt), einschließlich Patienten, denen bei einer perkutanen Koronarintervention ein Stent implantiert wurde in Kombination mit Acetylsalicylsäure (ASS)
- akuter Myokardinfarkt mit ST-Strecken-Hebung, in Kombination mit ASS bei medizinisch behandelten Patienten, für die eine thrombolytische Therapie infrage kommt.

Prävention atherothrombotischer und thromboembolischer Ereignisse bei Vorhofflimmern Bei erwachsenen Patienten mit Vorhofflimmern, bei denen wenigstens ein Risikofaktor für vaskuläre Ereignisse vorliegt, die keine Vitamin-K-Antagonisten-(VKA-)Therapie erhalten können und die ein geringes Blutungsrisiko aufweisen, ist Clopidogrel in Kombination mit ASS angezeigt zur Prophylaxe atherothrombotischer und thromboembolischer Ereignisse, einschließlich Schlaganfall.

Weitere Informationen sind im Abschnitt 5.1 enthalten

# 4.2 Dosierung und Art der Anwendung

Dosierung

Erwachsene und ältere Patienten

Plavix 75 mg Filmtabletten

Es werden einmal täglich 75 mg Clopidogrel gegeben.

Plavix 300 mg Filmtabletten

Diese 300 mg-Clopidogrel-Tablette ist als Aufsättigungsdosis vorgesehen.

Bei Patienten mit akutem Koronarsyndrom:

- Akutes Koronarsyndrom ohne ST-Strecken-Hebung (instabile Angina Pectoris oder Non-Q-Wave-Myokardinfarkt): Die Clopidogrel-Therapie sollte mit einer einmaligen Aufsättigungsdosis von 300 mg (Loading dose) begonnen werden und dann langfristig mit 75 mg einmal täglich fortgesetzt werden (in Kombination mit täglich 75-325 mg Acetylsalicylsäure [ASS]). Da höhere ASS-Dosierungen mit einem erhöhten Blutungsrisiko assoziiert waren, wird eine ASS-Dosis bis höchstens 100 mg empfohlen. Die optimale Behandlungsdauer ist nicht formal festgeschrieben. Klinische Studiendaten belegen eine Anwendung bis zu 12 Monaten, und der maximale Nutzen wurde nach 3 Monaten gesehen (siehe Abschnitt 5.1).
- Akuter Myokardinfarkt mit ST-Strecken-Hebung: Clopidogrel sollte einmal täglich in einer Dosis von 75 mg nach einer einmaligen Aufsättigungsdosis von 300 mg in Kombination mit ASS sowie mit oder ohne Thrombolytika gegeben werden. Die Therapie bei Patienten über 75 Jahre sollte ohne Aufsättigungsdosis beginnen.

Die Kombinationstherapie sollte so früh wie möglich nach Auftreten der Symptome initiiert und für mindestens vier Wochen fortgesetzt werden. Der Nutzen der Kombination von Clopidogrel mit ASS über vier Wochen hinaus wurde nicht untersucht (siehe Abschnitt 5.1).

Bei Patienten mit Vorhofflimmern sollte Clopidogrel einmal täglich in einer Dosis von 75 mg gegeben werden. ASS (75-100 mg täglich) sollte in Kombination mit Clopidogrel begonnen und weitergeführt werden (siehe Abschnitt 5.1).

Wenn eine Dosis vergessen wurde:

- Innerhalb von 12 Stunden nach der regulär geplanten Zeit: Patienten sollten die Dosis sofort einnehmen und die nächste Dosis dann wieder zur regulär geplanten
- Nach mehr als 12 Stunden: Patienten sollten die Dosis zum regulär vorgesehenen nächsten Einnahmezeitpunkt einnehmen und nicht die Dosis verdoppeln.

Kinder und Jugendliche

Clopidogrel darf bei Kindern nicht angewendet werden, da Bedenken zur Wirksamkeit vorliegen (siehe Abschnitt 5.1).

- Eingeschränkte Nierenfunktion Die therapeutische Erfahrung bei Patienten mit eingeschränkter Nierenfunktion ist bearenzt (siehe Abschnitt 4.4).
- Eingeschränkte Leberfunktion

Die therapeutische Erfahrung bei Patienten mit mäßiger Leberfunktionsstörung, die eine hämorrhagische Diathese aufweisen können, ist begrenzt (siehe Abschnitt 4.4).

Art der Anwendung

Zum Einnehmen.

Es kann unabhängig von den Mahlzeiten eingenommen werden

#### 4.3 Gegenanzeigen

- Überempfindlichkeit gegen den in Abschnitt 2 genannten Wirkstoff oder einen der in Abschnitt 6.1 genannten sonstigen Bestandteile,
- schwere Leberfunktionsstörungen,
- akute pathologische Blutung, wie bei Magen-Darm-Geschwüren oder intrakraniellen Blutungen

#### 4.4 Besondere Warnhinweise und Vorsichtsmaßnahmen für die Anwendung

Blutungen und hämatologische Störungen Wegen des Risikos für Blutungen und hämatologische Nebenwirkungen sollte sofort eine Bestimmung des Blutbildes und/oder ein anderes geeignetes Testverfahren erwogen werden, wenn während der Behandlung der klinische Verdacht auf eine Blutung entsteht (siehe Abschnitt 4.8). Wie auch andere thrombozytenaggregationshemmende Arzneimittel sollte Clopidogrel mit Vorsicht bei Patienten angewendet werden, die wegen eines Traumas, eines operativen Eingriffs oder anderer Erkrankungen ein erhöhtes Blutungsrisiko haben, sowie bei Patienten die ASS, Heparin, Glykoprotein-Ilb/Illa-Antagonisten oder nicht steroidale antiinflammatorische Arzneimittel (NSAR), einschließlich COX-2-Inhibitoren, oder selektive Serotonin-Wiederaufnahmehemmer (SSRI) oder andere mit einem Blutungsrisiko assoziierte Arzneimittel wie Pentoxifyllin erhalten (siehe Abschnitt 4.5). Diese Patienten sollten hinsichtlich jeglicher Blutungszeichen einschließlich okkulter Blutungen sorgfältig überwacht werden, besonders während der ersten Behandlungswochen und/oder nach invasiver kardialer Intervention oder Operation. Die gleichzeitige Anwendung von Clopidogrel mit oralen Antikoagulanzien wird nicht empfohlen, da Blutungen verstärkt werden können (siehe Abschnitt 4.5).

Wenn bei einem Patienten eine elektive Operation vorgesehen ist und ein thrombozytenaggregationshemmender Effekt vorübergehend unerwünscht ist, sollte Clopidogrel 7 Tage vor der Operation abgesetzt werden. Die Patienten sollten dem Arzt oder Zahnarzt mitteilen, dass sie Clopidogrel einnehmen, wenn ein operativer Eingriff geplant ist oder ein neues Arzneimittel genommen werden soll. Clopidogrel verlängert die Blutungszeit und sollte bei Patienten mit zu Blutungen neigenden Läsionen (besonders

2018

003345-31445

# Plavix® 75 mg Filmtabletten Plavix® 300 mg Filmtabletten

SANOFI 🗳

gastrointestinal und intraokulär) mit Vorsicht angewandt werden.

Die Patienten sind zu informieren, dass es bei Einnahme von Clopidogrei (allein oder in Kombination mit ASS) länger als sonst dauern könnte, bis eine Blutung zum Stillstand kommt, und dass sie dem Arzt jede ungewöhnliche Blutung (Lokalisation oder Dauer) melden sollten.

Thrombotisch-thrombozytopenische Purpura (TTP)

Nach der Einnahme von Clopidogrel wurde sehr selten eine thrombotisch-thrombozytopenische Purpura (TTP) beobachtet und dies manchmal bereits nach kurzer Einnahmedauer. Die TTP ist gekennzeichnet durch Thrombozytopenie und mikroangiopathische hämolytische Anämie in Verbindung mit neurologischen Symptomen, Nierenfunktionsstörungen oder Fieber. Eine TTP ist potenziell lebensbedrohlich und erfordert eine sofortige Behandlung einschließlich Plasmapherese.

#### Erworbene Hämophilie

Es wurde von erworbener Hämophilie nach der Einnahme von Clopidogrel berichtet. Im Falle einer bestätigten isolierten Verlängerung der aktivierten partiellen Thromboplastinzeit (aPTT) mit oder ohne Blutungen sollte eine erworbene Hämophilie in Betracht gezogen werden. Patienten mit der bestätigten Diagnose einer erworbenen Hämophilie müssen von einem Spezialisten versorgt und behandelt werden und Clopidogrel muss abgesetzt werden.

Vor kurzem aufgetretener Schlaganfall Nach akutem ischämischem Schlaganfall (weniger als 7 Tage zurückliegend) kann Clopidogrel nicht empfohlen werden, da hierfür keine Daten vorliegen.

# Cytochrom P450 2C19 (CYP2C19)

Pharmakogenetik: Bei Patienten, die langsame CYP2C19-Metabolisierer sind, wird bei empfohlener Clopidogrel-Dosierung weniger aktiver Metabolit von Clopidogrel gebildet, was einen verminderten Effekt auf die Thrombozytenfunktion zur Folge hat. Es sind Tests verfügbar, mit denen der CYP2C19-Genotyp des Patienten bestimmt werden kann

Da Clopidogrel teilweise durch CYP2C19 zu seinem aktiven Metaboliten verstoffwechselt wird, ist zu erwarten, dass der Gebrauch von Arzneimitteln, die die Aktivität dieses Enzyms hemmen, zu einem erniedrigten Spiegel des aktiven Metaboliten von Clopidogrel führt. Die klinische Relevanz dieser Wechselwirkung ist ungewiss. Als Vorsichtsmaßnahme sollte vom gleichzeitigen Gebrauch starker oder mäßig starker CYP2C19-Inhibitoren abgeraten werden (siehe Abschnitt 4.5 bez. einer Liste von CYP2C19-Inhibitoren, siehe auch Abschnitt 5.2).

# CYP2C8-Substrate

Vorsicht ist geboten bei Patienten, die gleichzeitig mit Clopidogrel und Substraten von CYP2C8 behandelt werden (siehe Abschnitt 4.5).

Kreuzreaktionen unter Thienopyridinen Patienten sollten auf eine Überempfindlichkeit gegen Thienopyridine (wie z.B. Clopidogrel, Ticlopidin, Prasugrel) in der Vorgeschichte untersucht werden, da Kreuzreaktionen unter Thienopyridinen berichtet worden sind (siehe Abschnitt 4.8). Thienopyridine können schwache bis schwere allergische Reaktionen, wie z.B. Hautausschlag, Angioödem, oder hämatologische Kreuzreaktionen, wie z.B. Thrombozytopenie und Neutropenie, verursachen. Bei Patienten, die bereits eine allergische Reaktion und/oder eine hämatologische Reaktion gegen ein anderes Thienopyridin gezeigt haben, kann ein erhöhtes Risiko für die Entwicklung der gleichen oder einer anderen Reaktion bestehen. Eine Überwachung von Patienten mit bekannter Allergie gegen Thienopyridine auf Zeichen einer Überempfindlichkeit wird angeraten.

#### Eingeschränkte Nierenfunktion

Es liegen bisher nur begrenzte therapeutische Erfahrungen mit Clopidogrel bei Patienten mit Nierenfunktionsstörungen vor. Daher ist Clopidogrel bei diesen Patienten mit Vorsicht anzuwenden (siehe Abschnitt 4.2).

# Eingeschränkte Leberfunktion

Es liegen bisher nur begrenzte Erfahrungen mit Clopidogrel bei Patienten mit mäßigen Leberfunktionsstörungen und damit möglicherweise verbundener hämorrhagischer Diathese vor. Daher ist Clopidogrel bei diesen Patienten mit Vorsicht anzuwenden (siehe Abschnitt 4.2).

# Sonstige Bestandteile

Plavix enthält Lactose. Patienten mit der seltenen hereditären Galactose-Intoleranz, Lactase-Mangel oder Glucose-Galactose-Malabsorption sollten dieses Arzneimittel nicht einnehmen.

Dieses Arzneimittel enthält hydriertes Rizinusöl, welches Magenverstimmung und Durchfall hervorrufen kann.

### 4.5 Wechselwirkungen mit anderen Arzneimitteln und sonstige Wechselwirkungen

Arzneimittel mit assoziiertem Blutungsrisiko: Es besteht ein erhöhtes Blutungsrisiko aufgrund des möglichen additiven Effekts. Die gleichzeitige Anwendung von Arzneimitteln mit assoziiertem Blutungsrisiko sollte mit Vorsicht erfolgen (siehe Abschnitt 4.4).

Orale Antikoagulanzien: Die gleichzeitige Anwendung von Clopidogrel und oralen Antikoagulanzien wird nicht empfohlen, da Blutungen verstärkt werden können (siehe Abschnitt 4.4).

Obwohl die Anwendung von Clopidogrel 75 mg/Tag weder die Pharmakokinetik von S-Warfarin noch die "International Normalized Ratio" (INR) bei Patienten, die eine Warfarin-Langzeittherapie erhalten, verändert, erhöht die gleichzeitige Anwendung von Clopidogrel mit Warfarin das Blutungsrisiko aufgrund unabhängiger Auswirkungen auf die Hämostase.

Glykoprotein-Ilb/Illa-Inhibitoren: Clopidogrel sollte mit Vorsicht bei Patienten angewendet werden, die gleichzeitig mit Glykoprotein-Ilb/Illa-Inhibitoren behandelt werden (siehe Abschnitt 4.4).

Acetylsalicylsäure (ASS): ASS hatte keinen Einfluss auf die Clopidogrel-vermittelte

Hemmung der ADP-induzierten Thrombozytenaggregation. Clopidogrel führte dagegen zu einer Potenzierung der Wirkung von ASS auf die kollageninduzierte Thrombozytenaggregation. Die gleichzeitige Gabe von zweimal täglich 500 mg ASS für einen Tag führte zu keiner signifikanten Zunahme der Clopidogrel-bedingten Verlängerung der Blutungszeit. Eine pharmakodynamische Wechselwirkung zwischen Clopidogrel und Acetylsalicylsäure, die zu einem erhöhten Blutungsrisiko führt, ist möglich. Deshalb sollte eine Kombinationstherapie nur mit Vorsicht durchgeführt werden (siehe Abschnitt 4.4). Allerdings sind Clopidogrel und ASS gemeinsam bis zu einem Jahr lang gegeben worden (siehe Abschnitt 5.1).

Heparin: In einer klinischen Studie mit gesunden Probanden war es unter Clopidogrel weder notwendig, die Heparin-Dosierung anzupassen, noch veränderte Clopidogrel den Einfluss von Heparin auf die Blutgerinnung. Die gleichzeitige Gabe von Heparin hatte keine Wirkung auf die Clopidogrelinduzierte Hemmung der Thrombozytenaggregation. Eine pharmakodynamische Wechselwirkung zwischen Clopidogrel und Heparin, die zu einem erhöhten Blutungsrisiko führt, ist möglich. Deshalb sollte eine Kombinationstherapie nur mit Vorsicht durchgeführt werden (siehe Abschnitt 4.4).

Thrombolytika: Die Unbedenklichkeit einer gleichzeitigen Gabe von Clopidogrel, direkten oder indirekten Thrombolytika (fibrinder nicht fibrinspezifisch) und Heparinen wurde bei Patienten mit akutem Herzinfarkt untersucht. Die Inzidenz von klinisch relevanten Blutungen entsprach derjenigen bei gleichzeitiger Gabe von thrombolytischen Substanzen und Heparin zusammen mit ASS (siehe Abschnitt 4.8).

NSAR: In einer klinischen Studie mit Probanden führte die gleichzeitige Gabe von Clopidogrel und Naproxen zu einem vermehrten okkulten gastrointestinalen Blutverlust. Aufgrund des Fehlens von Interaktionsstudien mit anderen NSAR ist jedoch derzeit nicht bekannt, ob bei allen NSAR ein erhöhtes Risiko für gastrointestinale Blutungen besteht. Demnach sollte die gleichzeitige Gabe von NSAR, einschließlich COX-2-Inhibitoren, und Clopidogrel mit Vorsicht erfolgen (siehe Abschnitt 4.4).

SSRI: Da SSRI die Aktivierung der Thrombozyten beeinflussen und das Blutungsrisiko erhöhen, sollte die gleichzeitige Gabe von SSRI mit Clopidogrel mit Vorsicht erfolgen.

Andere gleichzeitige Therapie: Da Clopidogrel teilweise durch CYP2C19 zu seinem aktiven Metaboliten verstoffwechselt wird, ist zu erwarten, dass der Gebrauch von Arzneimitteln, die die Aktivität dieses Enzyms hemmen, zu einem erniedrigten Spiegel des aktiven Metaboliten von Clopidogrel führt. Die klinische Relevanz dieser Wechselwirkung ist ungewiss. Als Vorsichtsmaßnahme sollte vom gleichzeitigen Gebrauch starker oder mäßig starker CYP2C19-Inhibitoren abgeraten werden (siehe Abschnitte 4.4 und 5.2).

Zu den Arzneimitteln, die starke oder mäßig starke CYP2C19-Inhibitoren darstellen, gehören z.B. Omeprazol und Esomeprazol,

003345-3144



Plavix® 75 mg Filmtabletten Plavix® 300 mg Filmtabletten

Fluvoxamin, Fluoxetin, Moclobemid, Voriconazol, Fluconazol, Ticlopidin, Carbamazepin und Efavirenz.

Protonenpumpen-Inhibitoren (PPI):

Die Anwendung von einmal täglich 80 mg Omeprazol entweder gleichzeitig mit Clopidogrel oder im Abstand von 12 Stunden verminderte die Exposition gegenüber dem aktiven Metaboliten um 45 % (Aufsättigungsdosis) und 40 % (Erhaltungsdosis). Die Abnahme war verbunden mit einer Reduktion der Hemmung der Thrombozytenaggregation um 39 % (Aufsättigungsdosis) und 21 % (Erhaltungsdosis). Esomeprazol hat vermutlich eine ähnliche Wechselwirkung mit Clopidogrel.

In Beobachtungsstudien und klinischen Prüfungen wurden widersprüchliche Daten zu den klinischen Auswirkungen dieser pharmakokinetischen (PK)/pharmakodynamischen (PD) Wechselwirkung, wie schwere kardiovaskuläre Ereignisse, berichtet. Als Vorsichtsmaßnahme sollte von der gleichzeitigen Anwendung von Omeprazol oder Esomeprazol abgeraten werden (siehe Abschnitt 4 4)

Eine weniger ausgeprägte Abnahme der Exposition gegenüber dem Metaboliten wurde mit Pantoprazol oder Lansoprazol beobachtet.

Die Plasmakonzentrationen des aktiven Metaboliten waren um 20 % (Aufsättigungsdosis) und 14 % (Erhaltungsdosis) während der gleichzeitigen Anwendung von einmal täglich 80 mg Pantoprazol reduziert. Dies war verbunden mit einer durchschnittlichen Abnahme der Hemmung der Thrombozytenaggregation um 15 % bzw. 11 %. Diese Ergebnisse weisen darauf hin, dass Clopidogrel zusammen mit Pantoprazol angewendet werden kann.

Es gibt keine Erkenntnisse, dass andere Arzneimittel, die die Magensäure reduzieren, wie  ${\rm H_2}$ -Blocker oder Antazida, die thrombozytenaggregationshemmende Wirkung von Clopidogrel beeinträchtigen.

# Andere Arzneimittel:

Es wurden zahlreiche weitere klinische Studien mit Clopidogrel und anderen gleichzeitig gegebenen Arzneimitteln durchgeführt, um mögliche pharmakokinetische und pharmakodynamische Wechselwirkungen zu untersuchen. Es wurden keine klinisch signifikanten pharmakodynamischen Wechselwirkungen beobachtet, wenn Clopidogrel zusammen mit Atenolol, Nifedipin oder einer Kombination aus Atenolol und Nifedipin gegeben wurde. Auch eine gleichzeitige Gabe von Phenobarbital oder Östrogen hatte keinen signifikanten Einfluss auf die Pharmakodynamik von Clopidogrel.

Die gleichzeitige Gabe von Clopidogrel hatte keinen Einfluss auf die Pharmakokinetik von Digoxin oder Theophyllin. Antazida veränderten die Resorationsrate von Clopidogrel nicht.

Die Ergebnisse der CAPRIE-Studie zeigen, dass Phenytoin und Tolbutamid, die durch CYP2C9 verstoffwechselt werden, zusammen mit Clopidogrel unbedenklich gegeben werden können.

CYP2C8-Substrate: Clopidogrel erhöht nachweislich die Repaglinidexposition bei

Probanden. In-vitro-Studien haben gezeigt, dass die gesteigerte Repaglinidexposition auf einer Inhibition von CYP2C8 durch den glucuronidierten Metaboliten von Clopidogrel beruht. Aufgrund des Risikos erhöhter Plasmakonzentrationen sollte die gleichzeitige Anwendung von Clopidogrel und Arzneimitteln, die primär über CYP2C8 metabolisiert werden (z. B. Repaglinid, Paclitaxel), mit Vorsicht erfolgen (siehe Abschnitt 4.4).

Abgesehen von den oben beschriebenen Informationen zu spezifischen Arzneimittelwechselwirkungen gibt es einige Arzneimittel, die Patienten mit atherothrombotischen Erkrankungen häufig gegeben werden, zu denen keine Interaktionsstudien mit Clopidogrel durchgeführt worden sind. Allerdings haben Patienten, die in klinische Studien mit Clopidogrel eingeschlossen wurden, eine Vielzahl weiterer Arzneimittel wie Diuretika. Betablocker, ACE-Hemmer, Kalziumkanalblocker, Cholesterinsenker, Koronar-Vasodilatatoren, Antidiabetika (einschließlich Insulin), Antiepileptika und GP-IIb/IIIa-Antagonisten erhalten ohne Hinweis auf klinisch relevante unerwünschte Interaktionen.

#### 4.6 Fertilität, Schwangerschaft und Stillzeit

#### Schwangerschaft

Da keine klinischen Daten über die Einnahme von Clopidogrel während der Schwangerschaft vorliegen, ist es als Vorsichtsmaßnahme vorzuziehen, Clopidogrel während der Schwangerschaft nicht anzuwenden.

Tierexperimentelle Studien lassen nicht auf direkte oder indirekte schädliche Auswirkungen auf Schwangerschaft, embryonale/fetale Entwicklung, Geburt oder postnatale Entwicklung schließen (siehe Abschnitt 5.3).

# Stillzeit

Es ist nicht bekannt, ob Clopidogrel in die menschliche Muttermilch übergeht. Tierexperimentelle Untersuchungen haben einen Übergang von Clopidogrel in die Muttermilch gezeigt. Als Vorsichtsmaßnahme sollte während der Plavix-Therapie abgestillt werden.

# Fertilität

In Tierstudien konnte nicht nachgewiesen werden, dass Clopidogrel die Fertilität beeinträchtigt.

#### 4.7 Auswirkungen auf die Verkehrstüchtigkeit und die Fähigkeit zum Bedienen von Maschinen

Clopidogrel hat keinen oder vernachlässigbaren Einfluss auf die Verkehrstüchtigkeit und die Fähigkeit zum Bedienen von Maschinen.

# 4.8 Nebenwirkungen

Zusammenfassung des Sicherheitsprofils
Die Sicherheit der Anwendung von Clopidogrel wurde im Rahmen klinischer Studien
an mehr als 44.000 Patienten untersucht.
Mehr als 12.000 dieser Patienten erhielten
das Arzneimittel ein Jahr oder länger. In der
CAPRIE-Studie erwies sich Clopidogrel in
einer Dosierung von 75 mg/Tag insgesamt
als vergleichbar mit ASS in einer Dosierung
von 325 mg/Tag, unabhängig von Alter, Geschlecht und ethnischer Zugehörigkeit. Die

in den Studien CAPRIE, CURE, CLARITY, COMMIT und ACTIVE-A beobachteten klinisch relevanten Nebenwirkungen werden nachfolgend diskutiert. Zusätzlich zu den Erfahrungen im Rahmen klinischer Studien wurden Arzneimittelnebenwirkungen spontan berichtet.

Blutungen sind sowohl in klinischen Studien als auch nach der Markteinführung die häufigsten berichteten Reaktionen, und zwar meistens im ersten Behandlungsmonat.

In der CAPRIE-Studie betrug die Gesamtinzidenz von Blutungen bei Patienten, die entweder mit Clopidogrel oder ASS behandelt wurden, 9,3%. Die Häufigkeit schwerer Blutungen war in der Clopidogrel-Gruppe und in der ASS-Gruppe vergleichbar.

In der CURE-Studie gab es keine zusätzlichen schweren Blutungen unter Clopidogrel plus ASS innerhalb von 7 Tagen nach koronarer Bypassoperation bei Patienten, die die antithrombozytäre Therapie mehr als 5 Tage vor dem Eingriff beendet hatten. Bei Patienten, die die Therapie innerhalb der letzten 5 Tage vor der Bypassoperation beibehalten hatten, betrug die Blutungsrate 9,6% für Clopidogrel plus ASS gegenüber 6,3% für Placebo plus ASS.

In der CLARITY-Studie war die Blutungsrate unter Clopidogrel plus ASS gegenüber Placebo plus ASS erhöht. Die Inzidenz schwerer Blutungen war in beiden Gruppen vergleichbar. Dieses Ergebnis war in allen Subgruppen, definiert nach Basischarakteristika und Art der fibrinolytischen oder Heparin-Therapie, konsistent.

In der COMMIT-Studie war die Rate nicht zerebraler schwerer Blutungen oder zerebraler Blutungen niedrig und ähnlich in beiden Gruppen.

In der ACTIVE-A-Studie war die Rate schwerer Blutungen in der Clopidogrel + ASS-Gruppe höher als in der Placebo + ASS-Gruppe (6,7 % vs. 4,3 %). Schwere Blutungen waren in beiden Gruppen hauptsächlich extrakraniellen Ursprungs (Clopidogrel + ASS-Gruppe: 5,3 %; Placebo + ASS-Gruppe: 3,5 %), vor allem aus dem Gastrointestinaltrakt (3,5 % vs. 1,8 %).

Es traten deutlich mehr intrakranielle Blutungen in der mit Clopidogrel + ASS behandelten Gruppe im Vergleich zu der Placebo + ASS-Gruppe auf (1,4 % bzw. 0,8 %). Es gab keinen statistisch signifikanten Unterschied zwischen den Gruppen in der Rate tödlicher Blutungen (Clopidogrel + ASS-Gruppe: 1,1 %; Placebo + ASS-Gruppe: 0,7 %) und hämorrhagischer Schlaganfälle (0,8 % bzw. 0,6 %).

Tabellarische Auflistung der Nebenwirkungen Nebenwirkungen, die entweder während klinischer Studien oder spontan berichtet wurden, sind in der Tabelle auf Seite 4 aufgelistet. Ihre Häufigkeit ist definiert unter Verwendung der folgenden Einteilung: häufig (≥ 1/100 bis < 1/10), gelegentlich (≥ 1/1.000 bis < 1/100), selten (≥ 1/10.000), nicht bekannt (Häufigkeit auf Grundlage der verfügbaren Daten nicht abschätzbar). Innerhalb jeder Häufigkeitsgruppe werden die Nebenwirkungen nach abnehmendem Schweregrad angegeben.

uar 2018

003345-31445

# Plavix® 75 mg Filmtabletten Plavix® 300 mg Filmtabletten



| Systemorganklasse | Häufig | Gelegentlich | Selten | Sehr selten,<br>nicht bekannt* |
|---|---|---|---|---|
| Erkrankungen des Blutes und<br>des Lymphsystems | | Thrombozytopenie,<br>Leukopenie,<br>Eosinophilie | Neutropenie, inklusive<br>schwerer Neutropenie | thrombotisch-thrombozytopenische<br>Purpura (TTP, siehe Abschnitt 4.4),<br>aplastische Anämie, Panzytopenie,<br>Agranulozytose, schwere Thrombo-<br>zytopenie, erworbene Hämophilie A<br>Granulozytopenie, Anämie |
| Herzerkrankungen | | | | Kounis-Syndrom (allergische vaso-<br>spastische Angina/allergischer<br>Myokardinfarkt) im Zusammenhang<br>mit einer Überempfindlichkeitsreak-<br>tion durch Clopidogrel* |
| Erkrankungen des Immunsystems | | | | Serumkrankheit, anaphylaktische<br>Reaktionen, kreuzreaktive Arznei-<br>mittel-Überempfindlichkeit unter<br>Thienopyridinen (wie z. B. Ticlopidin,<br>Prasugrel) (siehe Abschnitt 4.4)* |
| Psychiatrische Erkrankungen | | | | Halluzinationen, Verwirrtheit |
| Erkrankungen des Nervensystems | | intrakranielle Blutungen<br>(einige Fälle mit<br>tödlichem Ausgang),<br>Kopfschmerzen,<br>Parästhesien, Schwin-<br>del/Benommenheit | | Geschmacksstörungen, Ageusie |
| Augenerkrankungen | | Augenblutungen (kon-<br>junktival, okular, retinal) | | |
| Erkrankungen des Ohrs und des Labyrinths | | | Vertigo | |
| Gefäßerkrankungen | Hämatome | | | schwere Blutungen, Blutungen<br>operativer Wunden, Vaskulitis,<br>Hypotonie |
| Erkrankungen der Atemwege, des<br>Brustraums und Mediastinums | Epistaxis | | | Atemwegsblutungen<br>(Hämoptyse, Lungenblutungen),<br>Bronchospasmen, interstitielle<br>Pneumonie, eosinophile<br>Pneumonie |
| Erkrankungen des Gastro-<br>intestinaltrakts | gastrointestinale<br>Blutungen, Durchfall,<br>Bauchschmerzen,<br>Dyspepsie | Ulcus ventriculi<br>und Ulcus duodeni,<br>Gastritis, Erbrechen,<br>Übelkeit, Verstopfung,<br>Flatulenz | retroperitoneale<br>Blutungen | gastrointestinale und retroperito-<br>neale Blutungen mit tödlichem<br>Ausgang, Pankreatitis, Kolitis<br>(einschließlich ulzeröser und<br>lymphozytärer Kolitis), Stomatitis |
| Leber- und Gallenerkrankungen | | | | akutes Leberversagen, Hepatitis,<br>Leberwerte außerhalb der Norm |
| Erkrankungen der Haut und<br>des Unterhautzellgewebes | Bluterguss | Ausschlag, Juckreiz,<br>Blutungen der Haut<br>(Purpura) | | bullöse Dermatitis (toxische epidei male Nekrolyse, Stevens-Johnson Syndrom, Erythema multiforme, akut generalisiertes pustulöses Exanthem [AGEP]), Angioödem, Arzneimittel-induziertes Hypersensitivitätssyndrom, Arzneimittel-exanthem mit Eosinophilie und systemischen Symptomen (DRESS erythematöses oder exfoliatives Exanthem, Urtikaria, Ekzem, Lichen planus |
| Erkrankungen der Geschlechts-<br>organe und der Brustdrüse | | | Gynäkomastie | |
| Skelettmuskulatur-, Bindegewebs-<br>und Knochenerkrankungen | | | | Blutungen im Muskel- bzw.<br>Skelettbereich (Hämarthrose),<br>Arthritis, Arthralgie, Myalgie |
| Erkrankungen der Nieren und<br>Harnwege | | Hämaturie | | Glomerulonephritis, Anstieg des Serumkreatinins |
| Allgemeine Erkrankungen und Be-<br>schwerden am Verabreichungsort | Blutung an Punktionsstellen | | | Fieber |
| Untersuchungen | | Blutungszeit verlängert, Neutrophilenzahl vermindert, Thrombozytenzahl vermindert | | |

<sup>\*</sup>Angaben beziehen sich auf Clopidogrel mit Häufigkeit "nicht bekannt".

4 003345-31445



# Plavix® 75 mg Filmtabletten Plavix® 300 mg Filmtabletten

Meldung des Verdachts auf Nebenwirkun-

Die Meldung des Verdachts auf Nebenwirkungen nach der Zulassung ist von großer Wichtigkeit. Sie ermöglicht eine kontinuierliche Überwachung des Nutzen-Risiko-Verhältnisses des Arzneimittels. Angehörige von Gesundheitsberufen sind aufgefordert, jeden Verdachtsfall einer Nebenwirkung über das aufgeführte nationale Meldesystem anzuzeigen.

Deutschland Bundesinstitut für Arzneimittel und Medizinprodukte Abt. Pharmakovigilanz Kurt-Georg-Kiesinger-Allee 3 D-53175 Bonn Website: http://www.bfarm.de

Österreich Bundesamt für Sicherheit im Gesundheitswesen Traisengasse 5 A-1200 Wien Fax: +43 (0) 50 555 36207 Website: http://www.basg.gv.at

#### 4.9 Überdosierung

Eine Clopidogrel-Überdosis kann zu verlängerter Blutungszeit und anschließenden Blutungskomplikationen führen. Eine angemessene Therapie sollte in Erwägung gezogen werden, wenn Blutungen beobachtet werden.

Ein Antidot zu Clopidogrel ist bisher nicht bekannt. Wenn eine rasche Normalisierung der Blutungszeit notwendig ist, könnte eine Plättchentransfusion die Wirkung von Clopidogrel aufheben.

#### 5. PHARMAKOLOGISCHE EIGEN-SCHAFTEN

# 5.1 Pharmakodynamische Eigenschaften

Pharmakotherapeutische Gruppe: Thrombozytenaggregationshemmer, exkl. Heparin, ATC-Code: B01AC-04.

# Wirkmechanismus

Clopidogrel ist ein Prodrug. Einer seiner Metaboliten ist ein Inhibitor der Thrombozy tenaggregation. Clopidogrel muss durch CYP450-Enzyme metabolisiert werden, um den aktiven Metaboliten, der die Thrombozytenaggregation hemmt, zu bilden. Der aktive Metabolit von Clopidoarel hemmt selektiv die Bindung von Adenosindiphosphat (ADP) an dessen Thrombozytenrezeptor (P2Y<sub>12</sub>) und die nachfolgende ADP-vermittelte Aktivierung des Glykoprotein-(GP-)IIb/IIIa-Komplexes, so dass es zu einer Hemmung der Thrombozytenaggregation kommt. Aufgrund der irreversiblen Bindung sind Thrombozyten für den Rest ihrer Lebenszeit (ungefähr 7-10 Tage) beeinträchtigt und die Wiederherstellung der normalen Thrombozytenfunktion entspricht der Geschwindigkeit der Thrombozytenneubildung. Darüber hinaus hemmt Clopidogrel auch die durch andere Substanzen ausgelöste Thrombozytenaggregation, indem die Verstärkung der Thrombozytenaktivierung durch das freigesetzte ADP gehemmt wird.

Da der aktive Metabolit durch CYP450-Enzyme gebildet wird (einige davon unterliegen einem genetischen Polymorphismus oder können durch andere Arzneimittel gehemmt werden), werden nicht alle Patienten eine ausreichende Thrombozytenaggregationshemmung haben.

# Pharmakodynamische Wirkungen

Wiederholte Gaben von täglich 75 mg führten bereits ab dem ersten Tag zu einer ausgeprägten Hemmung der ADP-vermittelten Thrombozytenaggregation, die stetig zunahm und zwischen dem 3. und dem 7. Tag einen Steady State erreichte. Bei Erreichen des Steady State mit einer täglichen Dosierung von 75 mg betrug die durchschnittliche Hemmung zwischen 40% und 60%. Die Thrombozytenaggregation und Blutungszeit normalisierten sich im Allgemeinen innerhalb von 5 Tagen nach Beendigung der Therapie.

#### Klinische Wirksamkeit und Sicherheit

Die Wirksamkeit und Verträglichkeit von Clopidogrel wurden in 5 Doppelblindstudien mit über 88.000 Patienten untersucht: in der CAPRIE-Studie, ein Vergleich von Clopidogrel und ASS, und in den vier Studien CURE, CLARITY, COMMIT und ACTIVE-A, in denen Clopidogrel mit Placebo, jeweils in Kombination mit ASS und anderen Standardtherapien. verglichen wurde.

Kurz zurückliegender Myokardinfarkt (MI) oder Schlaganfall sowie nachgewiesene periphere arterielle Verschlusskrankheit An der CAPRIE-Studie nahmen 19.185 Patienten mit Atherothrombose teil, die durch einen kürzlich erfolgten Herzinfarkt (< 35 Tage), einen kürzlich erfolgten ischämischen Schlaganfall (zwischen 7 Tagen und 6 Monaten) oder durch nachgewiesene periphere arterielle Verschlusskrankheit (pAVK) in Erscheinung trat. Die Patienten erhielten nach Randomisierung entweder 75 mg/Tag Clopidogrel oder 325 mg/Tag ASS und wurden 1 bis 3 Jahre beobachtet. In der Herzinfarkt-Subgruppe erhielten die meisten Patienten in den ersten Tagen nach dem akuten Infarkt

Clopidogrel reduzierte signifikant die Inzidenz von erneuten ischämischen Ereignissen (kombinierter Endpunkt von Herzinfarkt, Schlaganfall und vaskulär bedingtem Tod) im Vergleich zu ASS. In der "Intention-totreat"-Analyse wurden in der Clopidogrel-Gruppe 939 Ereignisse und in der ASS-Gruppe 1.020 Ereignisse beobachtet (relative Risikoreduktion [RRR] von 8,7 % [95 % CI: 0.2 bis 16.41: p = 0.045). Dies bedeutet dass pro 1,000 Patienten, die 2 Jahre lang behandelt werden, bei zusätzlich 10 Patienten (CI: 0 bis 20) unter Clopidogrel im Vergleich zu ASS ein erneutes ischämisches Ereignis verhindert wird. Die Analyse der Gesamtmortalität als sekundärer Endpunkt zeigte keinen signifikanten Unterschied zwischen Clopidogrel (5,8%) und ASS (6,0%).

In einer Subgruppenanalyse nach dem entsprechenden qualifizierenden Ereignis (Herzinfarkt, ischämischer Schlaganfall, pAVK) schien der Nutzen am stärksten (statistisch signifikant, p = 0,003) in der pAVK-Gruppe ausgeprägt zu sein (insbesondere bei Patienten, die in ihrer Vergangenheit auch einen Herzinfarkt erlitten hatten, RRR = 23,7 %; CI: 8,9 bis 36,2) und schien geringer (kein signifikanter Unterschied zu ASS) ausgeprägt in der Schlaganfall-Gruppe

(RRR = 7,3%; Cl: -5,7 bis 18,7 [p = 0,258]). Bei Patienten, die ausschließlich wegen eines kürzlich erfolgten Herzinfarktes in die Studie aufgenommen wurden, war Clopidogrel zahlenmäßig unterlegen, aber nicht statistisch unterschiedlich zu ASS (RRR = -4,0%; Cl: -22,5 bis 11,7 [p = 0,639]). Darüber hinaus legt eine Subgruppenanalyse nach Alter nahe, dass der Nutzen von Clopidogrel bei Patienten über 75 Jahre geringer war als der bei Patienten ≤ 75 Jahre.

Da die CAPRIE-Studie nicht darauf ausgelegt wurde, die Wirksamkeit in den einzelnen Subgruppen zu evaluieren, ist unklar, ob die Unterschiede in der relativen Risikoreduktion je nach qualifizierendem Ereignis tatsächlich bestehen oder zufallsbedingt sind.

# Akutes Koronarsyndrom

In die CURE-Studie wurden 12.562 Patienten mit akutem Koronarsyndrom ohne ST-Strecken-Hebung (instabile Angina Pectoris oder Non-Q-Wave-Myokardinfarkt) eingeschlossen, die sich innerhalb von 24 Stunden nach der jüngsten Brustschmerzepisode oder ischämietypischen Beschwerden vorgestellt hatten. Zum Einschluss in die Studie mussten die Patienten entweder EKG-Veränderungen, vereinbar mit einer neu aufgetretenen Ischämie, erhöhte kardiale Enzyme oder mindestens zweifach erhöhte Troponin-I- oder -T-Spiegel aufweisen. Die Patienten wurden zu Clopidogrel (300 mg einmalige Aufsättigungsdosis mit anschließend 75 mg/Tag, n = 6.259) oder Placebo (n = 6.303), jeweils in Kombination mit ASS (75-325 mg einmal täglich) und anderen Standardtherapien, randomisiert. Die Patienten wurden bis zu einem Jahr lang behandelt. In der CURE-Studie wurden 823 (6,6%) Patienten begleitend mit GP-IIb/IIIa-Rezeptorantagonisten behandelt. Heparine wurden bei über 90 % der Patienten eingesetzt, und die relative Blutungsrate zwischen Clopidogrel und Placebo wurde durch die begleitende Heparin-Therapie nicht signifi-

Die Zahl der Patienten, die den primären Endpunkt (kardiovaskulärer [CV] Tod. Mvokardinfarkt [MI] oder Schlaganfall) erreichten. betrug in der Clopidogrel-Gruppe 582 (9,3%) und in der Placebo-Gruppe 719 (11,4%) - eine 20%ige Reduktion des relativen Risikos (95% CI von 10-28%; p = 0,00009) zu Gunsten der Clopidogrel-Gruppe. Die relative Risikoreduktion betrug 17%, wenn Patienten konservativ behandelt wurden, 29 %, wenn bei den Patienten eine perkutane transluminale koronare Angioplastie (PTCA) mit oder ohne Stent-Implantation durchgeführt wurde, und 10%, wenn eine aortokoronare Bypassoperation durchgeführt wurde. Neue kardiovaskuläre Ereignisse (primärer Endpunkt) wurden in den jeweiligen Studienintervallen 0-1, 1-3, 3-6, 6-9 und 9-12 Monate verhindert mit einer relativen Risikoreduktion von 22% (CI: 8,6; 33,4), von 32 % (CI: 12,8; 46,4), von 4 % (CI: -26,9; 26,7), von 6% (CI: -33,5; 34,3) bzw. von 14 % (CI: -31,6; 44,2). Über eine Behandlungsdauer von 3 Monaten hinaus verstärkte sich also der Nutzen, der in der Clopidogrel + ASS behandelten Gruppe beobachtet wurde, nicht weiter, wohingegen das Blutungsrisiko persistierte (siehe Abschnitt 4.4).

anuar 2018

003345-31445

# Plavix® 75 mg Filmtabletten Plavix® 300 mg Filmtabletten

SANOFI 🗳

Die Anwendung von Clopidogrel in der CURE-Studie war assoziiert mit einem verminderten Bedarf an thrombolytischer Therapie (RRR = 43,3%; Cl: 24,3%; 57,5%) und an GP-Ilb/Illa-Rezeptorantagonisten (RRR = 18,2%; Cl: 6,5%; 28,3%).

Die Zahl der Patienten, die den co-primären Endpunkt erreichten (CV-Tod, MI, Schlaganfall oder refraktäre Ischämie), betrug in der Clopidogrei-Gruppe 1.035 (16,5%) und in der Placebo-Gruppe 1.187 (18,8%) – eine relative Risikoreduktion zu Gunsten der Clopidogrei-Gruppe von 14% (95% CI von 6–21%, p = 0,0005). Dieser Nutzen war primär bedingt durch die statistisch signifikante Senkung der Herzinfarkt-Inzidenz (287 (4,6%) in der Clopidogrei-Gruppe und 363 [5,8%] in der Placebo-Gruppe). Auf die Rate der Rehospitalisierungen aufgrund von instabiler Angina Pectoris wurde keine Wirkung beobachtet.

Die Ergebnisse, die in Patientenpopulationen mit unterschiedlichen Charakteristika (z.B. instabile Angina Pectoris oder Non-Q-Wave-Myokardinfarkt, niedriger bis hoher Risikograd, Diabetes mellitus, Revaskularisationspflichtigkeit, Alter, Geschlecht etc.) erzielt wurden, waren konsistent mit den Resultaten der primären Analyse. Insbesondere konnte in einer Post-hoc-Analyse mit 2.172 Patienten (17 % der Gesamtpopulation der CURE-Studie), die einer Stent-Implantation unterzogen wurden, gezeigt werden, dass Clopidogrel im Vergleich zu Placebo eine signifikante RRR um 26,2% in Bezug auf den co-primären Endpunkt (CV-Tod, MI, Schlaganfall) und eine ebenfalls signifikante RRR um 23,9 % für den zweiten co-primären Endpunkt (CV-Tod, MI Schlaganfall oder refraktäre Ischämie) erzielte. Außerdem warf das Sicherheitsprofil von Clopidogrel in dieser Subgruppe keine besonderen Bedenken auf. Daher stehen die Ergebnisse dieser Untergruppe im Einklang mit den Ergebnissen der gesamten Studie.

Der Nutzen von Clopidogrel war unabhängig von anderen akut oder langfristig durch-geführten kardiovaskulären Therapien (z. B. Heparin/NMH, GP-Ilb/Illa-Rezeptorantagonisten, Lipidsenker, Betablocker und ACE-Inhibitoren). Die Wirksamkeit von Clopidogrel war unabhängig von der ASS-Dosis (75–325 mg einmal täglich).

Die Wirksamkeit und Verträglichkeit von Clopidogrel bei Patienten mit akutem ST-Hebungs-Myokardinfarkt wurden in zwei randomisierten, placebokontrollierten Doppelblindstudien, CLARITY und COMMIT, untersucht.

In die CLARITY-Studie wurden 3.491 Patienten innerhalb von 12 Stunden nach Beginn eines akuten ST-Hebungsinfarkts und geplanter thrombolytischer Therapie eingeschlossen. Die Patienten erhielten Clopidogrel (300-mg-Aufsättigungsdosis, gefolgt von 75 mg/Tag, n = 1.752) oder Placebo (n = 1.739), beide Gruppen in Kombination mit ASS (150 bis 325 mg als Aufsättigungsdosis, gefolgt von 75 mg bis 162 mg/Tag), eine fibrinolytische Substanz und, wo angezeigt, Heparin. Die Patienten wurden über 30 Tage nachbeobachtet. Der primäre Endpunkt war das Auftreten eines kombinierten Endpunkts: ein vor der Entlassung angio-

graphisch nachgewiesener Verschluss der infarktzugehörigen Arterie, Tod oder Reinfarkt vor der Koronarangiographie. Für Patienten, die keiner Angiographie unterzogen wurden, bestand der primäre Endpunkt aus Tod oder Reinfarkt bis Tag 8 oder bis zur Krankenhausentlassung. Der Anteil an Frauen in der untersuchten Patientenpopulation lag bei 19,7 %, der Anteil der Patienten ≥ 65 Jahre bei 29,2 %. Insgesamt erhielten 99,7 % der Patienten Fibrinolytika (fibrinspezifisch: 68,7 %, nicht fibrinspezifisch: 31,1 %), 89,5 % Heparin, 78,7 % Betablocker, 54,7 % ACE-Hemmer und 63 % Statine.

Fünfzehn Prozent (15,0%) der Patienten in der Clopidogrel-Gruppe und 21,7% in der Placebo-Gruppe erreichten den primären Endpunkt. Dies entspricht einer absoluten Risikoreduktion von 6,7 Prozentpunkten und einer Odds-Ratio-Reduktion von 36% zu Gunsten von Clopidogrel (95% Cl: 24, 47%; p < 0,001), hauptsächlich beruhend auf der Reduktion von Verschlüssen infarktbezogener Arterien. Dieser Vorteil war konsistent in allen präspezifizierten Subgruppen einschließlich Alter und Geschlecht der Patienten, Infarktlokalisation und Art des Fibrinolytikums oder Heparins.

In die COMMIT-Studie (2 x 2-faktorielles Design) wurden 45.852 Patienten eingeschlossen, die sich innerhalb von 24 Stunden nach Auftreten von Symptomen mit Verdacht auf Herzinfarkt und typischen EKG-Veränderungen (z.B. ST-Strecken-Hebung, ST-Strecken-Senkung oder Linksschenkelblock) vorstellten. Die Patienten erhielten Clopidogrel (75 mg/Tag, n = 22.961) oder Placebo (n = 22.891) in Kombination mit ASS (162 mg/Tag) für 28 Tage oder bis zur Krankenhausentlassung. Die co-primären Endpunkte waren Tod jeglicher Ursache bzw. das erste Auftreten eines Reinfarktes, eines Schlaganfalls oder Todes.

Der Anteil an Frauen in der untersuchten Patientenpopulation lag bei 27,8%, der Anteil der Patienten  $\geq 60$  Jahre bei 58,4% (26%  $\geq 70$  Jahre) und 54,5% erhielten Fibrinolytika.

Clopidogrel senkte signifikant das relative Risiko für Tod jeglicher Ursache um 7 % (p = 0,029) und das relative Risiko der Kombination aus Reinfarkt, Schlaganfall und Tod um 9% (p = 0,002), entsprechend einer absoluten Risikoreduktion von 0,5 % bzw. 0,9 %. Dieser Vorteil war konsistent über Alter, Geschlecht und mit oder ohne Anwendung von Fibrinolytika und wurde bereits nach 24 Stunden beobachtet.

# Vorhofflimmern

In die ACTIVE-W- und die ACTIVE-A-Studie, gesonderte Prüfungen innerhalb des ACTIVE-Programms, wurden Patienten mit Vorhofflimmern (VHF) aufgenommen, die wenigstens einen Risikofaktor für vaskuläre Ereignisse aufwiesen.

Auf Grundlage der Einschlusskriterien schlossen Ärzte Patienten in die ACTIVE-W ein, wenn diese Kandidaten für eine Therapie mit Vitamin-K-Antagonisten (VKA, wie z. B. Warfarin) waren. In die ACTIVE-A-Studie wurden Patienten aufgenommen, die keine VKA-Therapie erhalten konnten,

weil sie ungeeignet waren oder die Therapie ablehnten.

Die ACTIVE-W-Studie zeigte, dass eine Behandlung mit Vitamin-K-Antagonisten wirksamer war als mit Clopidogrel und ASS

Die ACTIVE-A-Studie (n = 7.554) war eine randomisierte, doppelblinde, placebokontrollierte Multicenter-Studie, die Clopidogrel 75 mg/Tag + ASS (n = 3.772) mit Placebo + ASS (n = 3.782) verglichen hat. Die empfohlene Dosis für ASS war 75–100 mg/Tag. Patienten wurden bis zu 5 Jahre behandelt.

Patienten, die im ACTIVE-Programm randomisiert wurden, zeichneten sich durch nachgewiesenes Vorhofflimmern aus, d.h. entweder permanentes VHF oder wenigstens zwei Episoden von intermittierendem VHF in den letzten sechs Monaten und wenigstens einen der folgenden Risikofaktoren:

Alter ≥ 75 Jahre oder Alter zwischen 55 und 74 Jahren und entweder Diabetes mellitus, der eine medikamentöse Therapie erfordert, einen bereits nachgewiesenen Myokardinfarkt oder eine bekannte koronare Herzkrankheit, behandelter systemischer Bluthochdruck, vorheriger Schlaganfall, transitorisch ischämische Attacke (TIA) oder nicht zerebraler systemischer Embolus, linksventrikulären Ejektionsfraktion < 45 % oder eine nachgewiesene periphere Verschlusskrankheit. Der mittlere CHADS₂-Score betrug 2.0 (Bereich 0 – 6).

Die wichtigen Ausschlusskriterien für Patienten waren peptisches Ulkus innerhalb der vorangegangenen 6 Monate, frührer intrazerebrale Blutungen, signifikante Thrombozytopenie (Plättchenzahl < 50 × 10<sup>9</sup>/l), Bedarf an Clopidogrel oder einem oralen Antikagulans (OAC) oder Unverträglichkeit gegenüber einem der beiden Wirkstoffe.

Dreiundsiebzig Prozent (73%) der in der ACTWE-A-Studie eingeschlossenen Patienten konnten aufgrund der ärztlichen Einschätzung, einer unzuverlässigen INR-Kontrolle ("International Normalized Ratio"), der Neigung zu Stürzen und Schädeltraumen oder eines spezifischen Blutungsrisikos keine VKA einnehmen; bei 26% der Patienten gründete sich die ärztliche Entscheidung auf der Ablehnung des Patienten, VKA einzuhehmen

Der Anteil an Frauen in der Patientengruppe lag bei 41,8%. Das Durchschnittsalter betrug 71 Jahre, 41,6% der Patienten waren ≥ 75 Jahre. Insgesamt 23,0% der Patienten erhielten Antiarrhythmika, 52,1% Betablocker, 54,6% ACE-Inhibitoren und 25,4% Statine

Die Anzahl der Patienten, die den primären Endpunkt erreichten (Zeitpunkt des ersten Auftretens von Schlaganfall, MI, nicht zerebraler systemischer Embolie, vaskulär bedingtem Tod), lag bei 832 (22,1%) in der Clopidogrel + ASS-Gruppe und bei 924 (24,4%) in der Placebo + ASS-Gruppe (relative Risikoreduktion 11,1%; 95% CI von 2,4% bis 19,1%; p = 0,013), vor allem durch die reduzierte Häufigkeit von Schlaganfällen. Schlaganfälle traten bei 296 Patienten (7,8%) auf, die Clopidogrel + ASS erhielten, und bei 408 Patienten (10,8%),

003345-31445



Plavix® 75 mg Filmtabletten Plavix® 300 mg Filmtabletten

die Placebo + ASS erhielten (relative Risikoreduktion 28,4%; 95% Cl von 16,8% bis 38,3%; p=0,00001).

#### Kinder und Jugendliche

In einer Dosis-Eskalationsstudie mit 86 Neugeborenen und Kleinkindern bis zu einem Alter von 24 Monaten mit einem Thrombose-Risiko (PICOLO) wurde Clopidogrel in den aufeinander folgenden Dosierungen 0,01, 0,1 und 0,2 mg/kg bei Neugeborenen und Kleinkindern und 0,15 mg/kg nur bei Neugeborenen untersucht. Die Dosis von 0,2 mg/kg führte zu einer mittleren prozentualen Hemmung von 49,3% (5 µM ADP-induzierte Thrombozytenaggregation), die damit vergleichbar ist mit der bei Erwachsenen, die täglich Plavix 75 mg einnehmen.

In einer randomisierten, doppelblinden Parallelgruppen-Studie (CLARINFT) wurden 906 pädiatrische Patienten (Neugeborene und Säuglinge) mit angeborenem zyanotischem Herzfehler nach systemisch-pulmonaler Shuntanlage randomisiert und erhielten entweder 0,2 mg/kg Clopidogrel (n = 467) oder Placebo (n = 439) neben gleichzeitiger Basistherapie bis zum Zeitpunkt der zweistufigen Operation. Die mittlere Zeit zwischen Shunt-Anlage und erster Anwendung der Studienmedikation betrug 20 Tage. Ungefähr 88 % der Patienten erhielten gleichzeitig ASS (in einem Bereich von 1 bis 23 mg/kg/Tag). Es gab keinen signifikanten Unterschied zwischen den Gruppen in Bezug auf die primären, kombinierten Endpunkte Tod, Shunt-Thrombose oder kardiovaskulärassoziierte Intervention vor einem Alter bis zu 120 Tagen nach einem thrombotischen Ereignis (89 [19.1%] in der Clopidogrel-Gruppe und 90 [20,5%] in der Placebo-Gruppe) (siehe Abschnitt 4.2). Blutungen waren die häufigste berichtete Nebenwirkung sowohl in der Clopidogrel- als auch in der Placebo-Gruppe: es gab iedoch keinen signifikanten Unterschied in der Blutungsrate zwischen den beiden Gruppen. In der Langzeitnachbeobachtung zur Klärung der Unbedenklichkeit erhielten 26 Patienten, bei denen im Alter von einem Jahr noch ein Shunt vorhanden war, Clopidogrel bis zu einem Alter von 18 Monaten. Sicherheitsbedenken wurden während dieser Langzeitnachbeobachtung nicht festgestellt.

Die CLARINET- und PICOLO-Studie wurden mit einer zubereiteten Clopidogrel-Lösung durchgeführt. In einer relativen Bioverfügbarkeitsstudie mit Erwachsenen zeigte diese Clopidogrel-Lösung im Vergleich zur zugelassenen Tablette eine ähnliche Größenordnung und eine leicht erhöhte Rate der Absorption, bezogen auf den hauptsächlich zirkulierenden (inaktiven) Metaboliten.

# 5.2 Pharmakokinetische Eigenschaften

# Resorption

Clopidogrel wird nach einmaliger und wiederholter Einnahme von täglich 75 mg rasch resorbiert. Mittlere Peakplasmaspiegel des unveränderten Clopidogrels (ungefähr 2,2–2,5 ng/ml nach einer einmaligen oralen Gabe von 75 mg) werden ungefähr 45 min nach der Einnahme erreicht. Bezogen auf die im Urin ausgeschiedenen Clopidogrel-Metaboliten beträgt die Resorptionsrate mindestens 50 %.

Clopidogrel und der hauptsächlich zirkulierende (inaktive) Metabolit binden *in vitro* reversibel an menschliche Plasmaproteine (jeweils zu 98 % und 94 %). *In vitro* bleibt die Bindung über einen weiten Konzentrationsbereich ungesättigt.

#### Biotransformation

Verteiluna

Clopidogrel wird weitgehend in der Leber metabolisiert. In vitro und in vivo wird Clopidogrel über zwei Hauptwege verstoffwechselt: Einerseits wird Clopidogrel durch Esterasen hydrolysiert, wobei das inaktive Carboxylsäurederivat entsteht (85 % der zirkulierenden Metaboliten), und andererseits wird ein zweiter Weg über mehrere Cytochrome P450 vermittelt. Clopidogrel wird zuerst zu einem 2-Oxo-Clopidogrel-Zwischenprodukt metabolisiert. Nachfolgende Metabolisierung des 2-Oxo-Clopidogrel-Zwischenproduktes ergibt die Bildung des aktiven Metaboliten (ein Thiolderivat von Clopidogrel). Der aktive Metabolit wird hauptsächlich durch CYP2C19 gebildet mit Beteiligung mehrerer anderer CYP-Enzyme einschließlich CYP1A2, CYP2B6 und CYP3A4. Der aktive Thiolmetabolit, der in vitro isoliert wurde, bindet schnell und irreversibel an Thrombozytenrezeptoren und hemmt dadurch die Thrombozytenaggregation.

 $\rm C_{max}$  des aktiven Metaboliten ist nach einmaliger Gabe der 300-mg-Aufsättigungsdosis doppelt so hoch wie nach 4-tägiger Gabe der 75-mg-Erhaltungsdosis.  $\rm C_{max}$  wird etwa 30–60 Minuten nach Einnahme erreicht.

# Elimination

Nach Gabe einer oralen Dosis von <sup>14</sup>C-markiertem Clopidogrel wurden beim Menschen innerhalb von 120 Stunden ca. 50 % im Urin und ca. 46 % im Stuhl ausgeschieden. Nach einer einmaligen oralen Gabe von 75 mg hat Clopidogrel eine Halbwertszeit von ungefähr 6 Stunden. Die Eliminationshalbwertszeit des hauptsächlich zirkulierenden (inaktiven) Metaboliten betrug sowohl nach einmaliger als auch nach wiederholter Gabe 8 Stunden.

# Pharmakogenetik

CYP2C19 ist sowohl an der Bildung des aktiven Metaboliten wie auch an der des 2-Oxo-Clopidogrel-Zwischenproduktes beteiligt. Die Pharmakokinetik des aktiven Metaboliten von Clopidogrel und der thrombozytenaggregationshemmende Effekt (gemessen mit Ex-vivo-Thrombozytenaggregationsassays) unterscheiden sich in Abhängigkeit vom CYP2C19-Genotyp.

Das CYP2C19\*1-Allel korrespondiert mit voll funktionsfähigem Metabolismus, während die CYP2C19\*2- und CYP2C19\*3-Allele mit einem nicht funktionsfähigen Metabolismus korrespondieren. Die CYP2C19\*2- und CYP2C19\*3-Allele machen die Mehrheit der Allele mit reduzierter Funktion bei kaukasischen (85%) und bei asiatischen (99%) Langsam-Metabolisierern aus. Andere Allele, die mit einem fehlenden oder verringerten Metabolismus verbunden sind, sind weniger häufig und schließen CYP2C19\*4, \*5, \*6, \*7 und \*8 ein. Ein Patient mit Langsam-Metabolisierer-Status trägt zwei Loss-of-Function-Allele, wie oben definiert. Die publizierten

Häufigkeiten für den langsamen CYP2C19-Metabolisierer-Genotyp sind etwa 2 % für Kaukasier, 4 % für Schwarze und 14 % für Chinesen. Es sind Tests verfügbar, mit denen der CYP2C19-Genotyp der Patienten bestimmt werden kann.

Eine Crossover-Studie mit 40 Gesunden. 10 aus jeder CYP2C19-Metabolisierer-Gruppe (ultraschnell, schnell, intermediär, langsam), untersuchte die Pharmakokinetik und die Hemmung der Thrombozytenaggregation unter Anwendung von 300 mg, gefolgt von 75 mg/Tag, und 600 mg, gefolgt von 150 mg/Tag, jeweils über 5 Tage (Steady State). Es wurden keine erheblichen Unterschiede in der Exposition gegenüber dem aktiven Metaboliten und der durchschnittlichen Hemmung der Thrombozytenaggregation zwischen den Ultraschnell-, Schnellund Intermediär-Metabolisierern beobachtet. Bei den langsamen Metabolisierern war die Exposition gegenüber dem aktiven Metaboliten im Vergleich zu schnellen Metabolisierern um 63-71 % vermindert.

Durch die 300-mg-/75-mg-Dosierung wurde die Hemmung der Thrombozytenaggregation in Langsam-Metabolisierern mit einer durchschnittlichen Inhibition der Plättchenaggregation (IPA; 5  $\mu\text{M}$  ADP) von 24% (24 Stunden) und 37 % (Tag 5) vermindert, im Vergleich zu einer durchschnittlichen IPA von 39 % (24 Stunden) und 58 % (Tag 5) bei schnellen Metabolisierern und 37 % (24 Stunden) und 60 % (Tag 5) bei intermediären Metabolisierern. Wenn langsame Metabolisierer 600 mg/150 mg erhielten, war die Exposition gegenüber dem aktiven Metaboliten von Clopidogrel größer als mit der 300-mg-/75-mg-Dosierung. Außerdem betrug die IPA 32% (24 Stunden) und 61% (Tag 5) und war damit höher als bei langsamen Metabolisierern, die die 300-mg-/ 75-mg-Dosierung erhielten, und vergleichbar mit den anderen CYP2C19-Metabolisierer-Gruppen, die die 300-mg-/75-mg-Dosierung erhielten. Eine geeignete Dosierung für diese Patientenpopulation wurde noch nicht in klinischen Ergebnisstudien ermittelt.

In Übereinstimmung mit den oben genannten Ergebnissen konnte in einer Meta-Analyse von 6 Studien mit 335 Clopidogrel-benandelten Patienten im Steady State gezeigt werden, dass die Exposition gegenüber dem aktiven Metaboliten um 28% bei Intermediär-Metabolisierern und um 72% bei Langsam-Metabolisierern reduziert war, während die Hemmung der Thrombozytenaggregation (5 μM ADP) mit Unterschieden in der IPA (Inhibition der Plättchenaggregation) von 5,9% bzw. 21,4% im Vergleich zu den schnellen Metabolisierern reduziert war

Der Einfluss des CYP2C19-Genotyps auf den klinischen Nutzen für Patienten, die mit Clopidogrel behandelt werden, wurde in prospektiven, randomisierten, kontrollierten Studien nicht untersucht. Es gab jedoch etliche retrospektive Auswertungen, die diesen Effekt in Patienten, die mit Clopidogrel behandelt wurden, untersucht haben und für die Genotypisierungen vorliegen: CURE (n = 2.721), CHARISMA (n = 2.428), CLARITY-TIMI 28 (n = 227), TRITON-TIMI 38 (n = 1.477) und ACTIVE-A (n = 601) sowie etliche veröffentlichte Kohortenstudien.

003345-31445

2018

# Plavix® 75 mg Filmtabletten Plavix® 300 mg Filmtabletten

In der TRITON-TIMI 38- und 3 Kohortenstudien (Collet, Sibbing, Giusti) hatte eine kombinierte Gruppe von Patienten mit entweder Intermediär- oder Langsam-Metabolisierer-Status eine höhere Rate an kardiovaskulären Ereignissen (Tod, Myokardinfarkt und Schlaganfall) oder Stentthrombosen im Vergleich zu den schnellen Metabolisierern.

In der CHARISMA- und einer Kohortenstudie (Simon) wurde eine erhöhte Ereignisrate nur bei den Langsam-Metabolisierern im Vergleich zu den schnellen Metabolisierern beobachtet.

In der CURE-, CLARITY-, ACTIVE-A- und einer Kohortenstudie (Trenk) konnte keine erhöhte Ereignisrate anhand des Metabolisierungsstatus festgestellt werden.

Keine dieser Studien hatte einen angemessenen Umfang, um Unterschiede in Bezug auf das klinische Ergebnis bei langsamen Metabolisierern festzustellen.

#### Spezielle Populationen

Die Pharmakokinetik des aktiven Metaboliten von Clopidogrel ist in diesen speziellen Populationen nicht bekannt.

#### Niereninsuffizienz

Nach wiederholter Clopidogrel-Gabe von 75 mg/Tag bei Personen mit schweren Nierenfunktionsstörungen (Kreatinin-Clearance von 5 bis 15 ml/min) war die Hemmung der ADP-induzierten Thrombozytenaggregation geringer (25 %) als bei Personen mit normaler Nierenfunktion, jedoch war die Verlängerung der Blutungszeit ähnlich wie bei Personen mit normaler Nierenfunktion, die 75 mg Clopidogrel pro Tag erhielten. Außerdem war die Verträglichkeit bei allen Patienten gut.

# Leberfunktionsstörung

Nach wiederholter Gabe von 75 mg Clopidogrel pro Tag über 10 Tage bei Patienten mit schweren Leberfunktionsstörungen ist die Hemmung der ADP-induzierten Thrombozytenaggregation vergleichbar mit der, die bei gesunden Patienten beobachtet worden ist. Die mittlere Verlängerung der Blutungszeit war auch in beiden Gruppen ähnlich.

# Rasse

Die Prävalenz von CYP2C19-Allelen, die eine mittelstarke oder schwache CYP2C19-Metabolisierung hervorrufen, ist unterschiedlich in Abhängigkeit von Rasse/Ethnie (siehe Abschnitt Pharmakogenetik). In der Literatur sind nur begrenzte Daten asiatischer Populationen verfügbar, um die klinischen Auswirkungen der CYP-Genotypen auf die klinischen Ergebnisse zu bewerten.

# 5.3 Präklinische Daten zur Sicherheit

In präklinischen Studien an Ratten und Pavianen wurden am häufigsten Veränderungen der Leberwerte beobachtet. Diese traten nach einer mindestens 25-fachen Überdosierung auf (im Vergleich zu der beim Menschen eingesetzten Tagesdosis von 75 mg) und sind auf eine Beeinflussung der metabolisierenden Leberenzyme zurückzuführen. Kein Effekt auf die metabolisierenden Leberenzyme wurde bei Menschen beobachtet, die Clopidogrel in der therapeutischen Dosis erhielten.

In sehr hohen Dosierungen wurde sowohl bei der Ratte als auch beim Pavian eine schlechte Magenverträglichkeit von Clopidogrel beobachtet (Gastritis, Magenschleimhauterosionen und/oder Erbrechen).

Mäuse erhielten 78 Wochen und Ratten 104 Wochen Dosen bis zu 77 mg/kg pro Tag (dies entspricht einer mindestens 25-fachen Exposition im Vergleich zu Menschen, die die therapeutische Dosis von 75 mg/Tag erhalten). Dabei zeigte sich kein Hinweis auf eine karzinogene Wirkung.

Clopidogrel wurde in einer Reihe von Invitro- und In-vivo-Untersuchungen auf Genotoxizität untersucht und zeigte keine aenotoxischen Effekte.

Clopidogrel hatte keinen Einfluss auf die Fertilität männlicher und weiblicher Ratten und es zeigte weder bei Ratten noch bei Kaninchen eine teratogene Wirkung. Bei laktierenden Ratten wurde unter Clopidogrel eine leicht verzögerte Entwicklung der Nachkommen beobachtet. Spezifische pharmakokinetische Studien mit radioaktiv markiertem Clopidogrel haben gezeigt, dass die Substanz selbst sowie ihre Metaboliten in die Muttermilch übertreten. Deshalb kann ein direkter Effekt (leichte Toxizität) oder ein indirekter Effekt (Geschmacksbeeinträchtigung) nicht ausgeschlossen werden.

# 6. PHARMAZEUTISCHE ANGABEN

# 6.1 Liste der sonstigen Bestandteile

Kern:

Mannitol (E 421)

Macrogol 6000 Mikrokristalline Cellulose

Hydriertes Rizinusöl

Hyprolose (5,0-16,0% Hydroxypropoxy-

Gruppen) Überzug:

Hypromellose (E 464)

Lactose-Monohydrat

Triacetin (E 1518)

Titandioxid (E 171)

Eisen(III)-oxid (E 172)

Poliermittel: Carnaubawachs

# 6.2 Inkompatibilitäten

Nicht zutreffend.

# 6.3 Dauer der Haltbarkeit

3 Jahre

# 6.4 Besondere Vorsichtsmaßnahmen für die Aufbewahrung

In PVC/PVDC/Aluminium-Blisterpackungen: Nicht über 30 °C lagern.

In Aluminium/Aluminium-Blisterpackungen: Für dieses Arzneimittel sind keine besonderen Lagerungsbedingungen erforderlich.

# 6.5 Art und Inhalt des Behältnisses

Plavix 75 mg Filmtabletten

PVC/PVDC/Aluminium-Blisterpackung oder Aluminium/Aluminium-Blisterpackung in Umkartons mit 7, 14, 28, 30, 84, 90 und 100 Filmtabletten.



Perforierte PVC/PVDC/Aluminium-Blisterpackung oder Aluminium/Aluminium-Blisterpackung zur Abgabe von Einzeldosen in Umkartons mit 50 x 1 Filmtablette.

# Plavix 300 mg Filmtabletten

Perforierte Aluminium/Aluminium-Blisterpackung zur Abgabe von Einzeldosen in Umkartons mit  $4 \times 1$ ,  $10 \times 1$ ,  $30 \times 1$  und  $100 \times 1$  Filmtablette.

Es werden möglicherweise nicht alle Packungsgrößen in den Verkehr gebracht.

#### 6.6 Besondere Vorsichtsmaßnahmen für die Beseitigung

Nicht verwendetes Arzneimittel oder Abfallmaterial ist entsprechend den nationalen Anforderungen zu beseitigen.

### 7. INHABER DER ZULASSUNG

Sanofi Clir SNC 54 rue La Boétie

F-75008 Paris – Frankreich

# 8. ZULASSUNGSNUMMERN

Plavix 75 mg Filmtabletten

EU/1/98/069/001a – Umkarton mit 28 Filmtabletten in PVC/PVDC/Aluminium-

Blisterpackungen

EU/1/98/069/001b – Umkarton mit 28 Filmtabletten in Aluminium/Aluminium-Blisterpackungen

EU/1/98/069/002a – Umkarton mit 50 × 1 Filmtablette in PVC/PVDC/

Aluminium-Blisterpackungen

EU/1/98/069/002b - Umkarton mit

50 x 1 Filmtablette in Aluminium/ Aluminium-Blisterpackungen

EU/1/98/069/003a – Umkarton mit

84 Filmtabletten in PVC/PVDC/Aluminium-

Blisterpackungen EU/1/98/069/003b – Umkarton mit

84 Filmtabletten in Aluminium/Aluminium-

Blisterpackungen

Blisterpackungen EU/1/98/069/004a – Umkarton mit

100 Filmtabletten in PVC/PVDC/Alumini-

um-Blisterpackungen

EU/1/98/069/004b – Umkarton mit

100 Filmtabletten in Aluminium/Aluminium-Blisterpackungen

EU/1/98/069/005a – Umkarton mit

30 Filmtabletten in PVC/PVDC/Aluminium-

Blisterpackungen EU/1/98/069/005b – Umkarton mit

30 Filmtabletten in Aluminium/Aluminium-

Blisterpackungen

EU/1/98/069/006a – Umkarton mit 90 Filmtabletten in PVC/PVDC/Aluminium-

Blisterpackungen

EU/1/98/069/006b – Umkarton mit 90 Filmtabletten in Aluminium/Aluminium-

Blisterpackungen EU/1/98/069/007a – Umkarton mit

14 Filmtabletten in PVC/PVDC/Aluminium-Blisterpackungen

EU/1/98/069/007b – Umkarton mit

14 Filmtabletten in Aluminium/Aluminium-Blisterpackungen

EU/1/98/069/011a – Umkarton mit 7 Filmtabletten in PVC/PVDC/Aluminium-Blisterpackungen

EU/1/98/069/011b – Umkarton mit 7 Filmtabletten in Aluminium/Aluminium-Blisterpackungen

003345-31445



Plavix® 75 mg Filmtabletten Plavix® 300 mg Filmtabletten

Plavix 300 mg Filmtabletten EU/1/98/069/008 - Umkarton mit 4 × 1 Filmtablette in perforierten Aluminium/Aluminium-Blisterpackungen zur Abgabe von Einzeldosen. EU/1/98/069/009 - Umkarton mit  $30 \times 1$  Filmtablette in perforierten Aluminium/Aluminium-Blisterpackungen zur Abgabe von Einzeldosen. EU/1/98/069/010 - Umkarton mit  $100 \times 1$  Filmtablette in perforierten Aluminium/Aluminium-Blisterpackungen zur Abgabe von Einzeldosen. EU/1/98/069/012 - Umkarton mit 10 × 1 Filmtablette in perforierten Aluminium/Aluminium-Blisterpackungen zur Abgabe von Einzeldosen

### 9. DATUM DER ERTEILUNG DER ZULASSUNG/VERLÄNGERUNG **DER ZULASSUNG**

Datum der Erteilung der Zulassung: 15. Juli 1998

Datum der letzten Verlängerung der Zulas-15. Juli 2008

# 10. STAND DER INFORMATION

Januar 2018

Ausführliche Informationen zu diesem Arzneimittel sind auf den Internetseiten der Europäischen Arzneimittel-Agentur http://www.ema.europa.eu/ verfügbar.

# **VERKAUFSABGRENZUNG**

Deutschland

Verschreibungspflichtig.

Österreich

Rezept- und apothekenpflichtig.

Für weitere Informationen zu diesem Arzneimittel wenden Sie sich bitte an den örtlichen Vertreter des Zulassungsinhabers:

Deutschland

Sanofi-Aventis

Deutschland GmbH

D-65926 Frankfurt am Main

Postanschrift:

Postfach 80 08 60

D-65908 Frankfurt am Main

Tel.: 0800 52 52 010

Tel. aus dem Ausland: +49 69 305 21 131

E-Mail: medinfo.de@sanofi.com

Österreich

sanofi-aventis GmbH

Leonard-Bernstein-Straße 10 A-1220 Wien

Telefon: +43 1 80 185-0

Zentrale Anforderung an:

Rote Liste Service GmbH

Fachinfo-Service

Mainzer Landstraße 55 60329 Frankfurt

003345-31445

Januar 2018

Until the information herein is released by Otsuka to the public domain, the contents of this document are Otsuka confidential information and should not be duplicated or re-distributed without prior written consent of Otsuka.